Page: 1

Protocol Number: MB102230 IND Number: 68,652

Ex-US Non-IND

EUDRACT Number 2014-004599-49

Date: 05-Feb-2015

Revised Date: 18-May-2016

# **Clinical Protocol MB102230**

A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Dapagliflozin as an Add-on to Insulin Therapy in Subjects with Type 1 Diabetes Mellitus - Study Two

Revised Protocol Number: 02 Incorporates amendment: 05

### **Study Director/Medical Monitor**

Lars Hansen, MD, PhD Route 206 & Province Line Road Lawrenceville, NJ 08543



24-hr Emergency Telephone Number Emergency Telephone Number



**Sponsor:** AstraZeneca AB, 151 85 Södertälje, Sweden Study being conducted by Bristol-Myers Squibb on behalf of AstraZeneca AB

### **Bristol-Myers Squibb Research and Development**

Avenue de Finlande 4 B-1420 Braine-l'Alleud, Belgium Route 206 & Province Line Road Lawrenceville, NJ 08543

This document is the confidential and proprietary information of Bristol-Myers Squibb Company and its global affiliates (BMS). By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS-sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis

within your organization or to your independent ethics committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (eg, amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to return it to BMS or promptly destroy it. All other rights reserved. References to BMS in this protocol may apply to partners to which BMS has transferred obligations, eg, a Contract Research Organization (CRO).

Replace all previous version(s) of the protocol with this revised protocol and please provide a copy of this revised protocol to all study personnel under your supervision, and archive the previous versions.

# **DOCUMENT HISTORY**

| Document | Date of Issue | Summary of Change |
|---|---|---|
| Revised Protocol<br>02 | 18-May-2016 | Incorporates Amendment 05 |
| Amendment 05 | 18-May-2016 | The primary purpose of this amendment is to provide study visit scheduling flexibility by allowing optional phone visits to be done at week 4, week 2 and for the Continuous Glucose Monitoring visits (weeks 10/11 and weeks 22/23) during the 24 week double blinded short term treatment period. Additional changes in this amendment include: • Adding an exploratory endpoint to compare the number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of >0.5% on dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin from baseline to Week 24 visit. • Updating the guidance on DKA assessments and reporting to include the following: − Reductions in insulin doses of more than 20% are not recommended regardless of glucose values. If blood glucose is repeatedly low and a 20% reduction in total daily insulin dose cannot be avoided the daily dietary carbohydrate intake should be increased, as well as during and/or after elevated physical activity. − Investigators are recommended to advise subjects to take extra insulin and extra carbohydrates if elevated ketones are registered and to continue to measure blood ketones. Study medication should be interrupted during sick days if necessary − For subjects who report elevated ketones/ketosis or a DKA, it is recommended that the investigator consider reeducation concerning DKA at the next scheduled visit, at an un-scheduled visit or by telephone contact • Adding that if total daily insulin dose is reduced upon initiation of study medication, attempts must be made to titrate insulin back to baseline total daily insulin dose. It is not recommended to reduce total daily insulin dose by more than 20% compared to baseline at any time during the study unless medically indicated and close attention should be paid, especially in these subjects, to symptoms of, and risk factors for developing DKA. • Revising the upper range of the Week -1 Visit: Central laboratory HbA1c to ≤ 10.5% • Adding multiple statistically related |

Clinical Protocol MB102230 BMS-512148 dapagliflozin

| Revised Protocol 06-May-2015 Revised Protocol 06-May-2015 The primary purpose of the amendment was to modify the Inclusion and Exclusion Criteria based on Fedding alignment that HbA1c may not drop more than 0.5% during the lead-ip phase. Adding guidance around requirements for performing the continue glucose monitoring (CGM) assessments, recording meal information or the that HbA1c may not drop more than 0.5% during the lead-ip phase. Additional changes in the amendment include: Adding guidance and and requirements for performing the continue glucose rounding the requirement that HbA1c may not drop more than 0.5% during the lead-ip hase. Additional changes in the amendment include: Additional c | Document | <b>Date of Issue</b> | Summary of Change |
|---|---|---|---|
| Amendment 03 O6-May-2015 The primary purpose of the amendment was to modify the Inclusion and Exclusion Criteria based on feedback from the European Medicines Agency (EMA). Specifically, the EMA has endorsed removing the requirement that HbA1c may not drop more than 0.5% during the leadiphase. Additional changes in the amendment include: • Adding guidance around requirements for performing the continual glucose monitoring (CGM) assessments, recording meal informatical and performing the 6-point self monitoring blood glucose (SMB) for subjects who are lead-in failures or who discontinue stumedication • Harmonizing the criteria for monitoring and discontinuing subjective function tests with the hepatic adjudication criterial and yof the screening or lead-in criterial and were not subsequent randomized within the applicable study visit windows (e.g. due to planned medical procedure, vacation plans, or employme commitments) • Added a 7 day window to the current Lead-in Period window of 56 days for subjects who have a one-time HbA1c retest at Week -1 | | | <ul> <li>Removing the PK Sampling required at the Day 1 visit</li> <li>Confirming that subjects are to record day and time of CGM sensor insertion if performed at home at week 11 and week 23</li> <li>Reinforcing that all results recorded in subject diary are to be reviewed by site staff during each study visit and that determination of a DKA event must be assessed and documented by the Principal Investigator or by a qualified sub-investigator</li> <li>Adding guidance on recording blood ketone and glucose values associated with events that are deemed not to be a DKA event</li> <li>Including local injections such as intramuscular or intra-articular in the systemic corticosteroid therapy exclusion criteria as well as adding drops to the topical corticosteroids that are allowed in the study</li> <li>Clarifying that the Data Monitoring Committee will periodically evaluate the incidence of hypoglycemia and DKA events, as well as AEs, laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects.</li> <li>Adding multiple updates, confirmations and additions in the Study</li> </ul> |
| Exclusion Criteria based on feedback from the European Medicines Agency (EMA). Specifically, the EMA has endorsed removing the requirement that HbA1c may not drop more than 0.5% during the leadiphase. Additional changes in the amendment include: • Adding guidance around requirements for performing the continue glucose monitoring (CGM) assessments, recording meal information and performing the 6-point self monitoring blood glucose (SMB for subjects who are lead-in failures or who discontinue stumedication • Harmonizing the criteria for monitoring and discontinuing subject with elevated liver function tests with the hepatic adjudication crite • Providing guidance on allowing subjects to rescreen if they did a fail any of the screening or lead-in criteria and were not subsequent randomized within the applicable study visit windows (e.g. due to planned medical procedure, vacation plans, or employme commitments) • Added a 7 day window to the current Lead-in Period window of 56 5 days for subjects who have a one-time HbA1c retest at Week -1 | | 06-May-2015 | Incorporates Amendment 03 |
| | Amendment 03 | 06-May-2015 | <ul> <li>Agency (EMA). Specifically, the EMA has endorsed removing the requirement that HbA1c may not drop more than 0.5% during the lead-in phase.</li> <li>Additional changes in the amendment include:</li> <li>Adding guidance around requirements for performing the continuous glucose monitoring (CGM) assessments, recording meal information, and performing the 6-point self monitoring blood glucose (SMBG) for subjects who are lead-in failures or who discontinue study medication</li> <li>Harmonizing the criteria for monitoring and discontinuing subjects with elevated liver function tests with the hepatic adjudication criteria</li> <li>Providing guidance on allowing subjects to rescreen if they did not fail any of the screening or lead-in criteria and were not subsequently randomized within the applicable study visit windows (e.g. due to a planned medical procedure, vacation plans, or employment commitments)</li> <li>Added a 7 day window to the current Lead-in Period window of 56 +</li> </ul> |
| Original Protocol 05-Feb-2015 Not applicable | Original Protocol | 05-Feb-2015 | Not applicable |

#### **SYNOPSIS**

#### **Clinical Protocol MB102230**

**Protocol Title:** A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Dapagliflozin as an Add-on to Insulin Therapy in Subjects with Type 1 Diabetes Mellitus - Study Two

# Investigational Products, Dose and Mode of Administration, Duration of Treatment with Investigational Products:

- Blinded dapagliflozin tablets 5 mg, and 10 mg administered orally for the 24-week double-blind short-term treatment period, and the 28-week subject- and site-blinded long-term treatment period of the study
- Matching placebo administered orally for the 24-week double-blind short-term treatment period, and the 28-week subject and site blinded long-term treatment period of the study.

#### **Study Phase: 3**

**Research Hypothesis:** After 24 weeks of oral administration of double-blind treatment, the change from baseline in hemoglobin A1c (HbA1c) with dapagliflozin plus insulin will be greater than placebo plus adjustable insulin in subjects with type 1 diabetes mellitus (T1DM) who have inadequate glycemic control. In this study, adjustments of insulin dose can be made as deemed appropriate to be consistent with good medical practice.

### **Objectives:**

#### **Primary Objective**

The primary objective of this study is to compare the change from baseline in HbA1c after 24 weeks of double-blinded treatment with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin.

### **Secondary Objectives:**

### **Efficacy**

- Compare the percent change from baseline in total daily insulin dose with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Compare the percent change from baseline in body weight with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Compare the change from baseline in the mean value of 24-hour glucose readings obtained from continuous glucose monitoring (CGM) with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Compare the change from baseline in mean amplitude of glucose excursion (MAGE) of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Compare the change from baseline in the percent of 24-hour glucose readings obtained from CGM that falls within the target range of > 70 mg/dL and ≤ 180 mg/dL with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Compare dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin for the proportion of subjects achieving an HbA1c reduction from baseline to Week 24 visit ≥ 0.5% without severe hypoglycemia events

Revised Protocol No.: 02

#### Safety

• To assess the proportion of subjects with hypoglycemia events and the frequency and severity of the hypoglycemia events with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin

• To evaluate the safety and tolerability by assessment of adverse events (AE), vital signs, diabetic ketoacidosis (DKA) events, physical examination findings, ECG, and laboratory values

#### **Other/Exploratory Objectives:**

- Assess the proportion of subjects with HbA1c reduction of at least 0.5% (≥ 0.5%) from baseline with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the proportion of subjects with HbA1c < 7.0% with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in fasting plasma glucose (FPG) with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in the percent of 24-hour glucose readings obtained from CGM that is within the hypoglycemic range of ≤ 70 mg/dL with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in seated systolic blood pressure with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment among subjects with hypertension at baseline, defined as seated SBP ≥ 140 mmHg and/or seated DBP ≥ 90 mmHg
- Assess the change from baseline in average glucose values measured by 6-point self monitored blood glucose (SMBG) with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in postprandial glucose values measured by 6-point SMBG with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in postprandial glucose values measured by CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline in standard deviation of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline to Week 24 in health status, as measured by the Euro Quality of life 5 dimensions 3 levels (EQ-5D-3L) questionnaire, between dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the changes from baseline to Week 24 in the summary score for treatment satisfaction and scores for perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively, as measured by the Diabetes Treatment Satisfaction Questionnaire status (DTSQs) between the dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- Assess the change from baseline to Week 24 in the fear of hypoglycemia as measured by the Hypoglycemia Fear Survey (HFS-II) Worry Subscale score between the dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- To explore the relationship between observed and/or model estimated pharmacokinetic measures of exposure (eg, AUCss, Cmax, Cmin) and efficacy and/or safety endpoints by using model-based approaches. This analysis will be provided in a separate report
- Compare the number of non-severe hypoglycemic events per subject in those achieving an HbA1c reduction of ≥ 0.5% on dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin from baseline to Week 24 visit.

**Study Design:** This trial is a randomized, double-blinded, three-arm, parallel-group, placebo-controlled, multicenter trial to evaluate the efficacy and safety of dapagliflozin, when added to ongoing insulin therapy, in subjects with T1DM and inadequate glycemic control. Approximately 768 subjects will be randomized in this trial. Due to regulatory requirements, approximately 160 subjects (of the 768 subjects) are planned to be be included from Japan.

Potential subjects will be assessed for eligibility criteria at the screening visit. Eligible subjects will enter an 8-week lead-in period in order to optimize their diabetes management based on individual subject challenge to glycemic control (including hyperglycemia, hypoglycemia, erratic meal/exercise patterns, as defined by the investigator) and to assess the variability in blood glucose profiles and frequency of hypoglycemic episodes at baseline. No placebo or study medication will be provided during the lead-in period. On Day 1, subjects who meet all the protocol-specific enrollment and randomization criteria will be randomized into one of the 3 blinded treatment arms (dapagliflozin 5 mg QD, dapagliflozin 10 mg QD, or placebo QD) in a 1:1:1 ratio. Randomization will be stratified to ensure equal representation across all treatment groups by the following: 1) current use of CGM (this refers to an unblinded/personal device which may already be in use before using the blinded device as part of the study and will be categorized as yes vs no); 2) method of insulin administration at baseline (multiple daily injections ([MDI] vs continuous subcutaneous insulin infusion [CSII]); and 3) baseline  $A1C \ge 7.5\%$  and 40.0% vs 4

Subjects will receive dapagliflozin 5 mg QD, 10 mg QD, or placebo QD for 24 weeks, followed by a 28-week subject- and site-blinded long-term treatment period. Besides study medications, subjects will be treated with MDI (three or more injections per day of basal and prandial insulin) or CSII. It is recommended that subjects reduce their daily insulin dose by up to 20% for both basal and bolus insulin after the first dose of study drug on Day 1 to reduce the risk of hypoglycemia, although in some cases it may be necessary to reduce insulin (particularly basal insulin) in advance of study drug administration. It is at the discretion of the investigator to determine the extent to which to reduce the insulin doses. Throughout the study (from the beginning of the lead-in period to the end of the long-term treatment period), insulin dose may be adjusted as deemed appropriate to be consistent with good medical practice according to SMBG readings, local guidance and individual circumstances. Subjects will be monitored closely with regard to safety parameters, including vital signs, safety laboratory tests, ECGs, and AEs.

Figure -1: Study Schematic



#### Notes:

• Eligible subjects should have the Day 1 randomization visit within  $56 \pm 5$  days of the Week -8 entry into lead-in period visit

• Subjects will receive the last dose of study medications on Week 52 visit and they will have the last follow-up visit on Week 56 visit (30 days after Week 52 visit)

Study Drug: includes both Investigational [Medicinal] Products (IP/IMP) and Non-investigational [Medicinal] Products (Non-IP/Non-IMP) as listed:

| Study Drug for MB102230 | | |
|-----------------------------------|---------|-----------|
| Medication | Potency | IP/Non-IP |
| Dapagliflozin Film Coated Tablets | 5mg | IP |
| Background Insulin | Varies | Non-IP |

### **Study Population:**

#### **Key Inclusion Criteria:**

- Diagnosis of T1DM. In addition, a central laboratory C-peptide < 0.7 ng/mL (0.23 nmol/L) is required</li>
- Ages 18 to 75 years, inclusive
- Insulin use for at least 12 months prior to screening per subject reported or medical records and:
  - O Method of insulin administration (MDI or CSII) must have been unchanged for at least 3 months prior to screening per subject reported or medical records. Subjects must be taking a total insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to screening
  - o If using MDI, the subject must be taking  $\geq 3$  injections per day
- HbA1c eligibility criteria include:
  - Screening Visit: Central laboratory HbA1c  $\geq$  7.7% and  $\leq$  11.0%
    - Note: a one-time repeat HbA1C is allowed for subjects in screening if their initial result is within  $\pm$  0.2% of the cut off values
  - Week -1 Visit: Central laboratory HbA1c  $\geq$  7.5 % and  $\leq$  10.5%
    - Note: a one-time repeat HbA1C is allowed for subjects in lead-in if their test result is within  $\pm$  0.2% of the cut off values
- BMI  $\geq 18.5 \text{ kg/m}^2$
- Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product
- WOCBP must agree to follow instructions for method(s) of contraception as outlined in the study
- Women must not be breastfeeding

### **Key Exclusion Criteria:**

- Target Disease Exceptions
  - o History of T2DM

Note: subjects with a previous misdiagnosis of T2DM in their medical history must have one of the following in order to be eligible for this trial:

- Positive autoantibodies for GAD65, phosphatase IA-2/IA2β, or zinc transporter 8 (ZnT8) (eg, autoimmune diabetes)
- Fasting c-peptide value below the lower limit of detection performed by the Central Laboratory
- History of maturity onset diabetes of young (MODY)
- Pancreatic surgery, chronic pancreatitis, or other pancreatic disorders that could result in decreased β-cell capacity (eg, pancreatogenous diabetes)
- o Previous use of dapagliflozin and/or any other SGLT-2 inhibitors
- Use of insulin-sensitizing agents, such as metformin and/or thiazolidinediones, within 2 months prior to the screening visit
- Use of any GLP-1 receptor agonist within the following timeframe prior to the screening visit:
  - i) 1 month for once or twice daily administration (eg, liraglutide)
  - ii) 2 months for once weekly administration
- Any non-insulin, antihyperglycemic agent use within 1 month prior to the Screening visit
- History of diabetes ketoacidosis (DKA) requiring medical intervention (eg, emergency room visit and/or hospitalization) within 1 month prior to the screening visit
- History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to the Screening visit
- o Frequent episodes of severe hypoglycemia as defined by more than one episode requiring medical assistance, emergency care (paramedics or emergency room care), and/or glucagon therapy administered by a third-party individual within 1 month prior to the screening visit
- Symptoms of poorly controlled diabetes that would preclude participation in this trial including but not limited to marked polyuria and polydipsia with greater than 10% weight loss during the 3 months prior to screening, or other signs and symptoms
- o History of Addison's disease or chronic adrenal insufficiency
- History of diabetes insipidus

#### • Medical History and Concurrent Diseases

- o Any of the following cardiovascular (CV)/vascular diseases within 6 months of the screening visit:
  - Myocardial infarction
  - Cardiac surgery or revascularization (coronary artery bypass surgery [CABG]/percutaneous transluminal coronary angioplasty [PTCA])
  - Unstable angina
  - Unstable congestive heart failure (CHF)
  - CHF New York Heart Association (NYHA) Class III or IV
  - Transient ischemic attack (TIA) or significant cerebrovascular disease
  - Unstable or previously undiagnosed arrhythmia
- Renal Disease:
  - History of unstable or rapidly progressing renal disease
  - Conditions of congenital renal glucosuria
  - Renal allograft
- Hepatic Diseases:
  - Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic
    insufficiency
- Hematological and Oncological Disease/Conditions:
  - History of hemoglobinopathy, with the exception of sickle cell trait (SA) or thalassemia minor; or chronic or recurrent hemolysis

930087408 3.0


v3.0

Known immunocompromised status, including but not limited to, individuals who have undergone
organ transplantation or who are positive for the human immunodeficiency virus

- Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 8 weeks prior to the screening visit
- Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma)
- History of bladder cancer
- History of radiation therapy to the lower abdomen or pelvis at any time

#### Physical and Laboratory Test Findings

- $\circ$  Aspartate aminotransferase (AST) > 3x upper limit of normal (ULN)
- o Alanine aminotransferase (ALT) > 3x ULN
- o Serum total bilirubin > 2.0x ULN unless exclusively caused by Gilbert's Syndrome
- O Calculated creatinine clearance (CrCl) < 60 mL/min as estimated by the Cockcroft-Gault formula, using laboratory measurements of serum creatinine collected at the screening visit [Creatinine clearance = [[140 age(yr)]\*weight(kg)/[72\*serum Cr(mg/dl)] (multiply by 0.85 for women]
- o Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women
- o Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody
- Abnormal Free T4

Note: abnormal TSH value at screening will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded. A one-time retest may be allowed after a minimum of 6 weeks following the adjustment of thyroid hormone replacement therapy in subject who have had a prior diagnosis of a thyroid disorder and who are currently receiving thyroid replacement therapy. Such cases should be discussed with the Sponsor prior to re-testing

#### Allergies and Adverse Drug Reaction

• Allergies or contraindication to the contents of dapagliflozin tablets or insulin

### • Sex and Reproductive Status

Women who are pregnant or breastfeeding

#### • Other Exclusion Criteria

- Prisoners or subjects who are involuntarily incarcerated
- Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
- Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program
- o History of bariatric surgery or lap-band procedure within 12 months prior to screening
- Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid (including local injections such as intramuscular or intra-articular, etc.) taken for > 4 weeks within 3 months prior to the Day 1 visit
  - NOTE: Topical (including drops) or inhaled corticosteroids are allowed
- O Any unstable endocrine, psychiatric or rheumatic disorders as judged by the investigator
- Volume-depleted subjects. Subjects at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should carefully monitor their volume status
- Subject who, in the judgment of the investigator, is found to be unlikely to comply with the protocol, or is unable to correctly self-administer subcutaneous insulin injections and/or manage their insulin pump, or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data (including during the lead-in period)
- Subject is currently abusing alcohol or other drugs or has done so within the last 6 months prior to the Day 1 visit


#### **Discontinuation of Subjects from Treatment:**

Subjects MUST discontinue study treatment for any of the following reasons:

- Withdrawal of informed consent (subject's decision to withdraw for any reason)
- Any AE, laboratory abnormality or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject
- Pregnancy
- Termination of the study by the Sponsor
- Loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness
- CrCl < 30 mL/min</li>
  - o If at any time the subject's CrCl (based on Cockroft-Gault) falls below 30 mL/min calculated at the central laboratory and confirmed at a repeated central laboratory measurement (to be obtained within 4 days, whenever possible) the subject should be discontinued from study medication
- Subjects experience at least one protocol-defined hypoglycemia episode that leads to a loss of consciousness and/or seizure as determined by the investigator
- Change of insulin administration method (eg, switch from MDI to CSII, or vice versa)
  - Subjects are not allowed to change their insulin administration methods (eg, from MDI to CSII or vice versa) throughout the study. Under certain situations (eg, the replacement of an insulin pump), the subjects who are on CSII may be on temporary use of MDI. They should restart CSII administration as early as feasible. The period of time when a subject on temporary use of MDI should not be more than 2 weeks
- Subjects with a central laboratory ALT and/or AST > 3xULN will be scheduled for a follow-up visit within 3 days following the receipt of the results. Subjects should be discontinued from study if the initial and repeat laboratory tests meet any of the following criteria:
  - $\circ$  ALT and/or AST are > 3x ULN and total bilirubin (TB) > 2x ULN
  - $\circ$  ALT and/or AST are > 5x ULN for  $\ge 14$  consecutive days, at any time after initial confirmatory results
  - o ALT and/or AST are > 10x ULN

#### **Study Assessments:**

#### **Primary Assessment:**

• Change from baseline in HbA1c

#### **Secondary Assessments:**

- Percent change from baseline to Week 24 in total daily insulin dose
- Percent change from baseline to Week 24 in body weight
- Change from baseline to Week 24 in the mean value of 24-hour glucose readings obtained from CGM
- Change from baseline to Week 24 in mean amplitude of glucose excursion of 24-hour glucose readings obtained from CGM
- Change from baseline to Week 24 in the percent of 24-hour glucose readings obtained from CGM that falls within the range of > 70 mg/dL and  $\le 180$  mg/dL
- Proportion of subjects achieving an HbA1c reduction from baseline to Week 24 visit ≥ 0.5% without severe hypoglycemia events


**Safety Assessments**: Safety assessments will be based on medical review of AE reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests. The incidence of observed AEs will be tabulated and reviewed for potential significance and clinical importance. Both hypoglycemia and DKA during the 24-week double-blinded short-term treament period and the 28-week subject- and site-blinded long-term period (the Sponsor will be unblinded during the long-term treatment period) will be assessed.

Subjects will receive a combined blood glucose and ketone meter, supplies and instructions on their use. Subjects should self-monitor their blood glucose consistent with local treatment guidelines (typically 4 times daily or when experiencing symptoms suggestive of hypoglycemia) and contact the investigator in the event of an unusually high or low blood glucose value. The investigator may require more frequent readings based on local clinical practice. The glucose values should be reviewed by the site to identify any unusual high or low values, and to confirm that the values are obtained from the subject.

Subjects will be advised to measure their blood ketones using a combined blood glucose and ketone meter provided by the Sponsor when they have potential symptoms/signs of DKA (eg, excessive thirst, nausea and vomiting, frequent urination, weakness or fatigue, fruity-scented breath, confusion, and/or consistently elevated blood glucose) and/or during acute illness. Subjects should be instructed to measure their ketones if symptoms occur, regardless of plasma glucose values. Subjects should contact the site for assistance with diabetes management in the event that the blood ketone reading is 0.6 mmol/L or above in accordance with the ketone meter user guide provided.

Subjects must also be instructed that if attempts to contact the site are unsuccessful or if they are in urgent need of medical attention, that they should seek medical attention. They should provide information to the health care provider on their participation in a placebo controlled clinical study evaluating the effects of the SGLT2i dapagliflozin in addition to their insulin treatment.

### **Exploratory Assessments**:

Subjects will be instructed to perform 6-point SMBG profiles according to the schedule presented in the study flow charts. 6-point SMBG profiles will be taken on any 3 days within one week before the scheduled visits, with three glucose measurements obtained preprandially (within 15 minutes prior to meal) and three glucose measurements obtained postprandially (1.5- 2 hours after start of the meal) for the three main meals of the day. Subjects will be provided with a diary to record their SMBG measurements and mealtimes.

CGM will be used periodically to measure the subject's interstitial glucose level according to the schedule presented in Study Flow Charts. A CGM sensor will be inserted subcutaneously at the Week -2 visit, Week -1 visit, Week 10 visit and Week 22 visit to allow monitoring for 2 weeks (for example: the Week -2 visit to the Day 1 visit [baseline]; the Week 10 office visit until the Week 12 office visit; and the Week 22 office visit until the Week 24 office visit.). The data will remain blinded to the subject, the investigator, and to the Sponsor during the recording and will be downloaded into a data file. Detailed procedures (including calibration) will be described in an operations manual and site staff will be fully trained on the use of CGM. Subjects will wear the sensor and perform calibration according to manufacturer's instructions. If a subject uses a CGM device prior to entry into the study, he/she may continue to use the device during the study in accordance with their usual diabetes management care. Such a subject will be required to also use the blinded CGM device according to protocol procedures.

#### **Outcomes Research Assessments:**

Patient reported outcomes (PROs) will be assessed at the Day 1 visit (prior to first dose), the Week 24 visit, and the Week 52 visit by EQ-5D-3L for generic health status, DTSQs for treatment satisfaction, and the HFS-II Worry subscale for worry about hypoglycemia and its negative consequences. The instruments/questions will be self-administered using paper and pencil questionnaires. The EQ-5D-3L is a generic, preference-based utility questionnaire and consists of two parts, the EQ visual analogue scale (VAS) and the EQ-5D-3L index. The EQ VAS ranges from 0 = worst possible health to 100 = best possible health. The EQ-5D-3L index is a questionnaire with five dimensions, which include mobility, self-care, usual activity, pain/discomfort and anxiety/depression. Each item has three levels: no problems, some problems and severe problems. The DTSQ has been developed to assess subjects' satisfaction with treatment and perception of change in hyper- and hypoglycaemia. The DTSQ status version (DTSQs) has 8 items. The HFS-II Worry Subscale is an 18-item questionnaire, in which responses are made on a 5-point Likert scale (where 0 = Never and 4 = Always). The HFS-II Worry Subscale has a score ranging from 0 to 72, with higher scores indicating increased fear of hypoglycaemia.


#### **Data Monitoring Committees:**

An external data monitoring committee (DMC) with multidisciplinary representation will be established to evaluate, on a periodic basis, the incidence of hypoglycemia and DKA events, as well as AEs, laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects. An independent reporting statistician not involved in the conduct of the study will be designated by BMS to provide the DMC with essential safety data during the study. The DMC responsibilities, authorities, and procedures will be documented in a DMC charter.

#### **Statistical Considerations:**

#### **Sample Size:**

With 243 subjects per treatment group with both baseline and at least one post baseline measurement, there is approximately 90% power to detect a difference in means of 0.35% between each dapagliflozin treatment group and placebo at the two-sided 0.0262 significance level (based on Dunnett and Tamhane step-up procedure), assuming a standard deviation (SD) of 1.1%. Assuming that 5% of subjects do not have a post-baseline assessment, a total of 768 subjects (256 subjects per treatment arm) need to be randomized to each dapagliflozin or placebo group in 1:1:1 ratio

Among those 768 subjects, approximately 160 of them will be from Japan in order to support population specific analyses.

A reduction in the primary endpoint of change from baseline in HbA1c of 0.35% was used to determine sample size as this represents a clinically meaningful improvement in glycemic control under the current study design with adjustable background insulin dose. A lesser degree of reduction in HbA1c in combination with other beneficial outcomes in secondary endpoints may also be clinically important.

### **Endpoints:**

#### Statistical Approach / Assumptions

The primary endpoint is the change in HbA1c from baseline to Week 24. The primary estimand for the primary endpoint is *treatment difference at Week 24 if subjects did not discontinue randomized treatment.* In order to maintain an overall Type I error rate of 5% for the endpoint, a Dunnett and Tamhane step-up procedure will be used, which allows for the correlation of 0.5 between the standard normal deviate for each comparison (Dunnett and Tamhane 1992). Applying the Dunnett and Tamhane procedure, statistical significance will be declared for both doses at the two-sided 5% level if the two-sided p-values from both pairwise comparisons are smaller than 5%. If the larger p-value among the two pairwise comparisons is greater than 5% and the smaller p-value is below 2.62%, then statistical significance will be declared for the latter comparison. The primary analysis of the change in HbA1c from baseline to Week 24 will be based on a longitudinal repeated measures analysis using 'direct likelihood'. The analysis will be based on the full analysis dataset who have a baseline assessment and any post-baseline double-blind treatment period assessment. The analysis will include all available data up to Week 24 or until premature discontinuation of randomized treatment, whichever occurs first. The analysis will be conducted regardless of insulin up-titration. The model is based on a missing at random (MAR) assumption with respect to missing data.

The SAS procedure PROC MIXED will be used. The preferred model will include the fixed categorical effects of treatment, week, randomization stratification factor (ie, one term for each combination of all stratification factors) and treatment-by-week interaction, as well as the continuous fixed covariates of baseline measurement and baseline measurement-by-week interaction. An unstructured matrix for the within-subject error variance-covariance will be used. The denominator degrees of freedom will be calculated according to the Kenward-Roger method. A number of back-up models will be defined in the statistical analysis plan in case of non-convergence of the preferred model or other issues. Point estimates and 95% confidence intervals for the mean change within each treatment group, as well as the difference in mean change between the dapagliflozin treatment group and placebo will be calculated. P-values for the difference in Week 24 estimates between each dapagliflozin group and placebo will be calculated

The ITT estimand, i.e., *treatment difference at Week 24 regardless of treatment discontinuation*, will be evaluated as the secondary estimand of the primary endpoint. The analysis of the ITT estimand will include all available data up to Week 24, regardless of insulin up-titration and regardless of premature discontinuation of randomized treatment.

Sensitivity analyses will be conducted for the primary efficacy endpoint to assess the robustness of the primary efficacy results, including sensitivity analysis with respect to the ITT estimand, sensitivity analyses based on

missing-not-at-random (MNAR) assumptions with respect to missing data, and sensitivity analysis with respect to insulin up-titration.

Statistical tests for secondary efficacy endpoints will be only conducted if there is a statistically significant difference in the primary endpoint for both pairwise comparisons, i.e., dapagliflozin 5mg vs. placebo and dapagliflozin 10mg vs. placebo. The same Dunnett and Tamhane step-up procedure will be applied to each secondary efficacy endpoint. Secondary efficacy endpoints will be tested in the order that they appear in the objectives section of the protocol and protocol synopsis. Statistical tests will be only performed for a given secondary endpoint if both comparisons for a proceeding secondary endpoint are significant. Otherwise, the testing procedure will stop at the secondary endpoint that does not reach statistical significance.

The percent change (using logarithmic transformation for the endpoint in the model) from baseline to Week 24 in total daily insulin dose and total body weight, the change from baseline to Week 24 in the mean value of 24-hour glucose readings obtained from CGM, mean amplitude of glucose excursion of 24-hour glucose readings obtained from CGM, and the percent of 24-hour glucose readings obtained from CGM that fall within the range of > 70 mg/dL and  $\le 180 \text{ mg/dL}$  will be analyzed using a longitudinal repeated measures analysis, similarly to the model used for the primary efficacy analysis. The proportion of subjects achieving an HbA1c reduction from baseline to Week  $24 \ge 0.5\%$  without severe hypoglycemia events will be analyzed using a logistic regression model with adjustment for baseline values. In addition to point estimates and 2-sided 95% confidence intervals, p-values will be calculated for all endpoints. Nominal p-values will be presented for endpoints where type 1 error is not controlled All secondary efficacy analyses will use subjects in the primary efficacy dataset (ie, full analysis dataset) who have a baseline assessment and any post-baseline double-blind treatment period assessment.

#### **Analysis and Reporting:**

There will be one study report at the end of short-term period and a second study report at the end of short-term plus long-term period.

The PK analysis may be provided in a separate report.


# TABLE OF CONTENTS

| TITLE PAGE | - |
|-------------------------------------------------------------------------|----|
| DOCUMENT HISTORY | |
| SYNOPSIS | |
| TABLE OF CONTENTS | |
| 1 INTRODUCTION AND STUDY RATIONALE | |
| 1.1 Study Rationale | |
| 1.1.1 Unmet Medical Need in Type 1 Diabetes Mellitus | |
| 1.1.2 Introduction of Dapagliflozin and Study Rationale | |
| 1.2 Research Hypothesis | |
| 1.3 Objectives | |
| 1.3.1 Primary Objectives | |
| 1.3.2 Secondary Objectives | |
| 1.3.2.1 Efficacy | |
| 1.3.2.2 Safety | |
| 1.3.3 Other/Exploratory Objectives | |
| 1.4 Product Development Background | |
| 2 ETHICAL CONSIDERATIONS | |
| 2.1 Good Clinical Practice | |
| 2.2 Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | |
| 2.3 Informed Consent | |
| 3 INVESTIGATIONAL PLAN | |
| 3.1 Study Design and Duration | |
| 3.2 Post Study Access to Therapy | |
| 3.3 Study Population | |
| 3.3.1 Inclusion Criteria | |
| 3.3.2 Exclusion Criteria | |
| 3.3.3 Women of Childbearing Potential | |
| 3.4 Concomitant Treatments | |
| 3.4.1 Prohibited and/or Restricted Treatments | |
| 3.4.2 Other Restrictions and Precautions | |
| 3.5 Discontinuation of Subjects from Treatment | 38 |
| 3.5.1 Discontinuation Guidelines due to Protocol-Defined Hypoglycemia | |
| Episode or Recurrent Hypoglycemia Episodes | 39 |
| 3.6 Post Study Drug Study Follow up | 39 |
| 3.6.1 Withdrawal of Consent | 4( |
| 3.6.2 Lost to Follow-Up | 40 |
| 4 STUDY DRUG | |
| 4.1 Investigational Product | 43 |
| 4.2 Non-investigational Product | |
| 4.3 Storage and Dispensing | |
| 4.4 Method of Assigning Subject Identification | 43 |
| 4.4.1 Subjects entering the 24-week double-blinded short-term treatment | |
| period | 44 |
| * | |

| | 4.4.2 Subjects entering the 28-week long-term subject and site blinded |
|---|---|
| | treatment period |
| 4.5 | Selection and Timing of Dose for Each Subject |
| 4.6 | Blinding/Unblinding |
| 4.7 | Treatment Compliance |
| | Destruction and Return of Study Drug |
| | 4.8.1 Destruction of Study Drug |
| | Return of Study Drug |
| 4.10 | Retained Samples for Bioavailability / Bioequivalence |
| | DY ASSESSMENTS AND PROCEDURES |
| 5.1 | Flow Chart/Time and Events Schedule |
| | 5.1.1 Retesting During Screening or Lead-in Period |
| | Study Materials |
| | Safety Assessments |
| | 5.3.1 Imaging Assessment for the Study |
| | 5.3.2 Self-Monitored Blood Glucose (SMBG) and Guidance on Management |
| | and Reporting of Hypoglycemia Episodes |
| | 5.3.2.1 Self-Monitored Blood Glucose (SMBG) |
| | 5.3.2.2 Guidance on Management and Reporting of Hypoglycemia |
| | Episodes |
| | 5.3.3 Self-Monitored Blood Ketone Testing and Guidance on Management and |
| | Reporting of Diabetic Ketoacidosis Episodes |
| | 5.3.4 Insulin Dosing Adjustment and Data Collection Guidelines |
| | 5.3.5 Guidance on Assessment of Urinary Infections and Hematuria |
| | 5.3.5.1 Guidance on Assessment of Urinary Infections |
| | 5.3.5.2 Guidance on Assessment of Hematuria |
| | 5.3.6 Guidance on Assessment of Cardiovascular Events |
| | 5.3.7 Guidance on Assessment of Hepatic Laboratory Abnormalities |
| | 5.3.8 Physical Examination |
| | 5.3.9 Blood Pressure and Heart Rate |
| | 5.3.10 Electrocardiograms |
| | 5.3.11 Guidance on Volume Depletion |
| | 5.3.12 Guidance on Monitoring Renal Function |
| | 5.3.13 Supplemental Visits |
| | 5.3.13.1 Early Treatment Discontinuation Visit |
| | 5.3.13.2 Early Treatment Discontinuation Follow-up (Off Treatment |
| | Procedures) |
| | 5.3.13.3 Other Supplemental (Unscheduled) Visits |
| 5 4 | Efficacy Assessments. |
| | Pharmacokinetic Assessments |
| | Pharmacogenomic/Pharmacogenetic Assessements |
| | Biomarker Assessments |
| | Outcomes Research Assessments |
| | 5.8.1 EQ-5D-3L |
| | 5.8.2 Diabetes Treatment Satisfaction Questionnaire |
| | 5.8.3 Hypoglycemia Fear Survey |
| | J.U.J IIVIOTIVEHIIU I'EUI DUI VEV |

| 5.9 Other Assessments | 77 |
|-----------------------------------------------------------|----------|
| 5.9.1 Weight | 77 |
| 5.9.2 Height and Body Mass Index (BMI) | 77 |
| 5.9.3 Diet and Exercise Counseling | 78 |
| 5.9.4 Pharmacodynamic Assessments | 78 |
| 5.9.4.1 Fasting Plasma Glucose | 78 |
| 5.9.4.2 6-point SMBG profiles | 78 |
| 5.9.4.3 Continuous Glucose Monitoring (CGM) | 79 |
| 5.10 Results of Central Laboratory Assessments | 80 |
| 6 ADVERSE EVENTS | 80 |
| 6.1 Serious Adverse Events | 81 |
| 6.1.1 Serious Adverse Event Collection and Reporting | 82 |
| 6.2 Nonserious Adverse Events | 83 |
| | 83 |
| 6.2.1 Nonserious Adverse Event Collection and Reporting | 83 |
| 6.3 Laboratory Test Result Abnormalities | 84 |
| 6.4 Pregnancy | |
| 6.5 Overdose | 84<br>84 |
| 6.6 Potential Drug Induced Liver Injury (DILI) | |
| 6.7 Other Safety Considerations | 85 |
| 6.7.1 AEs of Special Interest | 85 |
| 7 DATA MONITORING COMMITTEE AND OTHER EXTERNAL COMMITTEES | |
| | 85 |
| 7.1 Cardiovascular Adjudication Committee | 85 |
| 7.2 Hepatic Adjudication Committee | 86 |
| 7.3 DKA Adjudication Committee | 86 |
| 7.4 Data Monitoring Committee (DMC) | 86 |
| 8 STATISTICAL CONSIDERATIONS | 86 |
| 8.1 Sample Size Determination | 86 |
| 8.2 Populations for Analyses | 87 |
| 8.3 Endpoints | 88 |
| 8.3.1 Primary Endpoint | 88 |
| 8.3.2 Secondary Endpoints | 88 |
| 8.3.3 Safety | 88 |
| 8.3.4 Exploratory Endpoints | 89 |
| 8.4 Analyses | 89 |
| 8.4.1 Demographics and Baseline Characteristics | 90 |
| 8.4.2 Efficacy Analyses | 90 |
| 8.4.2.1 Primary Efficacy Analyses | 90 |
| 8.4.2.2 Secondary Efficacy Analyses | 91 |
| 8.4.2.3 Exploratory Efficacy Analyses | 91 |
| 8.4.3 Safety Analyses | 92 |
| 8.4.4 Pharmacokinetic Analyses | 92 |
| 8.4.5 Biomarker Analyses | 93 |
| 8.4.6 Outcomes Research Analyses | 93 |
| 8.4.7 Other Analyses | 93 |
| 8.5 Interim Analyses | 93 |
| 6.5 mermi Anaryses | 75 |

| BMS-512148 | MB102230<br>dapagliflozin |
|---|---|
| 9 STUDY MANAGEMENT | 93 |
| 9.1 Compliance | 93 |
| 9.1.1 Compliance with the Protocol and Protocol Revisions | 93 |
| 9.1.2 Monitoring | 94 |
| 9.1.3 Investigational Site Training | 94 |
| 9.2 Records | 94 |
| 9.2.1 Records Retention | 94 |
| 9.2.2 Study Drug Records | 95 |
| 9.2.3 Case Report Forms | 95 |
| 9.3 Clinical Study Report and Publications | 96 |
| 10 GLOSSARY OF TERMS | 97 |
| 11 LIST OF ABBREVIATIONS | 98 |
| 12 REFERENCES | 102 |
| APPENDIX 1 NEW YORK HEART ASSOCIATION FUNCTIONAL CLASS | 104 |
| APPENDIX 2 CENTRAL LABORATORY ASSESSMENTS | 105 |
| APPENDIX 3 SUSTAINED ELEVATED LIVER SAFETY ABNORMALITIES | |
| FLOW CHART | 110 |

#### 1 INTRODUCTION AND STUDY RATIONALE

### 1.1 Study Rationale

# 1.1.1 Unmet Medical Need in Type 1 Diabetes Mellitus

Type 1 diabetes mellitus (T1DM) is a serious chronic disorder that results in the destruction of insulin-producing pancreatic β-cells. T1DM accounts for approximately 5-10% of all cases of diabetes worldwide, and its incidence continues to increase. Patients with T1DM require lifelong insulin therapy due to their inability to produce endogenous insulin. Insulin requirements in these subjects vary widely and depend on several factors including body weight, activity level, and food intake.

People with T1DM must balance the goal of long-term glycemic control and reduction of complications of the disease with the day-to-day challenges of insulin therapy. The major limiting factor for restoring euglycemia is insulin-related hypoglycemia. Unfortunately, recent data suggest hypoglycaemia remains a common event, with 11.8% of subjects in a clinic registry study experiencing at least one episode of severe hypoglycemia resulting in seizure or loss of consciousness within the past 12 months. The occurrence of severe hypoglycemia did not appear to be related to hemoglobin A1C (HbA1c). However, the risk of recurrent hypoglycemia episodes in T1DM can be related to the degree of glycemic variability, which suggests that reducing the swings in glucose may be of importance in this population.

Intensive insulin therapy is also associated with weight gain and insulin resistance, as evidenced in the Diabetes Control and Complications Trial, where subjects in the intensive treatment arm gained an average of 4.6 kg more than the control group over the 5 year study. It has been postulated that the weight gain associated with intensive insulin treatment is related to reductions in urinary glucose excretion, increased appetite, and the ingestion of excess calories to manage or avoid hypoglycemia. Weight gain and insulin resistance may have a significant deleterious impact upon cardiovascular risk factors, at least in some people with T1DM, and has recently contributed to the concept of 'double diabetes."

Average HbA1c values greater than 8% have been reported in several large studies in people with T1DM, <sup>9,10</sup> suggesting a large proportion of the population are unable to achieve recommended glycemic levels with insulin alone because of the challenges associated with insulin therapy. Novel therapies used as an adjunct to insulin that improve glycemic control and provide important secondary benefits, such as reductions in insulin dose, hypoglycemia and glycemic variability, and attenuation of weight gain associated with insulin, address important unmet needs for people with T1DM.

### 1.1.2 Introduction of Dapagliflozin and Study Rationale

This Phase 3 study is designed to evaluate the efficacy and safety of dapagliflozin 5 mg and 10 mg as an add-on to insulin therapy when used in subjects with T1DM with inadequate glycemic control.


Dapagliflozin is a stable, competitive, reversible, highly selective, and orally active inhibitor of sodium glucose cotransporter 2 (SGLT-2), the major transporter responsible for renal glucose reabsorption. Dapagliflozin has been recently approved for the treatment of type 2 diabetes mellitus (T2DM). Dapagliflozin is marketed in 40 countries/regions, including the European Union (EU; 5 or 10 mg dapagliflozin), United States (5 or 10 mg dapagliflozin), and Australia (10 mg dapagliflozin only), and is under investigation for marketing in numerous countries around the world.

The mechanism of action (MOA) for dapagliflozin is different from and complementary to the mechanisms of existing medications in other drug classes for T2DM, resulting in the direct, and insulin-independent, elimination of glucose by the kidney. Furthermore, as SGLT-2 is almost exclusively expressed in the kidney, the highly selective nature of dapagliflozin minimizes the risk of off-target (ie, non-kidney) effects. Therefore, no effects are observed on glucose and/or other carbohydrate transport or absorption in any other organs, including the gut, and no other transporters are affected. As such, dapagliflozin offers an important additional strategy for improving glycemic control as an add-on to insulin in patients with T1DM.

Urinary glucose excretion induced by dapagliflozin depends upon the amount of glucose filtered by the kidney (Figure 1.1.2-1). This filtered load is the product of the plasma glucose concentration and the glomerular filtration rate (GFR). Therefore, the action of dapagliflozin is dependent upon the patient's plasma glucose and renal function, and is independent of the patient's beta cell function or insulin sensitivity, which translates into a relatively low risk of hypoglycemia. Furthermore, because the mechanism reduces hyperglycemia independently of insulin secretion or action, this approach to antidiabetic therapy provides an opportunity to achieve clinically important glycemic efficacy as an add-on to insulin in patients with T1DM.


Date: 18-May-2016

v 3.0 930087408 3.0

20

Figure 1.1.2-1: How Dapagliflozin Works (Mechanism of Action)



Multiple Phase 2 and Phase 3 studies, where dapagliflozin was used as monotherapy or in combination with other oral hypoglycemic agents or insulin in subjects with T2DM, have shown that there is a dose-dependent decrease in fasting plasma glucose (FPG) from baseline to Week 12 (Phase 2 studies) and Week 24 (Phase 3 studies) with dapagliflozin treatment. Dapagliflozin is also associated with a significant reduction of HbA1c from baseline compared to placebo (0.4-0.56% and 0.54-0.68% for the 5 and 10 mg doses, respectively 11).

In addition, dapagliflozin as add on therapy to insulin is now being investigated as a potential treatment for patients with T1DM with inadequate glycemic control (defined as HbA1c  $\geq$  7.5%). Dapagliflozin may be a clinically relevant adjunctive therapy for patients with T1DM given its insulin-independent mechanism of action. Because patients with T1DM are insulin deficient, insulin treatment is required for preventing ketoacidosis and ultimately for survival. Thus, dapagliflozin would not be a replacement for insulin therapy in the setting of T1DM. However, dapagliflozin reduces blood glucose levels by an insulin-independent mechanism and may be effective in improving glycemic control in patients with T1DM when used in combination with insulin. In the T1DM population, the inhibition of urinary glucose reabsorption via SGLT-2 inhibition is expected to produce a glucose lowering similar to that observed in the T2DM population, as well as the modest reductions in blood pressure and body weight. Furthermore, the amount of urinary glucose excreted following treatment with dapagliflozin is dependent upon the plasma glucose concentration,  $^{12}$  which may serve to blunt the excursions of glucose values over the course of the day (reduce glycemic variability).

The potential of dapagliflozin as a treatment option for the T1DM population was explored in a Phase 2a pilot study (MB102072). The MB102072 study was a randomized, double-blind, 5-arm, parallel-group, placebo-controlled exploratory trial to evaluate the safety, tolerability,

pharmacokinetics (PK) and pharmacodynamics (PD) of dapagliflozin in subjects with T1DM who had inadequate glycemic control on insulin therapy. Subjects taking insulin monotherapy who met the central laboratory enrollment requirement of HbA1c  $\geq 7.0\%$  and  $\leq 10.0\%$  were randomly assigned in a 1:1:1:1:1 ratio to one of 5 blinded treatment arms: placebo, 1 mg, 2.5 mg, 5 mg, or 10 mg of dapagliflozin once daily. Subjects received dapagliflozin or matching placebo for a total of 14 days and remained confined to the inpatient unit from Day -3 to Day 7, at which point they were discharged. Subjects then had outpatient visits on Day 10, Day 14, and a discharge visit on Day 21. In this pilot study, dapagliflozin was generally well tolerated at all doses in subjects with T1DM. Hypoglycemia events were frequent in this population during study treatment. Events were relatively balanced across treatment groups. Consistent with the known mechanism of action of dapagliflozin, dose-related increases in 24 hour urinary glucose were observed. Based upon the similar PK characteristics in subjects with T1DM compared to T2DM or healthy subjects, the exposure response relationship in terms of urinary glucose excretion appeared to be virtually identical in this T1DM population to that previously described in T2DM subjects, correcting for baseline differences in glycemic control and eGFR between the studies. Because dapagliflozin 5 mg was established as the minimally effective dose in T2DM and the marked similarities in the PK and PD response that drives efficacy, it is expected that dapagliflozin 5 mg will also be the minimally effective dose in subjects with T1DM. Evaluation of exploratory endpoints suggests a potential for dapagliflozin to improve glycemic control in subjects with T1DM as evidenced by:

- Dose-related trends toward reduction in FPG at Day 7
- Dose-related trends toward reduction in average daily glucose at Day 7 from continuous glucose monitoring (CGM)
- Trends to reduce glycemic variability over the day as evidenced by reduction in the standard deviation of 24-hour glucose values and reduction in the mean amplitude of glucose excursion (MAGE) determined from CGM at Day 7
- Trends towards increased percentage of CGM readings at Day 7 in the target range (> 70 mg/dl to  $\leq 180 \text{ mg/dl}$ )
- Trend towards reduction in total daily insulin dose with all dapagliflozin treatment

In completed clinical studies in subjects with both T2DM and T1DM, dapagliflozin was generally safe and well-tolerated. No clinically relevant changes from baseline were seen in either renal function or serum electrolytes in subjects treated with dapagliflozin. In Phase 2/3 studies in subjects with T2DM, the frequency of overall AEs was similar to placebo. In the Phase 2 study in subjects with T1DM (MB102072), the frequency of overall AEs was similar to placebo. Compared to subjects with T2DM, hypoglycemia was more frequent in subjects with T1DM, but the frequency of hypoglycemia was relatively balanced across dapagliflozin treatment and placebo groups. Urine ketone tests revealed frequent positive urine ketones in this study, with a possibly slight increase in subjects receiving dapagliflozin 10 mg. No diabetic ketoacidosis (DKA) was observed during the study period (from the start of study drugs to the end of follow-up).


930087408 3.0

v3.0

It is expected that dapagliflozin will exhibit an efficacy and safety profile in subjects with T1DM that will be similar to that observed in T2DM. In fact, dapagliflozin may be a potentially novel adjunct to insulin therapy for the treatment of T1DM. Dapagliflozin potently decreases HbA1c and may provide important secondary benefits, such as reductions in total daily insulin dose, hypoglycemia, and glycemic variability and may attenuate the weight gain associated with insulin use to address important unmet needs for people with T1DM.

### 1.2 Research Hypothesis

In subjects with T1DM that have inadequate glycemic control with insulin alone, the addition of dapagliflozin to adjustable insulin will result in a greater mean reduction in HbA1c after 24 weeks of double-blind treatment, as opposed to placebo plus adjustable insulin. In this study, adjustments of insulin dose can be made as deemed appropriate to be consistent with good clinical practice.

### 1.3 Objectives

# 1.3.1 Primary Objectives

The primary objective of this study is to compare the change from baseline in HbA1c between dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment.

### 1.3.2 Secondary Objectives

# 1.3.2.1 Efficacy

Six secondary efficacy objectives are identified:

- 1) Compare the percent change from baseline in total daily insulin dose with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 2) Compare the percent change from baseline in body weight with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 3) Compare the change from baseline in the mean value of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 4) Compare the change from baseline in mean amplitude of glucose excursions (MAGE) of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 5) Compare the change from baseline in the percent of 24-hour glucose readings obtained from CGM that falls within the target range of > 70 mg/dL and ≤ 180 mg/dL with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 6) Compare dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin for the proportion of subjects achieving an HbA1c reduction from baseline to Week 24 visit ≥ 0.5% without severe hypoglycemia events

### 1.3.2.2 Safety

1) To assess the proportion of subjects with hypoglycemia events and the frequency and severity of the hypoglycemia events with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin

2) To evaluate the safety and tolerability by assessment of AEs, vital signs, DKA events, physical examination findings, ECGs, and laboratory values

# 1.3.3 Other/Exploratory Objectives

- 1) Assess the proportion of subjects with HbA1c reduction of at least 0.5% ( $\geq 0.5\%$ ) from baseline with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 2) Assess the proportion of subjects with HbA1c < 7.0% with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 3) Assess the change from baseline in FPG with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 4) Assess the change from baseline in the percent of 24-hour glucose readings obtained from CGM that is in the hypoglycemic range of ≤ 70 mg/dL with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 5) Assess the change from baseline in seated systolic blood pressure with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment among subjects with hypertension at baseline, defined as seated SBP ≥ 140 mmHg and/or seated DBP ≥ 90 mmHg
- 6) Assess the change from baseline in average glucose values measured by 6-point (SMBG) with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 7) Assess the change from baseline in postprandial glucose values measured by 6-point self SMBG with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 8) Assess the change from baseline in postprandial glucose values measured by CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 9) Assess the change from baseline in standard deviation of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 10) Assess the change from baseline to Week 24 in health status, as measured by the Euro Quality of life 5 dimensions 3 levels (EQ-5D-3L) questionnaire, between dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment

11) Assess the changes from baseline to Week 24 in the summary score for treatment satisfaction and scores for perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively, as measured by the Diabetes Treatment Satisfaction Questionnaire status (DTSQs) between the dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment

- 12) Assess the change from baseline to Week 24 in the summary score of fear of hypoglycemia as measured by the Hypoglycemia Fear Survey (HFS-II) Worry Subscale between the dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 13) To explore the relationship between observed and/or model estimated pharmacokinetic measures of exposure (eg, AUCss, Cmax, Cmin) and efficacy and/or safety endpoints by using model-based approaches. This analysis will be provided in a separate report
- 14) Compare the number of non-severe hypoglycemic events per subject in those achieving an HbA1c reduction of  $\geq 0.5\%$  on dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin from baseline to Week 24 visit.

# 1.4 Product Development Background

Dapagliflozin has been designed as a potent and selective inhibitor of the renal sodium-glucose transporter, SGLT-2. Multiple Phase 2 and Phase 3 studies, where dapagliflozin was used as monotherapy or in combination with other oral hypoglycemic agents or insulin in subjects with T2DM, have shown that dapagliflozin is associated with a significant reduction of HbA1c from baseline compared to placebo (0.4-0.56% and 0.54-0.68% for 5 and 10 mg doses, respectively).

Results from the MB102009 and D1690C00006 studies, where dapagliflozin was added in subjects with T2DM receiving high doses of insulin, confirmed that dapagliflozin was effective in lowering HbA1c when combined with insulin in this population (HbA1c reduction of 0.6% relative to placebo).

Overall, dapagliflozin as monotherapy and in combination with other antidiabetic agents (metformin, sulfonylurea, thiazolidinedione, or insulin) was generally safe and well tolerated in subjects with T2DM. In Phase 2/3 studies, the frequency of overall AEs was similar to placebo. Most AEs were mild or moderate in intensity and resolved while continuing treatment. No clinically relevant changes from baseline were seen in either renal function or serum electrolytes in subjects treated with dapagliflozin. The frequency of genital infections and urinary tract infections was higher in subjects treated with dapagliflozin. Most of the genital infections and urinary tract infections were mild-to-moderate and easily treatable.

Besides data obtained from subjects with T2DM, results from MB102072, where dapagliflozin was added to insulin therapy in subjects with T1DM, showed that dapagliflozin 5 mg and 10 mg may improve glycemic control during a 2-week study period while reducing total daily insulin dose. In this pilot study, adverse events, including hypoglycemia and genitourinary infections, were generally balanced across treatment groups.

Additional clinical safety and efficacy information is available in the Investigator Brochure.

#### 1.5 Overall Risk/Benefit Assessment

Dapagliflozin is being developed as a potential new therapy for hyperglycemia in subjects with T1DM. Considering the mechanism of action of dapagliflozin, the design features of this study (ie, the inclusion, exclusion, and discontinuation criteria), and the planned safety procedures, participation in this study presents a minimal risk.

As noted above, dapagliflozin has been effective at lowering glucose and HbA1c in subjects with T2DM, when studied as monotherapy, as well as in combination with insulin or oral antidiabetic medications. In a recently concluded Phase 2a study, the combination therapy of dapagliflozin with insulin was assessed in subjects with T1DM with inadequate glycemic control. In that study, dapagliflozin was found to be well-tolerated. Results from the study also suggested that treatment with dapagliflozin as add-on to insulin may have potential to reduce glucose levels, decrease glycemic variability based on CGM, and reduce total daily insulin dose. Similar results were also reported in an 8-week study in which empagliflozin was added as an adjunct to insulin therapy in subjects with T1DM. <sup>13</sup>

#### **Potential risks**

The potential risks associated with dapagliflozin have been identified based upon the mechanism of action, the preclinical results, and the extensive clinical experience to date, including a study combining it with insulin when used in subjects with T1DM. The benefits and risks associated with the investigational drug and insulin are well established and presented in their approved Investigator Brochure and prescribing information respectively. No study procedure will put subjects at a risk beyond those ordinarily encountered during the performance of routine medical examinations or tests

#### Protection against risks

The present study has been designed with appropriate measures in place to monitor and minimize any of the potential health risks to participating subjects. In order to ensure the safety of all subjects participating in this study, the Sponsor will conduct a real-time review of all safety information from all ongoing clinical dapagliflozin studies as it becomes available. Safety signal detection will include the integration of all available sources of safety information, including clinical study data, AE reports, pre-clinical data, epidemiological studies and literature reports, and post-marketing reports to identify and characterize unrecognized safety risks or changes in those which are currently expected Adverse Drug Reactions. Any information that may affect the benefit-risk profile of dapagliflozin will be immediately communicated to relevant health authorities and appropriate actions will be taken regarding the clinical program as needed.

Given the potential increased risk of hypoglycemia when dapagliflozin is added on to insulin, it is <u>recommended</u> that subjects reduce their daily insulin doses by up to 20% for both basal and bolus insulin after the first dose of study drug on Day 1 following randomization to reduce the risk of hypoglycemia. In some cases it may be necessary to reduce insulin (particularly basal insulin) in advance of study drug administration. During the study, insulin dose may be adjusted


as deemed appropriate to be consistent with good clinical practice according to (SMBG) readings, local guidance and individual circumstances.

Safety will also be monitored by an external Data Monitoring Committee (DMC) with multidisciplinary representation, which will periodically evaluate the incidence of AEs (especially events of hypoglycemia and DKA), laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects. An independent reporting statistician not involved in the conduct of the study will be designated by Bristol-Myers Squibb (BMS) to provide the DMC with essential safety data during the study. The DMC responsibilities, authorities, and procedures will be documented in a DMC charter.

All studies which include dapagliflozin are subject to a carefully designed subject risk management plan. Investigators are also provided guidance on appropriate management of potential risks such as hypoglycemia, urinary tract infections and decreased renal function as mentioned in the plan. In addition, for this trial, investigators are provided guidance on appropriate managements and potentials risks associated with DKA.

### Potential benefits to subjects

As noted above, dapagliflozin added to background insulin therapy was well-tolerated in the Phase 2 study in subjects with T1DM (MB102072) and had a PK profile similar to the healthy and T2DM populations studied previously. Therefore, it is expected that the efficacy and safety profile of dapagliflozin in subjects with T1DM will be similar to that observed in T2DM subjects. Furthermore, because its mechanism is independent of insulin, dapagliflozin provides an opportunity to achieve clinically important glycemic efficacy in subjects with T1DM. In addition, all subjects will continue to receive insulin (dose can be adjusted) as active background therapy.

Subjects are also expected to receive some benefit in the form of increased medical care/attention when participating in study procedures, which includes multiple clinic visits and physical examinations over the 52 week study. Subjects will also receive counseling on diet and exercise. It is commonly observed that even subjects receiving placebo in diabetes studies show some improvement in glycemic control, likely due to their increased compliance to dietary and exercise counseling while they are participating in a clinical study.

### 2 ETHICAL CONSIDERATIONS

### 2.1 Good Clinical Practice

This study will be conducted in accordance with Good Clinical Practice (GCP), as defined by the International Conference on Harmonisation (ICH) and in accordance with the ethical principles underlying European Union Directive 2001/20/EC and the United States Code of Federal Regulations, Title 21, Part 50 (21CFR50).

The study will be conducted in compliance with the protocol. The protocol and any amendments and the subject informed consent form will receive Institutional Review Board/Independent Ethics Committee (IRB/IEC) approval/favorable opinion prior to initiation of the study.


All potential serious breaches must be reported to BMS immediately. A serious breach is defined as a violation of the conditions and principles of GCP in connection with the study or the protocol, which is likely to affect, to a significant degree, the safety or physical or mental integrity of the subjects of the study or the scientific validity of the study.

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

# 2.2 Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, consent form, subject recruitment materials (eg, advertisements), and any other written information to be provided to subjects. The investigator or BMS should also provide the IRB/IEC with a copy of the Investigator Brochure or product labeling information to be provided to subjects and any updates.

The investigator or BMS/AZ should provide the IRB/IEC with reports, updates and other information (eg, expedited safety reports, amendments, and administrative letters) according to regulatory requirements or institution procedures.

#### 2.3 Informed Consent

Investigators must ensure that subjects are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

In situations where consent cannot be given to subjects, their legally acceptable representatives (as per country guidelines) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the subject volunteers to participate.

BMS will provide the investigator with an appropriate (ie, Global or Local) sample informed consent form which will include all elements required by ICH, GCP and applicable regulatory requirements. The sample informed consent form will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

#### Investigators must:

- 1) Provide a copy of the consent form and written information about the study in the language in which the subject is most proficient prior to clinical study participation. The language must be non-technical and easily understood.
- 2) Allow time necessary for subject or subject's legally acceptable representative to inquire about the details of the study.
- 3) Obtain an informed consent signed and personally dated by the subject or the subject's legally acceptable representative and by the person who conducted the informed consent discussion.


4) Obtain the IRB/IEC's written approval/favorable opinion of the written informed consent form and any other information to be provided to the subjects, prior to the beginning of the study, and after any revisions are completed for new information.

- 5) If informed consent is initially given by a subject's legally acceptable representative or legal guardian, and the subject subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the subject.
- 6) Revise the informed consent whenever important new information becomes available that is relevant to the subject's consent. The investigator, or a person designated by the investigator, should fully inform the subject or the subject's legally acceptable representative or legal guardian, of all pertinent aspects of the study and of any new information relevant to the subject's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the subjects' signed ICF and, in the US, the subjects' signed HIPAA Authorization.

The consent form must also include a statement that BMS and regulatory authorities have direct access to subject records.

For minors, according to local legislation, one or both parents or a legally acceptable representative must be informed of the study procedures and must sign the informed consent form approved for the study prior to clinical study participation. The explicit wish of a minor, who is capable of forming an opinion and assessing this information to refuse participation in, or to be withdrawn from, the clinical study at any time should be considered by the investigator.

Minors who are judged to be of an age of reason must also give their written assent.

The rights, safety, and well-being of the study subjects are the most important considerations and should prevail over interests of science and society.

### 3 INVESTIGATIONAL PLAN

### 3.1 Study Design and Duration

This trial is a randomized, double-blinded, three-arm, parallel-group, placebo-controlled, multicenter trial to evaluate the efficacy and safety of dapagliflozin, when added to ongoing insulin therapy, in subjects with T1DM and inadequate glycemic control.

Potential subjects will be assessed for eligibility criteria at the screening visit. Eligible subjects will enter an 8-week lead-in period in order to optimize their diabetes management and assess the variability in blood glucose profiles and frequency of hypoglycemic episodes at baseline. No placebo or study medication will be provided during the lead-in period. On Day 1, subjects who meet all the protocol-specific enrollment and randomization inclusion criteria and meet none of the exclusion criteria will be randomized into one of the three blinded treatment arms (dapagliflozin 5 mg QD, dapagliflozin 10 mg QD, or placebo QD) in a 1:1:1 ratio.


Randomization will be stratified by the following factors to ensure equal representation across all treatment groups:

- Current use of CGM (this refers to an unblinded/personal device already being used, in addition to the blinded CGM device that will be required for participation in the study. Current use of CGM will be categorized as yes vs no)
- Method of insulin administration at baseline (multiple daily injections [MDI] defined as three or more injections per day vs continuous subcutaneous insulin infusion [CSII])
- Week -1 Visit (Baseline) A1C  $\geq$  7.5% and < 9.0% vs  $\geq$  9.0% and  $\leq$  10.5%

Subjects will receive dapagliflozin 5 mg QD, 10 mg QD, or placebo QD for 24 weeks, followed by a 28-week subject and site blinded long-term treatment period. Besides study medications, subjects will be treated with MDI (3 or more injections per day of basal and prandial insulin) or CSII.

It is <u>recommended</u> that subjects reduce their daily insulin dose by up to 20% for both basal and bolus insulin after the first dose of study medication to minimize the risk of hypoglycemia. In some cases it may be necessary to reduce insulin (particularly basal insulin) in advance of study drug administration. It is at the discretion of the investigator to determine the extent to which to reduce the insulin doses. Throughout the study (from the beginning of the lead-in period to the end of the long-term treatment period), insulin dose may be adjusted as deemed appropriate to be consistent with good clinical practice according to SMBG readings, local guidance, and individual circumstances. Subjects will be monitored closely with regard to safety parameters, including vital signs, safety laboratory tests, ECGs, and AEs.

The study design schematic is presented in Figure 3.1-1.


Date: 18-May-2016

930087408 3.0

v3.0

Figure 3.1-1: Study Design Schematic



#### Notes:

- Eligible subjects should have the Day 1 randomization visit within  $56 \pm 5$  days of the Week -8 entry into lead-in period visit
- Subjects will receive the last dose of study medications at the Week 52 Visit and they will have the follow-up visit at Week 56 (30 days after the Week 52 visit)

# 3.2 Post Study Access to Therapy

End of Lead-In Period/Entry into Short-term Treatment Period

At the end of the study, BMS/AZ will not continue to provide BMS supplied study drug to subjects/investigators unless BMS/AZ chooses to extend the study. The investigator should ensure that the subject receives appropriate standard of care to treat the condition under study.

### 3.3 Study Population

For entry into the study, the following criteria MUST be met.

### 3.3.1 Inclusion Criteria

- 1) Signed written Informed Consent
  - a) Subjects or their legally responsible representatives must be willing and able to give signed and dated written informed consent
  - b) Not applicable per Protocol Amendment 03 Subjects from Japan  $\geq$  18 years old and < 20 years old must have assent forms signed and dated by their parents or guardians


v3.0

930087408 3.0

### 2) Target Population

- a) Diagnosis of T1DM. In addition, the following criteria also needs to be met;
  - i) Central laboratory test of C-peptide < 0.7 ng/ml (0.23 nmol/L)
- b) Subject re-enrollment: This study does not permit the re-enrollment of a subject who has discontinued the study as a screen or lead-in failure

Note: Subjects who did not fail any of the screening or lead-in criteria and are not subsequently randomized within the applicable study visit windows (e.g. due to a planned medical procedure, vacation plans, or employment commitments) may rescreen after discussion and approval by the Sponsor.

- 3) Insulin use for at least 12 months prior to screening per subject report or medical records and
  - a) Method of insulin administration (MDI or CSII) must have been unchanged for at least 3 months prior to the screening visit per subject reported or medical records. Subjects must be taking a total insulin dose of  $\geq 0.3$  U/kg/day for at least 3 months prior to the screening visit
  - b) If on MDI insulin administration, subject must be taking  $\geq 3$  injections per day
- 4) HbA1c eligibility criteria include:
  - a) Screening visit: Central laboratory HbA1c  $\geq 7.7\%$  and  $\leq 11.0\%$

Note: a one-time repeat HbA1C is allowed for subjects in screening if their initial result is within  $\pm$  0.2% of the cut off values

b) Week -1 Visit: Central laboratory HbA1c  $\geq 7.5$  % and  $\leq 10.5$ %

Note: a one-time repeat HbA1C is allowed for subjects in lead-in if their test result is within  $\pm 0.2\%$  of the cut off values

To ensure adequate time is given to complete the repeat Week -1 A1C, a 7 day window (added to the current lead-in period window of 56 + 5 days) will be allowed

- 5) Body mass index (BMI)  $\geq 18.5 \text{ kg/m}^2$
- 6) Age and reproductive status
  - a) Men and women, ages 18 to 75 years, inclusive
  - b) Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product
  - c) Women must not be breastfeeding
  - d) WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with dapagliflozin plus 4 days (> 5 half-lives of dapagliflozin) plus 30 days (duration of ovulatory cycle) for a total of 34 days post-treatment completion
  - e) Males who are sexually active with WOCBP must agree to the following instructions for the duration of treatment with dapagliflozin plus 4 days (>5 half-lives of dapagliflozin) plus 90 days (duration of sperm turnover) for a total of 94 days post-treatment completion

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.

At a minimum, subjects must agree to the use of one method of highly effective contraception listed below:

- Male condoms with spermicide<sup>14</sup>
- Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena® by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
- Non-hormonal IUDs, such as ParaGard®
- Tubal ligation (not considered surgically sterile, see section 3.3.3)
- Vasectomy
- Complete abstinence\*

\*Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, females must still undergo pregnancy testing as described in this section.

### 3.3.2 Exclusion Criteria

### 1) Target Disease Exceptions

a) History of T2DM

Note: subjects with a previous misdiagnosis of T2DM in their medical history must have one of the following in order to be eligible for this trial:

- Positive autoantibodies for GAD65, phosphatase IA-2/IA2β, or zinc transporter 8 (ZnT8) (eg, autoimmune diabetes)
- Fasting c-peptide value below the lower limit of detection performed by the Central Laboratory
- b) History of maturity-onset diabetes of the young (MODY)
- c) Pancreatic surgery, chronic pancreatitis, or other pancreatic disorders that could result in decreased β-cell capacity (eg. pancreatogenous diabetes)
- d) Previous use of dapagliflozin and/or any other SGLT-2 inhibitors


v3.0 930087408 3.0

e) Use of insulin-sensitizing agents, such as metformin and/or thiazolidinediones, within 2 months prior to the screening visit

- f) Use of any GLP-1 receptor agonist within the following timeframe prior to the screening visit:
  - 1 month for once or twice daily administration (eg, liraglutide)
  - 2 months for once weekly administration
- g) Use of any non-insulin antihyperglycemic agent within 1 month prior to the screening visit
- h) History of DKA requiring medical intervention (eg, emergency room visit and/or hospitalization) within 1 month prior to the screening visit
- i) History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to the screening visit
- j) Frequent episodes of severe hypoglycemia as defined by more than one episode requiring medical assistance, emergency care (paramedics or emergency room care), and/or glucagon therapy administered by a third-party individual within 1 month prior to the screening visit
- k) Symptoms of poorly controlled diabetes that would preclude participation in this trial including, but not limited to, marked polyuria and polydipsia with greater than 10% weight loss during the 3 months prior to the screening visit, or other signs and symptoms of poor glycemic control
- 1) History of Addison's disease or chronic adrenal insufficiency
- m) History of diabetes insipidus

### 2) Medical History and Concurrent Diseases

- a) Any of the following cardiovascular (CV)/vascular disease within 6 months of the screening visit:
  - 1. Myocardial infarction
  - 2. Cardiac surgery or revascularization (coronary artery bypass surgery [CABG]/percutaneous transluminal coronary angioplasty [PTCA])
  - 3. Unstable angina
  - 4. Unstable congestive heart failure (CHF)
  - 5. New York Heart Association (NYHA) CHF Class III or IV
  - 6. Transient ischemic attack (TIA) or significant cerebrovascular disease
  - 7. Unstable or previously undiagnosed arrhythmia
- b) Renal disease:
  - 1. History of unstable or rapidly progressing renal disease
  - 2. Conditions of congenital renal glucosuria
  - 3. Renal allograft
- c) Hepatic diseases:
  - 1. Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency


- d) Hematological and oncological disease/conditions:
  - 1. History of hemoglobinopathy, with the exception of sickle cell trait (SA) or thalassemia minor; or chronic or recurrent hemolysis
  - 2. Known immunocompromised status, including but not limited to, individuals who have undergone organ transplantation or who are positive for the human immunodeficiency virus
  - 3. Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 8 weeks prior to the screening visit
  - 4. Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma)
  - 5. History of bladder cancer
  - 6. History of radiation therapy to the lower abdomen or pelvis at any time

### 3) Physical and Laboratory Test Findings

- a) Aspartate aminotransferase (AST) > 3x upper limit of normal (ULN)
- b) Alanine aminotransferase (ALT) > 3x ULN
- c) Serum total bilirubin (TB) > 2x ULN unless exclusively caused by Gilbert's Syndrome
- d) Calculated creatinine clearance (CrCl) < 60 mL/min as estimated by the Cockcroft-Gault formula, using laboratory measurements of serum creatinine collected at the screening visit [Creatinine clearance = [[140 age(yr)]\*weight(kg)/[72\*serum Cr(mg/dl)] (multiply by 0.85 for women)]
- e) Hemoglobin  $\leq 11.0 \text{ g/dL}$  (110 g/L) for men; hemoglobin  $\leq 10.0 \text{ g/dL}$  (100 g/L) for women
- f) Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody
- g) Abnormal Free T4

NOTE: abnormal TSH value at enrollment will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded. A one-time retest may be allowed, as determined by the investigator, after a minimum of 6 weeks following the adjustment of thyroid hormone replacement therapy in subjects who have had a prior diagnosis of a thyroid disorder and who are currently receiving thyroid replacement therapy. Such cases should be discussed with the Sponsor prior to re-testing. The subject must have all enrollment procedures and laboratory assessments performed as part of this re-test, and all of these must meet enrollment eligibility criteria. The subject's number will however remain the same as initially assigned.

#### 4) Allergies and Adverse Drug Reaction

a) Allergies or contraindication to the contents of dapagliflozin tablets or insulin

### 5) Sex and Reproductive Status

a) Women who are pregnant

### 6) Other Exclusion Criteria

a) Prisoners or subjects who are involuntarily incarcerated


v3.0 930087408 3.0

b) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

- c) Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program
- d) History of bariatric surgery or lap-band procedure within 12 months prior to screening
- e) Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid (including local injections such as intramuscular or intra-articular, etc.) taken for > 4 weeks within 3 months prior to the Day 1 visit
  - NOTE: Topical (including drops) or inhaled corticosteroids are allowed
- f) Any unstable endocrine, psychiatric or rheumatic disorders as judged by the investigator
- g) Volume-depleted subjects. Subjects at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics who cannot carefully monitor their volume status should be excluded from the study
- h) Subject who, in the judgment of the investigator, is found to be unlikely to comply with the protocol, or is unable to correctly administer subcutaneous insulin injections and/or manage their insulin pump, or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data (including during the lead-in period)
- i) Subject with any condition which, in the judgment of the investigator, may render the subject unable to complete the study or which may pose a significant risk to the subject
- j) Subject is currently abusing alcohol or other drugs or has done so within the last 6 months prior to the Day 1 visit
- k) Subject is a participating investigator, study coordinator, employee of an investigator or immediate family member of any of the aforementioned
- 1) Employee of BMS, AstraZeneca (AZ), or their relatives
- m) Administration of any other investigational drug within 30 days of the screening visit
- n) No clinical conditions or clinically significant abnormalities in any laboratory value(s) collected after screening and prior to randomization which, in the investigator's judgment, should preclude entry into the treatment period

Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.

### 3.3.3 Women of Childbearing Potential

A woman of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In additional, women under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40mIU/mL to confirm menopause.\*

\*Females treated with hormone replacement therapy (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and investigators should use their judgment in checking serum FSH levels. If the washout period exceeds 4 weeks, the subject must have all enrollment procedures and laboratory assessments repeated and all of these must meet enrollment eligibility criteria. The subject's number will however remain the same as initially assigned. If the serum FSH level is > 40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal:

- 1 week minimum for vaginal hormonal products, (rings, creams, gels)
- 4 week minimum for transdermal products
- 8 week minimum for oral products

Other parenteral products may require washout periods as long as 6 months.

### 3.4 Concomitant Treatments

### 3.4.1 Prohibited and/or Restricted Treatments

Once enrolled, subjects may not receive any of the following for the duration of the screening (qualification period), lead-in, double-blinded short-term and subject and site blinded long-term treatment periods:

- Antihyperglycemic medication (other than protocol required medication)
- Weight loss medication
- Newly initiated treatment with any systemic corticosteroid therapy (including local injections such as intramuscular or intra-articular,etc.) that will involve ≥ 5 days of therapy is not permitted (inhaled and topical, including drops, are allowed). The Medical Monitor should be consulted prior to beginning therapy with corticosteroids for subjects who require systemic corticosteroid treatment
- Acetaminophen (paracetamol) containing medications (such as Tylenol®) while using the CGM device and 24 hours prior to insertion

### 3.4.2 Other Restrictions and Precautions

- Subjects must comply with their prescribed dosing regimen to preserve study integrity and ensure subject safety
- Subjects should be cautioned that any new prescription medication or over-the-counter or herbal/nutritional therapies should be discussed thoroughly with the investigator, as concomitant use could result in alterations to their glycemic control and may place them at risk for significant hypoglycemic episodes


Date: 18-May-2016

• Subjects must make every attempt to adhere to the diet and exercise counseling (see Section 5.9.3) and to the study flow chart/time and event schedule (see Section 5.1)

• Women of child-bearing potential must immediately contact the investigator if they suspect they might be pregnant and if they have changed or plan to change their birth control method (see Section 6.4)

### 3.5 Discontinuation of Subjects from Treatment

Subjects MUST discontinue investigational product (and non-investigational product at the discretion of the investigator) for any of the following reasons:

- Subject's request to stop study treatment
- Withdrawal of informed consent (subject's decision to withdraw for any reason)
- Any clinical adverse event (AE), laboratory abnormality or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject
- Termination of the study by Bristol-Myers Squibb (BMS)/AstraZeneca (AZ)
- Loss of ability to freely provide consent through imprisonment or involuntarily incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness
- Unblinding a subject for any reason (emergency or non-emergency)
- Pregnancy
- Creatinine clearance < 30 mL/min
  - If at any time the subject's CrCl (based on Cockroft-Gault) falls below 30 mL/min calculated at the <u>central</u> laboratory and confirmed at a repeated central laboratory measurement (to be obtained within 4 days, whenever possible), the subject should be discontinued from study medication.
  - If at any time the subject's CrCl (based on Cockroft-Gault) falls below 30 mL/min calculated at <u>local</u> laboratory, a <u>central</u> laboratory CrCl should be obtained promptly. If the CrCl is confirmed by the central laboratory and persists at a repeated central laboratory measurement (to be obtained within 4 days, whenever possible), the subject should be discontinued from study medication.
- Subjects experience at least one protocol-defined hypoglycemia episode that leads to a loss of consciousness and/or seizure as determined by the investigator (see Section 3.5.1)
- Change of insulin administration method (eg, switch from MDI to CSII or vice versa)

  Note: Subjects are not allowed to change their insulin administration methods (MDI or CSII) throughout the study. Under certain situations (eg, the replacement of an insulin pump), the subjects who are on CSII may be on temporary use of MDI. They should restart CSII administration as early as feasible. The period of time when a subject is on temporary use of MDI should not be more than 2 weeks


Date: 18-May-2016

• Subjects with a central laboratory ALT and/or AST > 3x ULN will be scheduled for a follow-up visit within 3 days following the receipt of the result (see Appendix 3 for further guidance). Subjects should be discontinued from study if the initial and repeat laboratory tests meet any of the following criteria:

- ALT and/or AST are > 3x ULN and total bilirubin (TB) > 2x ULN
- ALT and/or AST are > 5x ULN for ≥ 14 consecutive days, at any time after initial confirmatory results
- ALT and/or AST are > 10x ULN

All subjects who discontinue study drug should comply with protocol specified follow-up procedures as outlined in Section 5 with the exception of the study drug and PK procedures. The only exception to this requirement is when a subject withdraws consent for all study procedures including post-treatment study follow-up or loses the ability to consent freely (ie, is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or physical illness).

If study drug is discontinued prior to the subject's completion of the study, the reason for the discontinuation must be documented in the subject's medical records and entered on the appropriate case report form (CRF) page.

# 3.5.1 Discontinuation Guidelines due to Protocol-Defined Hypoglycemia Episode or Recurrent Hypoglycemia Episodes

Subjects should not be discontinued from any treatment phase based on single episodes of hypoglycemia or symptoms of hypoglycemia unless clinically indicated (see the criteria below). The assessment of a single capillary glucose measurement (eg, fingerstick) or central laboratory glucose value should not be the sole assessment used to determine subject discontinuation due to hypoglycemia.

Subjects should be discontinued from study drug if they meet any of the following criteria:

- At least one hypoglycemia episode that leads to loss of consciousness and/or seizure
- Severe/recurrent hypoglycemia episodes where the possibility of down-titration of contributing concomitant medication(s) (other than double-blind study medication), and/or contributing factors (eg, excessive physical activity) have been evaluated and corrected.

NOTE: Dose titration of double-blind study drug is not permitted at any time during the short-term and long-term treatment period.

Section 5.3.2.2 provides additional guidance on management and reporting of hypoglycemia.

### 3.6 Post Study Drug Study Follow up

In this study, safety is a key endpoint of the study. Post treatment study follow-up is of critical importance and is essential to preserving subject safety and the integrity of the study. Subjects who discontinue study drug must continue to be followed for collection of outcomes and/or


survival follow-up data as required and in line with Section 5 until death or the conclusion of the study.

Therefore as such, all subjects who discontinue investigational product in the 24-week double-blinded short-term treatment period or in the subject- and site-blinded long-term treatment period should be asked to continue study participation for each scheduled visit for the remaining length of the study and complete all procedures as outlined in the Section 5 study flowchart, with the exception of study drug management and PK sampling. If continued study participation according to the protocol schedule is not possible, the investigator should contact the subject to discuss alternatives (eg, return to the clinic 30 days after discontinuation of study drug to perform the Week 56 visit post-treatment follow-up procedures as outlined in the Section 5 study flowchart or be contacted by telephone 30 days after discontinuation of study drug to evaluate the following safety assessments: AEs, hypoglycemia events, and DKA episodes. Please note that after the discontinuation of study drug, management of a subject's diabetes would be under the care and direction of the investigator and/or subject's healthcare providers.

The only exception to any of these follow-up methods are when a subject withdraws consent for all study procedures, including post-treatment study follow-up, or loses the ability to consent freely (ie, is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or physical illness).

Please utilize the Off-Treatment Short-Term and Off-Treatment Long-Term eCRF pages for this data completion.

### 3.6.1 Withdrawal of Consent

Subjects who request to discontinue study drug will remain in the study and must continue to be followed for protocol specified follow-up procedures. The only exception to this is when a subject specifically withdraws consent for any further contact with him/her or persons previously authorized by the subject to provide this information withdraws consent. Subjects should notify the investigator of the decision to withdraw consent from future follow-up **in writing**, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is from further treatment with study drug only or also from study procedures and/or post treatment study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the subject is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

### 3.6.2 Lost to Follow-Up

All reasonable efforts must be made to locate subjects to determine and report their ongoing status. This includes follow-up with persons authorized by the subject as noted above. Lost to follow-up is defined as the inability to reach the subject after a minimum of three documented phone calls, faxes, or emails, as well as lack of response by subject to one registered mail letter. All attempts should be documented in the subject's medical records. If it is determined that the subject has died, the site will use permissible local methods to obtain the date and cause of death.


If the investigator's use of a third-party representative to assist in the follow-up portion of the study has been included in the subject's informed consent, then the investigator may use a Sponsor-retained third-party representative to assist site staff with obtaining subject's contact information or other public vital status data necessary to complete the follow-up portion of the study. The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information. If after all attempts, the subject remains lost to follow-up, then the last known alive date as determined by the investigator should be reported and documented in the subject's medical records.

### 4 STUDY DRUG

Study drugs include both non-investigational medicinal products (NIMP) and investigational medicinal products (IMP) and can consist of the following:

- All products, active or placebo, being tested or used as a comparator in a clinical trial.
- Other drugs administered as part of the study that are critical to claims of efficacy (eg, background therapy, rescue medications)


Date: 18-May-2016 41

930087408 3.0

v3.0

| Table 4-1: | Study Drug for I and Site Blinded | MB102230 - Product Descripti<br>Long-term Treatment Period | luct Description -<br>rtment Period | Double-blinded Short-ter | Study Drug for MB102230 - Product Description - Double-blinded Short-term Treatment and Subject and Site Blinded Long-term Treatment Period |
|---|---|---|---|---|---|
| Product Description /<br>Class and Dosage Form | Potency | IP/Non-IMP | Blinded or Open<br>Label | Packaging/ Appearance | Storage Conditions (per label) |
| Dapagliflozin film-coated tablet | 5 mg | IP | Blinded | Green, plain, diamond<br>shaped, film coated tablet<br>(reference footnote below for<br>packaging) | Store at 15-25 degrees Celsius (59-77 degrees Fahrenheit); store in tightly closed container |
| Placebo for dapagliflozin<br>film- coated tablets | gm 0 | IP | Blinded | Green, plain, diamond<br>shaped, film coated tablet<br>(reference footnote below for<br>packaging) | Store at 15-25 degrees Celsius (59-77 degrees Fahrenheit); store in tightly closed container |
| Insulin | Varies | Non-IMP | Open Label | Based on manufactured product specifications | Based on manufactured product specifications |

Blinded dapagliflozin 10 mg kit contains 2 bottles of dapagliflozin 5 mg film-coated tablets (35 count) and 1 bottle of dapagliflozin film-coated tablets (35 count)

Blinded placebo kit contains 2 bottles of placebo for dapagliflozin film-coated tablets (35 count)

### 4.1 Investigational Product

An investigational product, also known as investigational medicinal product (IMP) in some regions, is defined as a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently than the authorized form, or used for an unauthorized indication, or when used to gain further information about the authorized form.

The investigational product should be stored in a secure area according to local regulations. It is the responsibility of the investigator to ensure that investigational product is only dispensed to study subjects. The investigational product must be dispensed only from official study sites by authorized personnel according to local regulations.

In this protocol, investigational products are: (also described in Table 4-1) dapagliflozin 5 mg and matching placebo tablets; insulin will not be provided by the Sponsor since it is part of the subject's standard of care.

- Blinded dapagliflozin 5 mg and 10 mg dose administered orally for the 24-week double-blinded short-term treatment period, and the 28-week subject- and site-blinded long-term treatment period of the study
- Matching placebo dose administered orally for the 24-week double-blinded short-term treatment period, and the 28-week subject- and site-blinded long-term treatment period of the study.

### 4.2 Non-investigational Product

Other medications used as support or escape medication for preventive, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as non-investigational products.

In this protocol, non-investigational product is: insulin.

### 4.3 Storage and Dispensing

The product storage manager should ensure that the study drug is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study drug arise, the study drug should not be dispensed and contact BMS immediately.

Study drug not supplied by BMS will be stored in accordance with the package insert.

Investigational product documentation (whether supplied by BMS or not) must be maintained that includes all processes required to ensure drug is accurately administered. This includes documentation of drug storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg., required diluents, administration sets).

### 4.4 Method of Assigning Subject Identification

JUI


CCI

# 4.4.1 Subjects entering the 24-week double-blinded short-term treatment period

Following completion of the lead-in period, subjects who meet the criteria will be randomly assigned by the IVRS at the Day 1 (randomization) visit, to one of the following 3 double-blind treatment arms in a 1:1:1 ratio using a centralized blocked randomization schedule:

- 1) Blinded dapagliflozin 5 mg
- 2) Blinded dapagliflozin 10 mg
- 3) Blinded placebo

Randomization will be stratified by:

- Current use of CGM (this refers to an unblinded/personal device already being used, in addition to the blinded CGM device that will be required for participation in the study. Current use of CGM will be categorized as yes vs no)
- Method of insulin administration at baseline (multiple daily injections [MDI] three or more injections per day vs continuous subcutaneous insulin infusion [CSII])
- Week -1 Visit (Baseline) HbA1c  $\geq 7.5\%$  and < 9.0% vs  $\geq 9.0\%$  and  $\leq 10.5\%$

Randomization schedules for both subject treatment and kits will be generated and kept by BMS.

# 4.4.2 Subjects entering the 28-week long-term subject and site blinded treatment period

Following completion of the 24-week double-blinded treatment period, subjects eligible for the long-term subject- and site-blinded treatment period will be continue in their same randomization assignment based on their original randomization grouping. Subjects that were assigned to the blinded dapagliflozin 5 mg arm will continue to receive blinded dapagliflozin 5 mg. Subjects that were assigned to the blinded dapagliflozin 10 mg arm will continue to receive blinded dapagliflozin 10 mg and subjects that were assigned to the blinded placebo arm will continue to receive blinded placebo. At all study visits when study drug is dispensed, each subject will be assigned a kit number by the IVRS. Kit numbers will be assigned non-sequentially and will correspond to the numbers printed on the containers and bottles containing study drug, and will be recorded on the appropriate eCRF. The IVRS will be available 24 hours per day, 7 days a week. Randomization schedules for both subject treatment and kits will be generated and kept by BMS.

### 4.5 Selection and Timing of Dose for Each Subject

Dapagliflozin 5 mg, 10 mg, or placebo will be administered orally, once daily for the 24-week double-blinded short-term treatment period and the 28-week subject- and site-blinded long-term treatment period.


### 4.6 Blinding/Unblinding

Blinding of treatment assignment is critical to the integrity of this clinical study. However, in the event of a medical emergency or pregnancy in an individual subject in which knowledge of the investigational product is critical to the subject's management, the blind for that subject may be broken by the investigator. The subject's safety takes priority over any other considerations in determining if a treatment assignment should be unblinded.

Before breaking the blind of an individual subject's treatment, the investigator should determine that the unblinded information is necessary (ie, that it will alter the subject's immediate management). In many cases, particularly when the emergency is clearly not related to the investigational product, the problem may be properly managed by assuming that the subject is receiving active product. It is highly desirable that the decision to unblind treatment assignment be discussed with the Medical Monitor, but the investigator always has ultimate authority for the decision to unblind. The investigator should only call in for emergency unblinding AFTER the decision to discontinue the subject has been made.

For this study, the method of unblinding for emergency purposes is the IVRS.

For information on how to unblind in case of an emergency, consult the IVRS manual.

In cases of accidental unblinding, contact the Medical Monitor and ensure every attempt is made to preserve the blind.

Any request to unblind a subject for non-emergency purposes should be discussed with the Medical Monitor.

### 4.7 Treatment Compliance

Each time study medication is dispensed, compliance will be reinforced. When study medication is returned, compliance will be assessed based upon the subject's interview and a count of the tablets returned. Compliance should be between  $\geq 80\%$  and  $\leq 120\%$ . The investigator (or designee) will record the amounts of study medication dispensed and returned at each visit, as well as document the reasons for non-compliance in the source document. The dates of all study medication dosing, including interruptions, missed doses or overdose, must be recorded on the eCRF. If the subject is not  $\geq 80\%$  compliant, the period of non compliance should be noted as a protocol deviation and the Sponsor should be notified. The subject should be re-educated regarding treatment compliance and/or recording dose.

### 4.8 Destruction and Return of Study Drug

### 4.8.1 Destruction of Study Drug

For this study, study drugs (those supplied by BMS or sourced by the investigator) such as partially used study drug containers, vials and syringes may be destroyed on site.

Any unused study drugs can only be destroyed after being inspected and reconciled by the responsible BMS Study Monitor unless study drug containers must be immediately destroyed as required for safety, or to meet local regulations (eg, cytotoxics or biologics).


On-site destruction is allowed provided the following minimal standards are met:

- On-site disposal practices must not expose humans to risks from the drug
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's standard operating procedures (SOPs) and a copy provided to BMS upon request
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing of the containers.
   The method of disposal (ie, incinerator, licensed sanitary landfill, or licensed waste disposal vendor) must be documented
- Accountability and disposal records are complete, up-to-date, and available for the Monitor to review throughout the clinical trial period

If conditions for destruction cannot be met the responsible BMS/Contract Research Organization (CRO) Study Monitor will make arrangements for return of study drug.

It is the investigator's responsibility to arrange for disposal of all empty and partially full containers, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

### 4.9 Return of Study Drug

If study drug will not be destroyed upon completion or termination of the study, all unused and/or partially used study drug that was supplied by BMS must be returned to BMS. The return of study drug will be arranged by the responsible BMS/CRO Study Monitor.

It is the investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

### 4.10 Retained Samples for Bioavailability / Bioequivalence

Not applicable.


# STUDY ASSESSMENTS AND PROCEDURES

# 5.1 Flow Chart/Time and Events Schedule

| Table 5.1-1: Flow | Flow chart for Protocol | <b>MB102230</b> | Protocol MB102230 - Qualification and Lead-in Period | tion and Le | ad-in Peri | po |
|---|---|---|---|---|---|---|
| Procedure | Qualification Period | | Lead-in Period (8 Weeks) | od (8 Weeks) | | Notes |
| | Screening Visit | Week -8 <sup>b</sup> | Week-4 <sup>b,c</sup> | Week -2 b | Week -1 <sup>d</sup> | |
| Eligibility Assessments | | | | | | |
| Subject reports to site | × | X | X | X | × | |
| Obtain informed consent | X | | | | | |
| Review inclusion/exclusion criteria | X | | | | × | |
| Review medical history | X | | | | | |
| General Procedures | | | | | | |
| Complete physical exam | × | | | | | Includes general appearance, head, eyes, ears, nose, throat, neck, cardiovascular, lungs, abdomen, lymph nodes, extremities, neurological, skin, and musculoskeletal. |
| Brief physical exam | | X | | | × | Includes cardiovascular, lungs, abdomen, and extremities, and any organ systems pertinent to the subject's signs, symptoms, or AEs |
| Body weight | X | X | | | × | |
| Height | × | | | | | |
| Body mass index (BMI) | X | | | | | |
| Electrocardiogram (ECG) | X | | | | | |
| Blood pressure and heart rate | X | X | | | X | 3 replicate measurements obtained at least 1 minute apart |
| Review concomitant medications/procedures | X | × | × | × | × | |

930087408

v3.0

| Table 5.1-1: Flow | Flow chart for Protocol | MB102230 | Protocol MB102230 - Qualification and Lead-in Period | tion and Le | ad-in Peri | po |
|---|---|---|---|---|---|---|
| Procedure | Qualification Period | | Lead-in Period (8 Weeks) | od (8 Weeks) | | Notes |
| | Screening Visit | Week-8 <sup>b</sup> | Week-4 <sup>b,c</sup> | Week -2 b | Week -1 <sup>d</sup> | |
| Contact IVR system | X | X | | | | |
| Provide dietary and exercise counseling | | X | X | × | X | |
| Dispense subject diaries and provide instructions | | X | X | × | X | |
| Review subject diaries | | | X | × | X | |
| Adjust insulin dose (as needed) | | × | X | × | X | |
| Dispense glucose and ketone meter and strips and provide training | | × | | | | |
| Dispense glucose and ketone strips | | | X | | | |
| Insert/calibrate CGM | | | | Xe | | If a lead-in subject fails lead-in prior to the Day 1 visit, the CGM will not be required to be completed between the week-2 visit and the Day 1 visit (Please refer to Section 5.9.4.3) |
| Replace CGM sensor,<br>download data to review<br>compliance, and provide<br>training | | | | | Xe | |
| Record Meals for 7 days - Second week of CGM. | | | | | Xe | If a lead-in subject fails lead-in prior to the Day I visit, the CGM will not be required to be completed between the week-2 visit and the Day I visit (Please refer to Section 5.9.4.3) |
| 6-point SMBG profiles | | | X | | | If a lead-in subject fails prior to the Day 1 visit, the 6-point SMBG profile will not be required between the week -1 visit and the |

v3.0 930087408

| Table 5.1-1: Flow | Flow chart for Protocol | <b>VIB102230</b> | Protocol MB102230 - Qualification and Lead-in Period | tion and Le | ad-in Peri | po |
|---|---|---|---|---|---|---|
| Procedure | Qualification Period | | Lead-in Period (8 Weeks) | d (8 Weeks) | | Notes |
| | Screening Visit | Week -8 <sup>b</sup> | Week-4 <sup>b,c</sup> | Week -2 b | Week -1 <sup>d</sup> | |
| | | | | | | Day 1 visit |
| | | | | | | Please refer to Section 5.9.4.2 in protocol |
| Safety Assessments | | | | | | |
| Assess AEs | | X | X | × | X | |
| Assess hypoglycemia episodes | | X | X | X | X | |
| Assess DKA | | X | X | X | X | |
| Laboratory Assessments | | | | | | |
| Blood standard safety<br>laboratory panel | X | | | | | |
| Urine standard safety panel (dipstick) | X | | | X | | |
| Pregnancy test (serum) WOCBP only | X | | | | | |
| Pregnancy test (urine) WOCBP only | | $X^g$ | $g^X$ | | | |
| Spot urine for glucose, albumin and creatinine quantification and determination of glucose: creatinine and albumin:creatinine ratios | × | | | | | |
| Fasting plasma glucose | X | | | | | |
| C-peptide | X | | | | | |
| HbA1c | X | | | | X | |
| Hepatitis screen panel | × | | | | | |
| TSH | X | | | | | |

Clinical Protocol

BMS-512148

| Table 5.1-1: Flov | How chart for Protocol | MB102230 | Protocol MB102230 - Qualification and Lead-in Period | tion and Le | ad-in Peri | po | 1-in Period |
|---|---|---|---|---|---|---|---|
| Procedure | Qualification Period | | Lead-in Period (8 Weeks) | d (8 Weeks) | | Notes | Notes |
| | Screening Visit | Week -8 <sup>b</sup> | Week-8 Week-4 <sup>b,c</sup> Week-2 <sup>b</sup> Week-1 | Week-2 b | Week -1 <sup>d</sup> | | Veek -1 <sup>d</sup> |
| Fasting serum lipids | X | | | | | | |

Screening visit may consist of 2 days. Second day is to collect lab work. The length of the Qualification period is ≤ 28 days.

Week -8 visit needs to be within 28 days of screening visit. Week -4 visit and Week -2 visit may be scheduled ± 3 days to allow flexibility of scheduling.

pregnancy kit and new week -4 visit diary should be given to the subject at the week -8 visit as well as additional glucose and ketone strips, if needed. Copies of completed diaries must be sent (scan, photo, fax) into the site prior to the phone visit so discussions can occur between the subject and site personnel about Optional Phone Visit - Week -4 visit can be done as a phone visit to allow flexibility for the subject in visit scheduling. If a phone visit is done, the home the data captured in the diaries.

Week -1 visit should be scheduled at least 7 days but not longer than 10 days after Week -2 visit to accommodate for CGM data collection.

If a lead-in subject fails lead-in prior to the Day 1 visit, the CGM and Meal Recording will not be required to be completed

These safety assessments; review of AEs, hypoglycemia events, and DKA episodes to be performed throughout the study according to the visit schedule as noted via "X"

g If an optional phone visit is planned for week -4, the home pregnancy kit should be given to the subject at the week -8 visit

930087408

| | | | 1 | | | | | |
|---|---|---|---|---|---|---|---|---|
| þ | Notes | | | | | | | Includes cardiovascular, lungs, abdomen, and extremities, and any organ systems pertinent to the subject's signs, symptoms, or AEs |
| t Perio | | Week 24/Early<br>Term Visit <sup>g</sup> | | X | | | | |
| eatmen | | Week 22 <sup>c, e</sup> | | × | | | | |
| rm Tre | | Week 18 <sup>c</sup> | | X | | | | |
| nort-te | riod | Week 12 <sup>f</sup> | | × | | | | × |
| lded Sl | ment Pe | Week 10 <sup>c,e</sup> | | X | | | | |
| ole-blir | n Treati | Week 8 <sup>c</sup> | | X | | | | |
| k Douk | ort-teri | Week 4 <sup>c</sup> | | X | | | | |
| 24-wee | inded Sl | Week 2 <sup>c,d</sup> | | X | | | | |
| 102230 - 2 | 24-week Double-blinded Short-term Treatment Period | Day 10<br>(Phone Visit) <sup>b</sup> | | | | | | |
| ol MB | 24-week | Week 1 <sup>b</sup> | | X | | | | X |
| Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | | Day 4<br>(Phone Visit) <sup>b</sup> | | | | | | |
| chart fo | | Day 2<br>(Phone Visit) | | | | | | |
| Flow | | Day 1 <sup>a</sup> | | X | X | X | | |
| Table 5.1-2: | Procedure | | Eligibility<br>Assessments | Subject reports to site | Review inclusion/exclusion criteria | Review medical history | General Procedures | Brief physical exam |

| Table 5.1-2: | Flow | chart fo | Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | ol MB1 | 02230 - 2 | 24-weel | k Doub | de-blin | ded Sh | ort-ter | m Tre | atment | t Perio | þ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | 7 | 24-week | 24-week Double-blinded Short-term Treatment Period | inded Sh | ort-tern | n Treatn | nent Per | iod | | | | Notes |
| | Day 1 <sup>a</sup> | Day 2<br>(Phone Visit) | Day 4<br>(Phone Visit) <sup>b</sup> | Week 1 <sup>b</sup> | Day 10<br>(Phone Visit) <sup>b</sup> | Week 2 <sup>c,d</sup> | Week 4 <sup>c</sup> | Week 8 <sup>c</sup> | Week 10 <sup>c,e</sup> | Week 12 <sup>f</sup> | Week 18 <sup>c</sup> | Week 22 <sup>c, e</sup> | Week 24/Early<br>Term Visit <sup>g</sup> | |
| Complete physical exam | × | | | | | | | | | | | | × | Includes general appearance, head, eyes, ears, nose, throat, neck, cardiovascular, lungs, abdomen, lymph nodes, extremities, neurological, skin, and musculoskeletal. |
| Body weight | X | | | X | | X | X | X | | X | X | | X | |
| Blood pressure and heart rate | × | | | X | | × | X | X | | × | X | | X | 3 replicate<br>measurements<br>obtained at least<br>1 minute apart |
| ECG | X | | | | | | | | | | | | X | |
| Review concomitant medications/procedures | X | X | X | X | X | X | X | X | X | X | X | X | X | |

| | | | ٠ | | |
|---|---|---|---|---|---|
| þ | Notes | | At Week 10 & 22. If subject is an early termination, then CGM is not required. If week 10 and week 22 are optional phone visits, please refer to footnote e below and Section 5.9.4.3 CGM. | At Week12 & 24. CGM Data Collection not needed if at Week 10/22 visit CGM insertion was not completed Please refer to Section 5.9.4.3 | Please refer to<br>Section 5.9.4.3 |
| t Perio | | Week 24/Early<br>Term Visit <sup>g</sup> | | Х <sub>Р</sub> | Xh |
| atmen | | Week 22 <sup>c, e</sup> | X <sub>P</sub> | | |
| rm Tre | | Week 18 <sup>c</sup> | | | |
| nort-te | riod | Week 12 <sup>f</sup> | | ×p | X |
| nded Sl | ment Pe | Week 10 <sup>c,e</sup> | × | | |
| ole-blir | m Treat | Week 8 c | | | |
| k Doul | hort-teri | Week 4 <sup>c</sup> | | | |
| 24-wee | inded Sl | Week 2 <sup>c,d</sup> | | | |
| 102230 - 3 | 24-week Double-blinded Short-term Treatment Period | Day 10<br>(Phone Visit) <sup>b</sup> | | | |
| ol MB1 | 24-week | Week 1 <sup>b</sup> | | | |
| Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | | Day 4<br>(Phone Visit) <sup>b</sup> | | | |
| chart fo | | Day 2<br>(Phone Visit) | | | |
| Flow | | Day 1 <sup>a</sup> | | × | |
| Table 5.1-2: | Procedure | | Insert/calibrate CGM | CGM Data collection,<br>data upload, and<br>review | Record Meals for 7 days - Second week of CGM. |

| Table 5.1-2: | Flow | chart fo | Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | ol MB1 | 02230 - 2 | 24-wee] | k Doub | le-blin | ded Sh | ort-ter | m Tre | atmeni | t Perio | p |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | 7 | 4-week | 24-week Double-blinded Short-term Treatment Period | inded Sk | ort-tern | n Treati | nent Per | iod | | | | Notes |
| | Day 1 <sup>a</sup> | Day 2<br>(Phone Visit) | Day 4<br>(Phone Visit) <sup>b</sup> | Week 1 <sup>b</sup> | Day 10<br>(Phone Visit) <sup>b</sup> | Week 2 <sup>c,d</sup> | Week 4 <sup>c</sup> | Week 8 <sup>c</sup> | Week 10 <sup>c,e</sup> | Week 12 <sup>f</sup> | Week 18 <sup>c</sup> | Week 22 <sup>c, e</sup> | Week 24/Early<br>Term Visit <sup>g</sup> | |
| 6-point SMBG profiles | × | | | | | | | | | X | | | Xh | See Section 5.9.4.2 |
| Provide dietary and exercise counseling | × | | | × | | × | × | × | | × | × | | × | |
| Dispense subject<br>diaries and provide<br>instructions | × | | | × | | × | × | X | × | × | X | × | × | At Day 1, collect Lead-In Period diaries and dispense the first diaries in the Short Term Treatment Period |
| Re-dispense blood glucose and ketone strips and provide training (as needed) | × | | | | | | X | X | | × | X | | X | |
| Review subject diaries | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Adjust insulin dose (as needed) | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Collection of short-<br>term diaries. Dispense<br>long-term diaries. | | | | | | | | | | | | | × | |

| Table 5.1-2: | Flow | chart fo | r Protoco | ol MB1 | Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | 24-wee | k Doub | ole-blin | ded Sh | ort-ter | m Tre | atmen | t Perio | d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 7 | 24-week | 24-week Double-blinded Short-term Treatment Period | inded Sk | hort-tern | n Treatr | nent Per | iod | | | | Notes |
| | Day 1 <sup>a</sup> | Day 2<br>(Phone Visit) | Day 4<br>(Phone Visit) <sup>b</sup> | Week 1 <sup>b</sup> | Day 10<br>(Phone Visit) <sup>b</sup> | Week 2 <sup>c,d</sup> | Week 4 <sup>c</sup> | Week 8 <sup>c</sup> | Week 10 <sup>c,e</sup> | Week 12 <sup>f</sup> | Week 18 <sup>c</sup> | Week 22 <sup>c, e</sup> | Week 24/Early<br>Term Visit <sup>g</sup> | |
| | × | | | | | | | | | | | | × | Completed prior to any other procedures. For Day 1 visit assessment to be completed prior to first dose |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | |

| Table 5.1-2: | Flow | Flow chart for | | ol MB1 | Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | 24-weel | k Doub | le-blin | ded Sh | ort-ter | m Tre | atment | t Perio | þ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | 7 | 4-week | 24-week Double-blinded Short-term Treatment Period | nded Sh | ort-tern | 1 Treatn | nent Per | iod | | | | Notes |
| | Day 1 <sup>a</sup> | Day 2<br>(Phone Visit) | Day 4<br>(Phone Visit) <sup>b</sup> | Week 1 <sup>b</sup> | Day 10<br>(Phone Visit) <sup>b</sup> | Week 2 <sup>c,d</sup> | Week 4 <sup>c</sup> | Week 8 <sup>c</sup> | Week 10 <sup>c,e</sup> | Week 12 <sup>f</sup> | Week 18 <sup>c</sup> | Week 22 <sup>c, e</sup> | Week 24/Early<br>Term Visit <sup>g</sup> | |
| Laboratory<br>Assessments | | | | | | | | | | | | | | |
| Pregnancy test (urine) WOCBP only | × | | | | | | × | × | | × | × | × | × | Home pregnancy test kits sent home with WOCBP subjects to perform monthly pregnancy tests between visits and record results |
| Blood standard safety laboratory panel | X | | | | | | X | X | | X | X | | X | |
| Urine standard safety panel (dipstick) | X | | | | | | X | X | | | X | | | |
| Spot urine for glucose, albumin and creatinine quantification and determination of glucose: creatinine and albumin:creatinine ratios | × | | | | | | | | | × | × | | × | |
| FPG | X | | | X | | | | | | × | | | X | |

| Table 5.1-2: | Flow | chart fo | Flow chart for Protocol MB102230 - 24-week Double-blinded Short-term Treatment Period | ol MB1 | 02230 - 2 | 4-weel | k Doub | le-blin | ded Sh | ort-ter | m Tre | atment | t Perio | p |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | (4) | 24-week | 24-week Double-blinded Short-term Treatment Period | nded Sh | ort-tern | n Treatn | nent Per | iod | | | | Notes |
| | Day 1 <sup>a</sup> | Day 2<br>(Phone Visit) | Day 4<br>(Phone Visit) <sup>b</sup> | Week 1 <sup>b</sup> | Day 10<br>(Phone Visit) <sup>b</sup> | Week 2 <sup>c,d</sup> | Week 4 <sup>c</sup> | Week 8 <sup>c</sup> | Week 10 <sup>c,e</sup> | Week 12 <sup>f</sup> | Week 18 <sup>c</sup> | Week 22 <sup>c, e</sup> | Week 24/Early<br>Term Visit <sup>g</sup> | |
| FFA | × | | | | | | | | | | | | X | |
| A1C | | | | | | | × | × | | × | × | | × | |
| Fasting serum lipids | X | | | | | | | | | X | | | X | |
| PK sampling | | | | | | | | | | × | × | | $\mathbf{x}^{1}$ | Refer to Section 5.5 |
| Clinical Drug Supply | | | | | | | | | | | | | | |
| Randomize | X | | | | | | | | | | | | | |
| Dispense study drug | X | | | | | | X | X | | X | | | X | |
| Contact IVR system | × | | | | | | Xm | Xm | | Xm | | | X <sub>m</sub> * | *Also, call if<br>subject is<br>having an early<br>termination visit |
| Review study<br>medication compliance | X | | | X | | X | X | X | | X | X | | X | |
| Review study drug<br>dosing | | × | × | | × | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 1 visit should be within 56 days +/- 5 days of the Week -8 visit. If a retest of A1C is done at Week -1, a 7 day window (added to the current lead-in period window of 56+5 days) will be allowed

 $<sup>^{</sup>b}$  Visits may be scheduled  $\pm$  1 days to allow flexibility of scheduling.

 $<sup>^{\</sup>rm c}$  Visits may be scheduled  $\pm\,3$  days to allow flexibility of scheduling.

be sent (scan, photo, fax) into the site prior to the phone visit so discussions can occur between the subject and site personnel about the data captured in the Optional Phone Visit - Week 2 visit can be done as a phone visit to allow flexibility for the subject in visit scheduling. If a phone visit is done, the blood pressure, heart rate and body weight will not be done. A new week 2 diary should be given to the subject at the week 1 visit. Copies of completed diaries must

Optional Phone Visit - Week 10 visit and/or Week 22 visit can be done as a phone visit to allow flexibility for the subject in visit scheduling. If a phone visit is the subject at week 8 and/or week 18. The CGM sensor should be self inserted by the subject at home at week 11 for the first CGM wear in the short term period and/or at week 23 for the second CGM wear in the short term period and should be worn for 7 days. In those subjects having optional phone visits, this visit to confirm the insertion was done correctly. If the self-insertion is not done or no data is on the device at the week 12 and/or week 24 visit, then the done, the week 10 visit will move to be performed at week 11 and/or week 22 visit will move to be performed at week 23. CGM sensors (4) should be given to means that the CGM device would be worn for 7 days instead of the full 14 days Site personnel should call the subject for the week 11 visit and/or week 23 subject gets a new sensor inserted at the site and wears it for 7 days. After the 7 days of CGM wear is completed, following the week 12 visit, the subject will retain the sensor until returning to the site for the week 18 visit. After the week 24 visit, the subject will return the sensor to the site within 7 days of removal. If an optional phone visit is to be done, a new week 10 diary should be given at week 8 and/or a new week 22 diary should be given at week 18. Week 12 visit should be scheduled at least 14 days after Week 10 visit in order to collect a full 14-day CGM data, but not longer than 17 days. Sensors need to be changed 7 days after insertion. Subjects will be trained at the Week-1 visit to change the sensor. An ad-hoc visit may be performed if assistance is needed. If a subject performs sensor change on his/her own, the site should call to remind the subject to change the sensor 7 days after insertion.

Week 24 visit should be scheduled at least 14 days after Week 22 visit in order to collect full 14-day CGM data, but not longer than 17 days. Sensors need to be changed 7 days after insertion. Subjects will be trained at the Week-1 visit to change the sensor. An ad-hoc visit may be performed if assistance is needed. If a subject performs sensor change on his/her own, the site should call to remind the subject to change the sensor 7 days after insertion. If a randomized subject terminates the study any time prior to the Week 24 visit, the CGM, Recording Meals, and 6-point SMBG will not be required for the early termination visit. However, CGM, Recording Meals, and 6-point SMBG are expected to be performed at Week 12 and 24 off treatment visit, if the subject decides to continue with the study procedures If an optional phone visit is to be done at week 10, the subject diary should be given to the subject at week 8 and/or a new week 22 diary should be given at

For the Day 1 visit - it will be recommended that subjects reduce their daily insulin dose by up to 20% for both basal and bolus insulin after the first dose of study drug, although in some cases it may be necessary to reduce insulin (particularly basal insulin) in advance of study drug administration.

These safety assessments; review of AEs, hypoglycemia events, and DKA episodes to be performed throughout the study according to the visit schedule as noted via "X."

PK samples should be collected if the visit is being used as an early termination visit or if it is the subject's regularly scheduled week 24 visit and the subject is currently taking study medication. In the event that the subject discontinues study medication but continues in the study, any PK samples required at visits should not be done

If visit is during the "off-treatment" or the Post Study Drug Study Follow-up phase (Section 3.6), the IVRS does not have to be contacted

| Table 5.1-3: Flow chart for 1 | rt for Proto | col MB102 | 230 - 28-w | eek Subject- ar | nd Site-Blinded Lo | Protocol MB102230 - 28-week Subject- and Site-Blinded Long-term Treatment Period |
|---|---|---|---|---|---|---|
| Procedure | 28-we | ek Subject ar | nd Site blinde | 28-week Subject and Site blinded Long-term Treatment Period | atment Period | Notes |
| | Week 32 <sup>a</sup> | Week 40 <sup>a</sup> | Week 48 <sup>a</sup> | Week 52 <sup>a</sup> / ET<br>Visit For<br>Long- term | Week 56 <sup>a</sup> Follow-up (for both ST and LT periods) | |
| Subject reports to site | X | X | X | X | X | |
| General Procedures | | | | | | |
| Brief physical exam | | X | | | × | Includes cardiovascular, lungs, abdomen, and extremities, and any organ systems pertinent to the subject's signs, symptoms, or AEs |
| Complete physical exam | | | | × | | Includes general appearance, head, eyes, ears, nose, throat, neck, cardiopvascular, lungs, abdomen, lymph nodes, extremities, neurological, skin, and musculoskeletal. |
| Body weight | X | X | X | X | X | |
| Blood pressure and heart rate | X | × | × | × | × | |
| ECG | | | | X | | |
| Review concomitant medications/procedures | X | X | X | X | X | |
| Provide dietary and exercise counseling | X | X | X | X | | |
| Dispense study diaries and provide instructions | X | X | X | X | | |
| Re-dispense blood glucose and ketone strips and provide retraining (as needed) | X | X | X | X | | |
| Review subject diaries | X | X | X | X | X | |

| Table 5.1-3: Flow chan | rt for Proto | col MB102 | 230 - 28-w | eek Subject- ar | nd Site-Blinded Lo | Flow chart for Protocol MB102230 - 28-week Subject- and Site-Blinded Long-term Treatment Period |
|---|---|---|---|---|---|---|
| Procedure | 28-we | ek Subject an | d Site blinde | 28-week Subject and Site blinded Long-term Treatment Period | atment Period | Notes |
| | Week 32 <sup>a</sup> | Week 40 <sup>a</sup> | Week 48 <sup>a</sup> | Week 52 <sup>a</sup> / ET<br>Visit For<br>Long- term | Week 56 <sup>a</sup> Follow-up (for both ST and LT periods) | |
| Adjust insulin dose (as needed) | X | X | X | X | | |
| Collection of long-term treatment period diaries | | | | | X | |
| Administer EQ-5D-3L, DTSQs, and HFS-II | | | | X | | Completed prior to any other procedures |
| Safety Assessment | | | | | | |
| Assess AEs | X | × | X | × | X | |
| Assess hypoglycemia episodes | X | X | X | X | X | |
| Assess DKA | X | X | X | X | X | |
| Laboratory Assessments | | | | | | |
| Pregnancy test (urine) WOCBP only | X | × | × | × | × | Home pregnancy test kits and pregnancy logs sent home with WOCBP to perform monthly pregnancy tests between visits and record results in log book. |
| Blood standard safety laboratory panel | | × | | X | X | |
| Urine standard safety (dipstick) | | X | | X | X | |
| Spot urine for glucose, albumin and creatinine quantification and determination of glucose: creatinine and albumin:creatinine ratios | | | | X | × | |
| FPG | | | | X | X | |

| Table 5.1-3: | Flow chai | rt for Proto | col MB102 | 230 - 28-w | eek Subject- ar | nd Site-Blinded La | Flow chart for Protocol MB102230 - 28-week Subject- and Site-Blinded Long-term Treatment Period |
|---|---|---|---|---|---|---|---|
| Procedure | | 28-we | ek Subject ar | nd Site blinde | 28-week Subject and Site blinded Long-term Treatment Period | atment Period | Notes |
| | | Week 32 <sup>a</sup> | Week 40 <sup>a</sup> | Week 48 <sup>a</sup> | Week 52 <sup>a</sup> / ET<br>Visit For<br>Long- term | Week 56 <sup>a</sup> Follow-up (for both ST and LT periods) | |
| A1C | | × | × | × | X | X | |
| FFA | | | | | X | | |
| Fasting lipid panel | | | | | × | | |
| Clinical Drug Supply | | | | | | | |
| Dispense study drug | | X | X | | | | |
| Contact IVR system | | X <sub>c</sub> | X <sub>c</sub> | | X <sub>c</sub> * | X | *Also, call if subject is having an early termination visit |
| Review study medication compliance | | X | X | X | X | | |

Visits may be scheduled  $\pm$  5 days to allow flexibility of scheduling with the exception of Week 56 visit. Week 56 visit cannot be scheduled earlier than 30 days of week 52 visit or last dose of study drug but can have a longer window of 5 days.

b These safety assessments; review of Adverse Events, hypoglycemia events, and DKA episodes, to be performed throughout the study according to the visit schedule as noted via "X."

c If visit is during the "off-treatment" the Post Study Drug Study Follow-up phase (Section 3.6), the IVRS does not have to be contacted

### 5.1.1 Retesting During Screening or Lead-in Period

Retesting of laboratory parameters and/or other assessments during the Screening or Lead-in period will not be permitted (this does not include parameters that require a confirmatory result).

### Retesting is limited to HbA1C and free T4 as described in Section 3.3.

Any new result will override the previous result (ie, the most current result prior to randomization) and is the value by which study inclusion will be assessed, as it represents the subject's most current, clinical state.

### 5.2 Study Materials

BMS will supply the sites with the following materials as allowed per local regulations.

- Blood glucose/ketone meters. One (1) meter will be provided to each study subject at lead-in and one meter will be provided to each investigative site
- Glucose and ketone test strips
- Lancets
- Glucose control solutions
- CGM devices and software to download data (see paragraph at the end of this section)
- Subject education and site support materials (eg, CGM instruction manuals)
- Electronic case report forms (eCRFs) (Serious Adverse Event [SAE] Forms, Pregnancy Surveillance Forms, Events of Special Interest]
- Subject alert cards
- Study drug inventory control forms
- Site file
- Subject diary:
  - Full diary review by site staff is required for this study during each visit
  - Use of subject diaries are mandatory for the study and will be maintained by each study subject for documentation of 6-point SMBG results and SMBGs from the Day 1 visit to the Week 2 visit, insulin doses, meal times during specific weeks of CGM monitoring, day/time of CGM sensor insertion if performed at home at Weeks 11 and 23, study medication dosing, ketone testing, DKA symptoms, hypoglycemia episodes, and if applicable WOCBP urine pregnancy results
    - ♦ 6-point SMBG profiles: see Section 5.9.4.2
    - ♦ SMBG: see Section 5.3.2.1
    - ♦ Subjects are to be instructed to document their insulin dose in their study diaries during the protocol-defined time period as outlined in Section 5.3.4. eCRF pages will be provided to the sites so they can record the data obtained from the diaries in the study database
      - Subjects who have not recorded all of their insulin doses should be assessed by the study staff for their ability to comply with the protocol. The diaries are to be maintained to ensure subject safety and must be completed by the subject


throughout the study. Compliance with prescribed insulin administration and diary completion should be assessed and re-enforced at every visit

- Subjects are to record their meal times in their diary during the following time periods:
  - Week -1 to Day 1 prior to randomization
  - o Week 11 to Week 12
  - O Week 23 to Week 24
- ◆ Subjects are to record day and time of CGM sensor insertion if performed at home at week 11 and week 23
- ♦ The dates, time, and number of tablets of study medication taken by the subject are to be recorded in the study diary. Electronic CRF pages will be provided to the sites so they can record the data obtained from the diaries in the study database
- ♦ Subjects are to record any hypoglycemic symptoms they may experience and SMBG values if they conducted the test when they had symptoms in their diaries. All events recorded in subject diary will be reviewed by site staff according to Section 5.3.2
- ◆ Any ketone testing performed by the subject, symptoms potentially associated with DKA, and relevant events (Section 5.3.3) are to be recorded in the diary. All results recorded in subject diary will be reviewed by site staff during each study visit. Determination of a DKA event must be assessed and documented by the Principal Investigator or by a qualified sub-investigator.
- Any other materials as locally required or agreed upon

The central laboratory will provide all laboratory-related materials including home pregnancy testing kits for WOCBP to the study sites.

Materials related to the CGM will be provided by a central vendor. Dexcom Inc is planned to be the provider of these devices; however, the Sponsor may change the provider as needed. Below is a summary of selected information related to the specifications of the planned CGM system:

### Model No (range)/Name:

- STK-GL-(00l to 099) / mg/dL, Dexcom G4 PLATINUM Receiver Kit
- STK-GL-(101 to 199) / mmol/L, Dexcom G4 PLATINUM Receiver Kit
- STR-GL-(002 to 099) / mg/dL, Dexcom G4 PLATINUM Replacement Receiver Kit
- STR-GL-(101 to 199) / mmol/L, Dexcom G4 PLATINUM Replacement Receiver Kit
- STT-GL-(00l to 010) / Dexcom G4 PLATINUM Transmitter Kit
- STS-GL-(00l to 144) / Dexcom G4 PLATINUM Sensor
- MT21190 / Dexcom Studio

All the information for devices used in this study is available from the vendor(s).


### 5.3 Safety Assessments

Safety assessments will include adverse event reporting, as well as marked abnormalities in clinical laboratory tests. Please refer to Appendix 2 for details on central laboratory assessments.

The procedures described in the sections that follow will also be completed to ensure subject's safety.

### 5.3.1 Imaging Assessment for the Study

Not applicable.

# 5.3.2 Self-Monitored Blood Glucose (SMBG) and Guidance on Management and Reporting of Hypoglycemia Episodes

Any incidental findings of potential clinical relevance that are not directly associated with the objectives of the protocol should be evaluated and handled by the investigator as per standard medical/clinical judgment.

### 5.3.2.1 Self-Monitored Blood Glucose (SMBG)

Combination glucose and ketone meters will be supplied to each study site. At the entry into the lead-in period, subjects will receive a glucose and ketone meter, supplies and instruction on their use. Testing supplies will be provided to allow for blood glucose and ketone testing for the duration of the study. Subjects should bring their glucose meter with them to each study visit to ensure that it is functioning properly and for review of SMBG results. Subjects may keep the glucose meters at the end of the study. It is strongly preferred that subjects use the meter provided by the Sponsor. If a subject uses another meeting to perform this test, these results will be captured on an eCRF page.

Subjects should self-monitor their blood glucose at least 4 times per day (generally before breakfast, lunch, dinner, and bedtime), and in the occurrence of hypoglycemic symptoms, and to contact the investigator in the event of an unusually high or low blood glucose value. In addition, study subjects should comply with the site's instructions with regard to self-monitoring of blood glucose and insulin adjustments accordingly and should report to the site blood glucose values and/or signs and symptoms suggestive of a hypoglycemic episode.

Subjects should attempt to enter all valid SMBG values into the CGM in order for the calibration of the system.

The glucose values should be reviewed by the site to identify any unusual high or low values, and to confirm that the values (from the glucose and ketone meter's memory and/or from the subject's hypoglycemia portion in the diary) were obtained from the subject. If fingerstick glucose values are discordant from glycemic control assessed by the central laboratory or with clinical symptoms, the subject's glucose and ketone meter should be tested and the procedure for using it reviewed with the subject.


### 5.3.2.2 Guidance on Management and Reporting of Hypoglycemia Episodes

Hypoglycemia may be an expected event in subjects who are treated for diabetes. Subjects and their family members must be aware of the possibility that hypoglycemia may occur and the dangers associated with low blood sugar.

Study subjects must be properly instructed on the recognition and management of hypoglycemia. Subjects should record any hypoglycemic symptoms in their diaries. They should be encouraged to measure, when possible, their blood glucose values when they have symptoms of hypoglycemia. Subjects should carry with them easily ingestible forms of carbohydrate at all times in order to treat an event of hypoglycemia should it occur.

During clinical trials, subjects frequently report symptoms of hypoglycemia when asked, even when treated with placebo or medications not otherwise associated with hypoglycemia. As hypoglycemia is an important event associated with diabetes therapy, all episodes which could be consistent with the clinical definition of hypoglycemia as assessed by the investigator should be documented and reported on the appropriate eCRF page.

Hypoglycemia eCRF pages will be used to document all reported episodes of hypoglycemia. The investigator is responsible for questioning the subject about all symptoms reported on the hypoglycemia portion of the diary and for determining if they meet the clinical definition of hypoglycemia. Only symptoms and/or blood glucose values deemed by the investigator to meet the definition of hypoglycemia should be reported on the hypoglycemia eCRF pages. Signs and symptoms of hypoglycemia, hypoglycemia episodes or discontinuation due to hypoglycemia should not be reported on the AE eCRF page, unless the event fulfills protocol criteria for an SAE (see Section 6.1.1), in which case an SAE form must be completed in addition to the hypoglycemia eCRF pages for hypoglycemia.

## 5.3.3 Self-Monitored Blood Ketone Testing and Guidance on Management and Reporting of Diabetic Ketoacidosis Episodes

Diabetic ketoacidosis is an expected event in subjects with T1DM. Subjects and their family members must be aware of the possibility that DKA may occur and the dangers associated with DKA.

Dapagliflozin reduces blood glucose by urinary excretion of glucose, thus representing a daily removal of a substantial amount of carbohydrate from the body. We estimate (from insulin:carbohydrate ratios) that the amount of glucose excreted in the urine in subjects on dapagliflozin may correspond to the glycemic effect achieved from as much as 20% of a subject's total daily insulin dose and, therefore, insulin dose reductions will have opposite glycemic effects compared to those of dapagliflozin. Furthermore, since DKA is caused by gross insulin deficiency and is mechanistically unrelated to glucose levels per se (as can be seen in euglycemic DKA), reductions in insulin doses of more than 20% are not recommended regardless of glucose values. If subjects have repeatedly low blood glucose and could otherwise not avoid a 20% reduction in total daily insulin dose, they are recommended to increase their daily dietary carbohydrate intake. Similarly, subjects should be reminded that during/after elevated physical activity/exercise, dapagliflozin continues to remove glucose in addition to what


is being consumed by the physical activity. Therefore, additional (re-) fueling with carbohydrates is important and should generally be preferred over higher than usual reductions in subjects' insulin doses.

As noted above, subjects will receive a combined glucose and ketone meter and sufficient supplies for testing at the entry into the lead-in period. Subjects will also be trained in the procedure of conducting blood ketone testing according to the manufacturer's specifications. Subjects will be advised to measure their blood ketones using the glucose and ketone meter provided by the Sponsor when they have potential symptoms/signs of DKA, including but not limited to: excessive thirst, nausea and vomiting, frequent urination, weakness or fatigue, fever, fruity-scented breath, confusion, and/or consistently elevated blood glucose, and/or during acute illness. Subjects should be instructed to measure their ketones if symptoms occur, regardless of plasma glucose values. Blood ketone test results, symptoms potentially associated with DKA, and relevant risk factors (eg, missed insulin injection, insulin pump malfunction, infection, heart attack, etc) should be recorded in the subject diary.

Study subjects must be properly instructed on the recognition and management of DKA. Subjects should contact the site for assistance with diabetes management in the event that the blood ketone reading is 0.6 mmol/l or above according to the glucose/ketone meter user guide. The investigator is recommended to advise the subject to take extra insulin and extra carbohydrate if elevated ketones are registered and continue to measure blood ketones. If deemed necessary, dosing of study medication should be interrupted during sick days. The action, follow-up, and monitoring plan will be at the discretion of the investigator and will depend on his/her judgment of severity based on signs/symptoms of DKA, risk factors, relevant contributing factors, and blood glucose (with the caveat that the blood glucose may be lower than would be otherwise expected given elevated ketone levels). ). It is recommended that for subjects who report elevated ketones/ketosis, the investigator considers re-education concerning DKA at the next scheduled visit, at an un-scheduled visit or by telephone contact, as appropriate.

Subjects must also be instructed that if attempts to contact the site are unsuccessful or if they are in urgent need of medical attention, that they should seek medical attention. They should provide information to the health care provider on their participation in a placebo controlled clinical study evaluating the effects of the SGLT2i dapagliflozin in addition to their insulin treatment.

The blood ketone values should be reviewed by the site to identify any unusual high values, and to confirm that the values (from the glucose and ketone meter's memory and/or from the subject's diary) were obtained from the subject. If fingerstick blood values are discordant from glycemic control assessed by the central laboratory or with clinical symptoms, the subject's glucose and ketone meter should be tested and the procedure for using it reviewed with the subject. Investigators will examine if any of the elevated ketone values from the subject's diary are associated with a DKA event. If yes, investigators will document all DKA related symptoms, relevant risk factors, and available laboratory test results (including blood ketone values and blood glucose values measured by the glucose/ketone meter) on the DKA eCRF pages and report


this event to the Sponsor. Blood ketone and glucose values associated with events deemed not to be a DKA event should be recorded on the non-DKA eCRF log page.

In addition the Sponsor will utilize Standardized Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs) based on a list of pre-defined terms in MeDRA to identify potential DKA events. The list of these terms are included in the Data Monitoring Committee (DMC) Charter. Investigators will further evaluate these cases and if the event is determined to be DKA, the investigator will complete the DKA eCRF.

Regarding the reporting of DKA events, it is important to distinguish ketosis from DKA. Low levels of ketosis, in which blood or urine ketone values are elevated, can occur in individuals who follow a low-carbohydrate, high-fat diet (eg, dietary ketosis) or after prolonged periods of fasting. However, ketosis is a benign condition if symptoms are absent and the blood pH remains buffered within normal limits (eg, no acidosis). In contrast, DKA episode may be confirmed when subjects have potential symptoms/signs of DKA (polyuria, polydipsia, weight loss, vomiting, abdominal pain, signs of volume depletion on physical examination), marked hyperglycemia (although DKA has been reported in individuals with normal or mildly elevated plasma glucose levels as well), elevated blood/urine ketone values, and a metabolic acidosis characterized by low arterial blood pH values, decreased serum bicarbonate, and an increased anion gap. The combination of specific symptoms/signs of DKA and elevated blood/urine ketone values may be suggestive of DKA, recognizing that some subjects may not have lab test results (eg, blood gas measurement) to confirm acidosis.

During clinical trials, subjects frequently report symptoms of DKA when asked, even when treated with placebo or medications not otherwise associated with DKA. The investigator is responsible for questioning the subject about all DKA related symptoms reported on the subject diary and for determining if they meet the clinical definition of DKA. Only the episodes deemed by the investigator to meet the definition of DKA should be reported on the DKA eCRF pages. Signs and symptoms of DKA, DKA episodes, or discontinuation due to DKA should not be reported on the AE eCRF page, unless the event fulfills protocol criteria for an SAE (see Section 6.1.1), in which case an SAE form must be completed in addition to the DKA eCRF pages. If a DKA episode occurs in a subject that fails screening, the DKA eCRF pages do not need to be completed. However, if the event meets the protocol criteria for an SAE, the SAE form must be completed. For subjects who experience a DKA it is recommended that the investigator schedules a telephone or site visit for re-education in prevention of ketosis and DKA.

A DKA Adjudication Committee, blinded to the treatment of the subjects, will independently adjudicate all the DKA events reported by investigators during the study period. A separate Adjudication Manual will define and describe the procedure for the handling, reporting, and classification of these cases.

The key goals of treating DKA include correcting dehydration, hyperglycemia, and electrolyte imbalance, and identifying and appropriately treating comorbid precipitating events. Subjects with DKA should be carefully monitored until significant improvement in the symptoms,


normalization of blood acidity (eg, pH > 7.3), and improvement/absence of ketones in blood or urine.

### 5.3.4 Insulin Dosing Adjustment and Data Collection Guidelines

Adjustment of a subject's pre-existing insulin dosing regimen may be required during the conduct of this study, due to changes in diet, activity, emotional stress during the study, as well as potential effects of dapagliflozin to reduce blood glucose and thereby insulin requirements.

During the lead-in period, subjects will be advised to self-monitor their blood glucose consistent with local treatment guidelines. The method of documentation for glucose results will be based on local clinic practice. Glucose control will be reviewed by the investigator at each visit. Insulin dose may be adjusted as deemed appropriate to be consistent with good medical practice according to SMBG readings, local guidance and individual circumstances.

It is recommended that subjects reduce their daily insulin dose by up to 20% for both basal and bolus insulin after the first dose of study drug to minimize the risk of hypoglycemia. It is at the discretion of the investigator to determine the extent to which to reduce the insulin doses. In some cases it may be necessary to reduce insulin (particularly basal insulin) in advance of study drug administration. If total daily insulin dose is reduced upon initiation of study medication, attempts must be made to titrate insulin back to baseline total daily insulin dose. It is not recommended to reduce total daily insulin dose by more than 20% compared to baseline at any time during the study unless medically indicated and close attention should be paid, especially in these subjects, to symptoms of, and risk factors for developing DKA (See also Section 5.3.3). Subjects are to be instructed to document their daily individual insulin doses and self-monitor glucose values at least 4-times every day (before breakfast, lunch, dinner, and bedtime) during the first 2 weeks. This information will be used to facilitate appropriate insulin dose adjustment and ensure subject safety. For the rest of the study period (both short-term and long-term), subjects will be advised to continue self-monitoring their blood glucose as per local guidelines. Glucose control will be reviewed by the investigator at each visit. Insulin dose may be adjusted as deemed appropriate to be consistent with good medical practice according to SMBG readings, local guidance, and individual circumstances. The glycemic control goals may be individualized based upon a subject's personal target and stability of glycemic control at baseline.

Subjects are not allowed to change their insulin administration methods (MDI or CSII) throughout the study unless a subject using an insulin pump needs to replace the pump. Under this situation, the subject may temporarily use MDI and should restart CSII administration as early as feasible. The period of time a subject is on temporary use of MDI should not be more than 2 weeks.

### **Insulin Dosing Recording**

At the following time periods the subjects will be instructed to record all their individual doses of (basal and bolus) insulin in their study diary.

• Week -2 visit up to the Day 1 visit prior to randomization


- Day 1 visit after randomization up to the Week 2 visit
- Week 10 visit up to the Week 12 visit
- Week 22 visit to up the Week 24 visit

The site will review these diary entries and record the total basal and total bolus daily dose of insulin the subject received on the eCRF. For statistical analysis purposes the total daily dose is defined as the sum of all these individual doses of insulin (both basal and bolus) during a 24-hour period.

Subject's daily individual insulin doses and self-monitored glucose values collected from Day 1 visit (after randomization) to the Week 2 visit will be used to facilitate appropriate insulin dose adjustment and ensure patient safety.

At the following time periods subjects will be instructed to record the minimum and maximum total daily insulin dose range (basal plus bolus) taken for each week in their study diary:

- Week -8 visit up to the Week -2 visit
- Week 2 visit up to the Week 10 visit
- Week 12 visit up to the Week 22 visit
- Week 24 visit up to the Week 56 visit

The site will review these diary entries and record the weekly ranges subject received of insulin on the eCRF.

### 5.3.5 Guidance on Assessment of Urinary Infections and Hematuria

### 5.3.5.1 Guidance on Assessment of Urinary Infections

The following is presented to assist in the classification and management of urinary tract infections. It is not intended to supplant investigators' clinical judgment: It is at the discretion of an investigator to determine whether and when to send an initial urine culture.

Study drug should be withheld in subjects with clinical evidence of a UTI or presumed urosepsis until the course of treatment of the infection has been completed and clinical recovery has occurred.

It is recommended that a urine culture be obtained by local laboratory within 7 days of clinical recovery from all <u>treated</u> urinary tract infections. Whether or not additional therapy is prescribed because of culture results should be determined by investigator judgment, after consultation with the Medical Monitor.

It is the investigator's responsibility to report, as applicable based on the investigator's judgment and the subject's medical history, related adverse events as defined in Section 6. Additional information, including but not limited to completion of supplemental eCRFs or questionnaires may be requested for certain adverse events and/or laboratory abnormalities which are reported/identified during the course of the study.


### Asymptomatic Bacteriuria

During enrollment, treatment and follow up of subjects in this trial, the investigator may discover a subject with asymptomatic bacteriuria. Asymptomatic bacteriuria is defined as the presence of ≥ 10<sup>5</sup> colony forming units/mL of bacteria, in a properly collected voided urine specimen, without signs or symptoms typically attributed to urinary tract infection. Asymptomatic bacteriuria is prevalent among diabetic women, and is associated with pyuria in 70% of cases. Neither guidelines from the Infectious Diseases Society of America (IDSA), US Preventive Services Task Force, <sup>15,16</sup> nor the European Association of Urology <sup>17</sup> recommend screening for or treatment of, asymptomatic bacteriuria in non-pregnant diabetic patients. In this study, the central laboratory will report urinary dipstick test results for hemoglobin but will not routinely report the results of urinary dipstick tests for leukocyte esterase as a screening test for pyuria in surveillance urine examinations.

### 5.3.5.2 Guidance on Assessment of Hematuria

During the course of the study, hematuria should be investigated according to local standards and best clinical practices for a possible cause.

If **NO** common cause is identified, subjects should be further investigated based on American Urological Association (AUA) guidelines or equivalent local standard of care and best practices, which could include referral to a urologist and undergoing evaluation that may include abdominal computed tomography (CT), urine cytology, and an NMP-22 urine test. The subject should continue to be randomized/receive investigational product treatment during these investigations (unless otherwise contraindicated).

It is the investigator's responsibility to report, as applicable based on the investigator's judgment and subject's medical history, related adverse events as defined in Section 6. Additional information, including but not limited to completion of supplemental eCRFs or questionnaires may be requested for certain adverse events and/or laboratory abnormalities which are reported/identified during the course of the study.

### 5.3.6 Guidance on Assessment of Cardiovascular Events

A Clinical Events Committee (CEC), blinded to the treatment of the subjects, will independently adjudicate certain cardiovascular adverse events, and they will operate in accordance with a dedicated Clinical Events Committee Charter/Manual of Operations:

Events related to the following will be sent to the CEC for adjudication.

Death, including:

- Cardiovascular death
- Non-cardiovascular death

Myocardial infarction (MI), including:

• ECG and/or cardiac enzymes confirmed MI

Revised Protocol No.: 02 Date: 18-May-2016

- Sudden death
- Percutaneous coronary intervention (PCI)-related MI
- Coronary artery bypass graft (CABG)-related MI
- MI diagnosed via pathologic criteria
- Silent MI

Fatal and non-fatal stroke, including:

- Ischemic stroke
- Hemorrhagic stroke

Serious Adverse Events of the following:

- Heart failure
- Cardiac arrhythmia
- Unstable angina
- Unplanned arterial revascularization (coronary, carotid and peripheral)
- Cardiac arrest with successful resuscitation
- Deep vein thrombosis (DVT) and pulmonary emboli (PE)
- Systemic non-stroke arterial embolism/thrombosis including systemic arterial occlusion
- Non-traumatic amputation of the lower limb. Only events above the ankle will be considered for adjudication.

In order to provide the independent CEC with appropriate and adequate information for adjudication of the listed events, please consult the Adjudication Reference Manual for Primary Investigators and Study Staff.

### 5.3.7 Guidance on Assessment of Hepatic Laboratory Abnormalities

An independent Hepatic Adjudication Committee, blinded to the treatment of the subjects, will determine the probability that drug-induced liver injury (DILI) is the cause of liver-related abnormalities, included, but not limited to:

- AST and/or ALT > 3x ULN and total bilirubin (TB) > 2x ULN (within 14 days of the AST and/or ALT elevation)
- Hepatic events timely related to death (within 30 days before death)
- AST and/or ALT > 10x ULN

### Hepatic disorders leading to discontinuation from study drug and/or death

Liver laboratory abnormalities such as elevated AST and/or ALT with or without TB Elevations


A separate Adjudication Charter will define and describe the procedure for the handling, reporting and classification of these cases.

The following is presented to assist in the evaluation and management of hepatic laboratory values. It is not intended to supplant the investigator's clinical judgment. Subjects who experience ALT and/or AST values > 3x ULN confirmed with a repeated test will have the following performed within 3 days of the confirmed laboratory results:

- AE assessment
- Physical examination for jaundice and other signs of liver diseases
- Review of relevant risk factors and current history focusing on possible causes of the increased ALT and/or AST and/or TB, including:
  - Use of suspect concomitant medication [including over-the-counter (ie, acetaminophen/paracetamol), herbal and vitamin preparations]
  - Recent alcohol consumption or recreational drug/narcotic use
  - Recent unaccustomed physical exertion
  - Occupational or environmental exposure to hepatotoxins
  - Other conditions which may cause liver diseases or which may cause abnormal test results
- Specialized liver laboratory panel (see Appendix 2)
  - should only be done once for elevated liver enzymes per Appendix 3 Sustained Elevated Liver Safety Abnormalities Flow Chart unless liver discontinuation panel is required

Additional information, including but not limited to completion of supplemental eCRFs or questionnaires, may be requested for certain adverse events and/or laboratory abnormalities which are reported /identified as part of the hepatic safety surveillance.

For subjects who are discontinued from study medication as a result of sustained elevated liver safety abnormalities, as described in Section 3.5, additional blood sampling must be done within 3 days of the confirmed laboratory results (see Appendix 3), in conjunction with an Early Treatment Discontinuation (End-of-Treatment) visit, in addition to the procedures noted above. A referral consultation to a hepatologist or gastroenterologist (specializing in liver abnormalities) should be obtained. Any additional tests and/or examinations should be carried out at the discretion of the Investigator. Any further investigations and laboratory results for subjects with abnormal laboratory values at the follow-up visit should be made available to the Sponsor upon request.

### 5.3.8 Physical Examination

 A brief physical examination should include cardiovascular, lungs, abdomen, and extremities, and any organ systems pertinent to the subject's signs, symptoms, or adverse events

A complete physical examination should include general appearance, head, eyes, ears, nose, throat, neck, cardiovascular, lungs, abdomen, lymph nodes, extremities, neurological, skin, and musculoskeletal

The individual performing the physical examinations must be licensed by state or national law (or applicable local law) to perform this procedure.

#### 5.3.9 Blood Pressure and Heart Rate

Blood pressure (BP) and heart rate (HR) measurements must be taken consistently throughout the study. Only the right or the left arm should be used when measuring these parameters. The arm that was used should be documented, along with the observer's initials; the same arm should be used at each visit. The subject should be in a seated position, allowing at least 5 minutes of rest before measurement. Blood pressure should be measured with the subject's arm resting on a table, and with subject's back supported and feet flat on the floor.

Blood pressure and HR will be determined from three replicate measurements obtained at least 1 minute apart. The average BP and HR will be determined from these 3 replicate measurements and reported in the eCRF.

All measurements should occur at least 8 hours after the last ingestion of caffeine, alcohol, or nicotine.

## 5.3.10 Electrocardiograms

Electrocardiograms will be performed as noted in Section 5.1. The investigator should review and assess all ECGs for any clinically significant abnormalities, and initial and date the report. The screening ECG must be assessed, and initialed and dated by the investigator prior to randomizing the subject. In preparation for the ECG, there should be minimal interference between the skin surface and the electrode. Alcohol should be used to prepare the skin at each electrode site. Thick chest hair should be shaved to ensure sufficient contact. Before attaching electrodes to pick-up points, electrode gel should be applied to the electrodes. The electrodes should be placed on bony areas, avoiding large muscle masses, to achieve better tracings as described below. The subject must be supine and should refrain from movement during the ECG recording. The subject and the electrodes (including the neutral electrode) should not be exposed to conducting objects, even if grounded.

- RL: On the right leg (inside calf, midway between knee and ankle)
- LL: On the left leg (inside calf, midway between knee and ankle)
- RA: Right arm (on the inside)
- LA: Left arm (on the inside)
- V1: 4th intercostal space, at right sternal margin
- V2: 4th intercostal space, at left sternal margin
- V3: Midway between V2 and V4
- V4: 5th intercostal space at left midclavicular line


930087408 3.0

v3.0

- V5: Same transverse level at V4, at anterior axillary line
- V6: Same transverse level at V4, at left midaxillary line

One original ECG print-out should be kept in the medical chart and a copy, assessed, initialed and dated by the investigator, should be maintained in the source documents for the study.

## 5.3.11 Guidance on Volume Depletion

Dapagliflozin has a modest diuretic effect. The risk of volume depletion is enhanced when two diuretics are used in combination and in subjects that otherwise are at risk for volume depletion. Therefore, caution should be exercised when administering dapagliflozin to subjects at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics. These subjects should be carefully monitored for of volume status, electrolytes, and renal function.

## 5.3.12 Guidance on Monitoring Renal Function

#### Creatinine clearance (CrCl, based on Cockroft-Gault) ≥ 45 ml/min and < 60 ml/min:

- At all scheduled and unscheduled visits, patients should be asked for symptoms of volume depletion, as well as other AEs, and vital signs should be assessed (including blood pressure measurement).
- Renal function should be monitored by central lab at all scheduled and unscheduled visits.

#### Creatinine clearance (CrCl, based on Cockroft-Gault) ≥ 30 ml/min and < 45 ml/min:

- If the creatinine clearance (CrCl, based on Cockroft-Gault) falls below 45 ml/min, the patient should be scheduled for a re-test within 4 days, whenever possible.
  - If the re-test CrCl (based on Cockroft-Gault) is ≥ 45 ml/min the patient can resume the normal visit schedule.
  - If re-test CrCl is still < 45 ml/min, the Investigator should consider re-testing CrCl within one to two weeks, whenever possible.
- In addition, the Investigator should consider evaluating the subjects for potentially reversible causes of renal dysfunction including: concurrent use of NSAIDS, antibiotics, or other medications known to affect creatinine clearance; volume depletion; urinary tract infection and obstructive uropathy. Further re-testing and evaluation should be done every second week until stabilization.

#### Creatinine clearance (CrCl, based on Cockroft-Gault) < 30 ml/min:

See Section 3.5 for re-testing instructions and possible need for study medication discontinuation.


Any subject that is discontinued from study medication due to deterioration in renal functions should be monitored closely by the investigator until abnormalities stabilize and the subject is asymptomatic.

## 5.3.13 Supplemental Visits

#### 5.3.13.1 Early Treatment Discontinuation Visit

#### Subjects discontinued from the double-blinded short-term treatment period

Any subject who discontinues study medication during the 24-week double-blinded short-term treatment period must have the Week 24/Early Termination (ET) visit completed. The Week24/ET visit eCRF will also need to be completed and a Week 24/ET visit laboratory kit will need to be used to collect ET visit blood and urine samples. The IVRS must be called to record the subject status (ie, discontinuation status).

## Subjects discontinued from the subject and site blinded long-term treatment period

Any subject who discontinues study medication during the 28-week subject- and site-blinded long-term treatment period must have the Week 52/ET visit completed. The IVRS must be called to record the subject status (ie, discontinuation status). The Week 52/ET visit eCRF will also need to be completed and a Week 52/ET visit laboratory kit will need to be used to collect ET Visit blood and urine samples.

## 5.3.13.2 Early Treatment Discontinuation Follow-up (Off Treatment Procedures)

As described in Section 3.6, all subjects who discontinue investigational product during the 24-week double-blinded short-term treatment period or the subject- and site-blinded long-term treatment period are expected to continue study participation for each scheduled visit for the remaining length of the study and complete all procedures as outlined in the Section 5.1 study flowchart (with the exception of study drug management and PK sampling). If continued study participation according to the protocol schedule is not possible, the investigator should contact the subject to discuss alternatives (eg, return to the clinic 4 weeks/at least 30 days after discontinuation of study drug to perform the week 56 post treatment follow-up procedures as outlined in Section 5.1 study flowchart or be contacted by telephone 30 days after discontinuation of study drug to evaluate the following safety assessments: AEs, hypoglycemia events, and DKA episodes). Please note that after the discontinuation of study drug, management of the subject's diabetes would be under the care and direction of the investigator and/or subject's healthcare providers.

Please utilize the post treatment follow up pages in the eCRF post treatment section for this data completion.

#### 5.3.13.3 Other Supplemental (Unscheduled) Visits

At any time during the trial, the investigator may, at his/her discretion, arrange for a subject to have an unscheduled (supplemental) assessment(s), especially in the case of AEs that require follow-up. If a subject is seen for an unscheduled assessment, the appropriate Supplemental Pages of the eCRF must be completed.


930087408 3.0

v3.0

#### 5.4 Efficacy Assessments

The procedures described in the sections that follow will completed to capture information for efficacy assessments.

#### 5.5 Pharmacokinetic Assessments

PK samples will be obtained prior to dosing at the Weeks 12, 18, and 24 visits.

Please refer to the central laboratory instructions for sample collection and processing

#### 5.6 Pharmacogenomic/Pharmacogenetic Assessements

Pharmacogenetic samples may be collected as covered in the pharmacogenetic blood sample amendment (Amendment 01), where applicable.

#### 5.7 Biomarker Assessments

Not applicable.

#### 5.8 Outcomes Research Assessments

Patient-reported outcomes (PROs) will be assessed as indicated in Table 5.1-2 and Table 5.1-3. The instruments/questions will be self-administered using paper and pencil questionnaires. The following PROs will be assessed in this trial:

- EQ-5D-3L for generic health status
- Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) for treatment satisfaction
- **Hypoglycemia Fear Survey (HFS-II)** for worries to avoid hypoglycemia and its negative consequences

PROs will be filled out prior to any other site activities and encounters with the study physician. The subjects will be instructed to complete the PRO questionnaires independently. The site will have a designated quiet space for subjects to use when completing the assessments. Each center should allocate responsibility for PRO assessment to a specified individual (eg, a research nurse). The research nurse or appointed individual should stress the information is confidential.

It is important that the value and relevance of health-related quality of life (HRQoL) data are explained carefully to participating subjects so that they are motivated to comply with data collection. The research nurse or appointed individual should also stress that the information is confidential. Therefore, if the subject has any medical problems s/he should discuss them with the doctor or research nurse separately from their PRO assessment.

The instructions for completion of questionnaires are:

- It should be completed before any investigations or discussions about the status of the subject's disease with the clinic staff
- The subject should complete it her/himself without any intervention from family, friends, center staff etc


v3.0 930087408 3.0

- Only one answer to every question should be checked
- Center personnel should not review the responses to the questionnaire with the subject or with any other center staff

Following completion, the nurse or appointed individual may quickly scan the questionnaire visually for completeness and should confirm verbally with the subject that the questionnaire has been completed fully.

#### 5.8.1 EQ-5D-3L

The EQ-5D-3L is a generic, preference-based utility questionnaire and consists of two parts, the EQ visual analogue scale (VAS) and the EQ-5D-3L index. The EQ VAS ranges from 0 = worst possible health to 100 = best possible health. The EQ-5D-3L index is a five dimension questionnaire. The dimensions consist of mobility, self-care, usual activity, pain/discomfort and anxiety/depression. Each item has three levels: no problems, some problems and severe problems.

#### 5.8.2 Diabetes Treatment Satisfaction Questionnaire

The Diabetes Treatment Satisfaction Questionnaire (DTSQ) has been developed to assess patient's satisfaction with treatment and perception of change in hyper- and hypoglycaemia <sup>18</sup>. The DTSQ status version (DTSQs) has 8 items.

## 5.8.3 Hypoglycemia Fear Survey

The Hypoglycemia Fear Survey (HFS-II) includes two subscales, of which one is an 18-item Worry Subscale that measures worries about hypoglycemia and its negative consequences (ie, describe specific concerns that patients may have about their hypoglycemic episodes). Responses are made on a 5-point Likert scale where 0 = Never and 4 = Always. The Worry Subscale has a score range of 0 to 72, with higher scores indicating increased fear of hypoglycaemia. The HFS-II is a widely used measure in clinical trials, has been translated into more than 20 languages, and has demonstrated reliability and validity. <sup>19</sup>

#### 5.9 Other Assessments

#### 5.9.1 Weight

Body weight will be measured according to the schedule presented in the study flow chart/time and event schedule (see Section 5.1) and will be recorded in the eCRF. The study-site staff should use a digital precision scale if possible, and record the weight in kilograms or pounds to the first decimal point (eg, 69.3 kg). The subject should wear a standard hospital-type gown or equivalent light indoor clothing, shoes removed, and bladder empty for the body weight measurement at each visit. Subjects should be weighed on the same scale at all visits.

## 5.9.2 Height and Body Mass Index (BMI)

 Measurement of height should be performed with the subject's shoes removed. The subject's knees should be straightened, head held erect and eyes forward


v3.0 930087408 3.0

• BMI is used as an index of obesity and is a method of defining normal body weight and excess body fat. BMI is determined by weight (kg) divided by height (m) squared

#### Method of BMI calculation:

- Use actual height and weight
- To calculate BMI:
  - convert pounds (lbs) to kilograms (kg = lb / 2.2)
  - convert inches (in) to meters (in x 0.0254)
  - BMI = (weight in kg) / (height in meter)  $^2$

## 5.9.3 Diet and Exercise Counseling

Starting at entry into the lead-in period (Week -8 visit), subjects will be instructed on a diet and an exercise program in accordance with the American Diabetes Association (ADA) or similar local guidelines to be followed for the study duration.

A registered dietitian, registered nurse, physician, certified diabetes educator (CDE), nutritionist, or other qualified member of the study team who has appropriate documented training, will provide this counseling.

## 5.9.4 Pharmacodynamic Assessments

#### 5.9.4.1 Fasting Plasma Glucose

Blood samples will be drawn for measurement of fasting plasma glucose concentrations according to the schedule presented in study flow chart/time and event schedule (see Section 5.1).

#### 5.9.4.2 6-point SMBG profiles

Subjects will be instructed to perform 6-point SMBG profiles as described below. <u>It is strongly preferred that subjects use the meter provided by the Sponsor</u>. If a subject uses another meter to perform this test, the site must try to determine the medium that the meter reports in (ie, plasma glucose vs. whole blood glucose). This information and results will be captured on an eCRF page. If subjects do not use the meter provided by the Sponsor, they should be instructed to continue using the same meter for all subsequent visits to avoid increasing variability.

Profiles will be obtained on any 3 days within a week before the Week -4 visit, Day 1 visit, Week 12 visit, and Week 24 visit, according to the schedules presented in study flow chart/time and event schedule (see Section 5.1). Each separate 6-point SMBG profile encompasses 1 day within one week before the scheduled visits, with three glucose measurements obtained preprandially (within 15 minutes prior to meal) and three glucose measurements obtained postprandially (1.5 - 2 hours after the start of the meal) for the three main meals of the day. Subjects will be provided with a diary to record these SMBG measurements and mealtimes, and eCRFs will available for the investigator sites to capture these results.


Date: 18-May-2016 78

If a lead-in subject fails prior to the Day 1 visit, the 6-point SMBG profile will not be required between the week -1 visit and the Day 1 visit.

If a randomized subject terminates the study any time prior to the Week 24 visit, the 6-point SMBG profile will not be required for the early termination visit. However, the 6-point SMBG is expected to be performed at Week 12 and 24 off treatment visit, if the subject decides to continue with the study procedures.

## 5.9.4.3 Continuous Glucose Monitoring (CGM)

CGM measures the subject's interstitial glucose level using electrodes that measure an electric signal produced by glucose oxidase reaction. The system records data approximately every 5 minutes. CGM will be used periodically to measure the subject's interstitial glucose level according to the schedule presented in study flow chart/time and event schedule (see Section 5.1).

A CGM sensor will be inserted subcutaneously at the Week - 2 visit, at the Week - 1 visit (and removed prior to the first dose on the Day 1 visit), and at the Week 10 and Week 22 visits to allow for monitoring of a 2 week time period (for example: the Week -2 visit to the Day 1 visit [baseline]; the Week 10 office visit until the Week 12 office visit; and the Week 22 office visit until the Week 24 office visit.) <u>During those periods, subjects will document their three main meal times in the diary every day.</u> Subjects should be trained to perform sensor replacement at Week-1 visit. In addition, at Week-1, sites should upload the sensor data to check subject's compliance with wearing the device.

The sensor requires at least one SMBG values to be entered every 12 hours for calibration during use. At a minimum, a SMBG value obtained in the morning (eg, fasting or pre-breakfast measurement) should be entered, as well as a value in the evening (eg, pre- or post-dinner measurement). Subjects may be instructed to use results from the 4 daily SMBG measures to fulfill this criteria. Every 7 days the sensor needs to be replaced and subjects can return to the site for assistance on this, if needed. If the subject needs assistance with sensor replacement, an ad-hoc visit should be performed; if this occurs a data upload is also recommended at this time. If subjects opt to perform sensor replacement at home, sites should call subject 7 days after insertion as a reminder. Please refer to the CGM Manual for further instructions on data uploads during an ad-hoc visit.

The data will remain blinded to the subject, the investigator, and to the Sponsor during the recording and will be downloaded into a data file. The downloaded file should be printed and reviewed by the site for review of monitoring compliance. The subjects should make every attempt to be at or greater than 100% compliant with use of the device. If a subject is not compliant, the reason should be discussed with the subject, documented in source notes, and the subject should be re-educated about the importance of CGM compliance.

Detailed procedures (including calibration) will be described in an operations manual and site staff will be fully trained on the use of CGM. Subjects will be instructed on use of the device and calibration according to manufacturer's instructions. Subjects will wear the sensor and perform calibration according to manufacturer's instructions.


930087408 3.0

v3.0

If a subject uses a CGM device prior to entry into the study, he/she may continue to use their personal device during the study in accordance with their usual diabetes management care. Such a subject will be required to also use the blinded CGM device according to protocol procedures.

If a lead-in subject fails lead-in prior to the Day 1 visit, the CGM will not be required to be completed between the week -2 visit and the Day 1 visit. In addition, the meal recording for 7 days will not be required between the week -1 visit and the Day 1 visit.

If a randomized subject terminates the study any time prior to the Week 24 visit, the CGM and meal recording for 7 days during the second week of CGM will not be required for the early termination visit. However, CGM and meal recording is expected to be performed at week 12 and week 24 off treatment visits, if the subject decides to continue with the study procedures after discontinuation of study drug.

## 5.10 Results of Central Laboratory Assessments

Blood and urine samples will be obtained at specified time points for laboratory evaluations (see Appendix 2). The central laboratory for this study will perform the analysis of all scheduled laboratory tests and will provide reference ranges for these tests. The central laboratory will provide specific instructions for collection, processing, packaging, and shipping of all samples.

During the short-term double-blind treatment periods (Day 1 to Week 24), the HbA1c, continuous glucose monitoring values, and urinary glucose values, including spot urine for glucose, albumin and creatinine quantification, determination of glucose:creatinine and albumin:creatinine ratios, and urine glucose dipstick values, will be masked to the Sponsor and will not be available to the investigator. During the long-term subject- and site-blinded treatment period, (after Week 24 and through Week 56), the above measurements will be unmasked to the Sponsor. However, these values will still not be available to the investigator, except for the HbA1c values, until after study completion. HbA1c values will be provided to the investigator during the subject- and site-blinded treatment period.

#### 6 ADVERSE EVENTS

An *Adverse Event (AE)* is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product.

The causal relationship to study drug is determined by a physician and should be used to assess all adverse events (AE). The casual relationship can be one of the following:

- Related: There is a reasonable causal relationship between study drug administration and the AE
- Not related: There is not a reasonable causal relationship between study drug administration and the AE


The term "reasonable causal relationship" means there is evidence to suggest a causal relationship.

AEs can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more AEs.)

#### 6.1 Serious Adverse Events

A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:

- results in death
- is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
- requires inpatient hospitalization or causes prolongation of existing hospitalization (see **NOTE** below)
- results in persistent or significant disability/incapacity
- is a congenital anomaly/birth defect
- is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the subject or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above). Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.) Potential drug induced liver injury (DILI) is also considered an important medical event. (See Section 6.6 for the definition of potential DILI).

Suspected transmission of an infectious agent (eg, pathogenic or nonpathogenic) via the study drug is an SAE.

Although pregnancy, overdose, cancer, and potential drug induced liver injury (DILI) are not always serious by regulatory definition, these events must be handled as SAEs. (See Section 6.1.1 for additional information on reporting pregnancies).

#### NOTE:

The following hospitalizations are not considered SAEs in BMS clinical studies:

- a visit to the emergency room or other hospital department < 24 hours, that does not result in admission (unless considered an important medical or life-threatening event)
- elective surgery, planned prior to signing consent
- admissions as per protocol for a planned medical/surgical procedure
- routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy)


• medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases

• admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (eg, lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason)

## 6.1.1 Serious Adverse Event Collection and Reporting

The Investigator Brochure (IB) includes Reference Safety Information to determine expectedness of SAEs for expedited reporting. Following the subject's written consent to participate in the study, all SAEs, whether related or not related to study drug, must be collected, including those thought to be associated with protocol-specified procedures. All SAEs must be collected that occur during the screening period and within 30 days of discontinuation of dosing.

The investigator should report any SAE that occurs after these time periods and that is believed to be related to study drug or protocol-specified procedure.

An SAE report should be completed for any event where doubt exists regarding its seriousness.

If the investigator believes that an SAE is not related to study drug, but is potentially related to the conditions of the study (such as withdrawal of previous therapy or a complication of a study procedure), the relationship should be specified in the narrative section of the SAE Report Form.

SAEs, whether related or not related to study drug, and pregnancies must be reported to the AstraZeneca within 24 hours. SAEs must be recorded on the SAE Report Form and pregnancies must be recorded on a Pregnancy Surveillance Form (electronic or paper forms). When using paper forms, the reports are to be transmitted via email or confirmed facsimile (fax) transmission to:



Note: All numbers redirect to the same recipient – so chose the most convenient number.

For studies capturing SAEs through electronic data capture (EDC), electronic submission is the required method for reporting. The paper forms should be used and submitted immediately, only in the event the electronic system is unavailable for transmission. When paper forms are used, the original paper forms are to remain on site.

**SAE Telephone Contact** (required for SAE and pregnancy reporting): Contact should be made to AZ or its designee. Refer to provided Contact Information list.


930087408 3.0

v3.0

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports should include the same investigator term(s) initially reported.)

If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, a follow-up SAE report should be sent within 24 hours to AstraZeneca using the same procedure used for transmitting the initial SAE report.

All SAEs should be followed to resolution or stabilization.

#### 6.2 Nonserious Adverse Events

A *nonserious adverse event* is an AE not classified as serious.

## 6.2.1 Nonserious Adverse Event Collection and Reporting

The collection of nonserious AE information should begin at initiation of study drug. Nonserious AE information should also be collected from the start of a placebo lead-in period or other observational period intended to establish a baseline status for the subjects.

Nonserious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious (see Section 6.1.1). Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study drug and for those present at the end of study drug as appropriate. All identified nonserious AEs must be recorded and described on the nonserious AE page of the CRF (paper or electronic).

Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.

See Section 6.7.1 regarding the collection and reporting of non-serious events necessary to meet the post-marketing commitments required by the FDA.

## 6.3 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the nonserious AE CRF page or SAE Report Form (paper or electronic) as appropriate:

- Any laboratory test result that is clinically significant or meets the definition of an SAE
- Any laboratory test result abnormality that required the subject to have study drug discontinued or interrupted


• Any laboratory test result abnormality that required the subject to receive specific corrective therapy

It is expected that wherever possible, the clinical, rather than laboratory term, would be used by the reporting investigator (eg, anemia versus low hemoglobin value).

## 6.4 Pregnancy

If, following initiation of the investigational product, it is subsequently discovered that a study subject is pregnant or may have been pregnant at the time of study exposure, including during at least 5 half-lives (approximately 3 days) after product administration, the investigator must immediately notify the BMS (or designee) Medical Monitor of this event and complete and forward a Pregnancy Surveillance Form to AZ (or designee) within 24 hours and in accordance with SAE reporting procedures described in Section 6.1.1.

In most cases, the study drug will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for subject safety).

In the rare event that the benefit of continuing study drug is thought to outweigh the risk, after consultation with BMS and/or AZ, the pregnant subject may continue study drug, after a thorough discussion of benefits and risk with the subject.

Protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (eg, x-ray studies). Other appropriate pregnancy follow-up procedures should be considered if indicated.

Follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcomes and, where applicable, offspring information must be reported on the Pregnancy Surveillance Form

Any pregnancy that occurs in a female partner of a male study participant should be reported to AZ. Information on this pregnancy will be collected on the Pregnancy Surveillance Form.

#### 6.5 Overdose

An overdose is defined as the accidental or intentional administration of any dose of a product that is considered both excessive and medically important. All occurrences of overdose must be reported as an SAE (see Section 6.1.1 for reporting details).

## 6.6 Potential Drug Induced Liver Injury (DILI)

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event. All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 6.1.1 for reporting details).

Potential drug induced liver injury is defined as:

Aminotransferase (ALT or AST) elevation > 3x upper limit of normal (ULN)

**AND** 


Date: 18-May-2016 84

Total bilirubin (TB) > 2x ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

#### AND

No other immediately apparent possible causes of aminotransferase elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic

## 6.7 Other Safety Considerations

Any significant worsening noted during interim or final physical examinations, electrocardiograms, x-ray filming, any other potential safety assessment required or not required by protocol should also be recorded as a nonserious or serious AE, as appropriate, and reported accordingly.

## 6.7.1 AEs of Special Interest

Event categories of special interest for this study may include, but are not limited to, hypoglycemia, fractures, hepatobiliary adverse events, genital infections, urinary tract infections, volume depletion, worsening renal function, hypersensitivity, and DKA.

For the purposes of regulatory reporting, the following events must be reported within 24 hours regardless of whether the events are classified as serious or non-serious:

#### Liver test abnormalities accompanied by jaundice or hyperbilirubinemia

This category of events include all AEs where hepatocellular damage (with elevations of ALT or AST > 3x ULN) is combined with hepatic dysfunction (with elevation of total bilirubin > 2x ULN) or jaundice. With respect to LFT abnormalities, both central-lab results and adverse events will be monitored

For each non-serious event in this category, notify the Medical Monitor within 24 hours to discuss next steps in reporting.

# 7 DATA MONITORING COMMITTEE AND OTHER EXTERNAL COMMITTEES

## 7.1 Cardiovascular Adjudication Committee

An Independent Adjudication Committee, blinded to the treatment of subjects, will classify cardiovascular adverse events, such as, but not limited to, death, myocardial infarction, and stroke reported in the study (see Section 5.3.6 for more details).

A separate Adjudication Charter will define and describe the procedure for the handling, reporting and classification of these events.


Date: 18-May-2016 85

## 7.2 Hepatic Adjudication Committee

An Independent Adjudication Committee, blinded to the treatment of the subjects, will determine the probability that drug-induced liver injury (DILI) is the cause of liver-related abnormalities, including but not limited to:

- AST and/or ALT > 3X ULN and TB >2 X ULN (within 14 days of the AST and/or ALT elevation)
- Hepatic events timely related to death (within 30 days before death)
- AST and/or ALT > 10X ULN

A separate Adjudication Charter will define and describe the procedure for the handling, reporting, and classification of these events.

## 7.3 DKA Adjudication Committee

A DKA Adjudication Committee, blinded to the treatment of the subjects, will independently adjudicate all the DKA events reported by investigators during the study period.

A separate Adjudication Manual will define and describe the procedure for the handling, reporting, and classification of these cases.

## 7.4 Data Monitoring Committee (DMC)

An external DMC with multidisciplinary representation will be established to evaluate, on a periodic basis, the incidence of hypoglycemia and DKA events, as well as AEs, laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects. An independent reporting statistician not involved in the conduct of the study will be designated by BMS to provide the DMC with essential safety data during the study.

The DMC responsibilities, authorities, and procedures will be documented and followed according to the DMC charter.

#### 8 STATISTICAL CONSIDERATIONS

#### 8.1 Sample Size Determination

The primary endpoint is the change from baseline in HbA1c to Week 24

With 243 subjects per treatment group with both baseline and at least one post baseline measurement, there is approximately 90% power to detect a difference in means of 0.35% between each dapagliflozin treatment group and placebo at the two-sided 0.0262 significance level (based on Dunnett and Tamhane step-up procedure), assuming a standard deviation (SD) of 1.1%. Assuming that 5% of subjects do not have a post-baseline assessment, a total of 768 subjects (256 subjects per treatment arm) need to be randomized to each dapagliflozin or placebo group in 1:1:1 ratio.

Among those 768 subjects, approximately 160 of them are planned to be from Japan in order to support population specific analyses.


A reduction in the primary endpoint of change from baseline in HbA1c of 0.35% was used to determine the sample size, as this represents a clinically meaningful improvement in glycemic control under the current study design with adjustable background insulin dose. A lesser degree of reduction in HbA1c in combination with other beneficial outcomes in secondary endpoints may also be clinically important.

## 8.2 Populations for Analyses

The following datasets will be used for analyses:

- **Enrolled subjects dataset**: The enrolled subjects dataset includes data collected from all subjects who signed informed consent.
- <u>Lead-in subjects dataset</u>: The lead-in subjects dataset includes data collected from all subjects who have at least one vital sign measurement during the lead-in period.
- <u>Full analysis dataset</u>: The full analysis dataset will consist of all randomized subjects who took at least one dose of double-blind study medication during the short-term double-blind period. Whenever using the full analysis dataset, subjects will be presented in the treatment group to which they were randomized at the start of the short-term double-blind treatment period (even if the treatment they received was different).
- Evaluable subjects dataset: The evaluable subjects dataset will be a subset of the full analysis dataset through exclusion of subjects with important protocol deviations. Important protocol deviations are those that have the potential to impact the results of the primary analysis. Detailed exclusion criteria for the evaluable subjects dataset will be specified in the SAP. All decisions to exclude data from the full analysis dataset to form the evaluable subjects dataset will be made prior to the unblinding of the study.
- Treated subjects dataset: The treated subjects dataset consists of all subjects who received at least one dose of double-blind study medication during the short-term double-blind treatment period. The treated subjects dataset would include any subject who accidentally received double-blind study medication but was not randomized in the study. These subjects will be included in analyses using the treated subject dataset in the treatment they received. For randomized subjects, all analyses using the treated subject dataset will be presented by randomized treatment group, except in cases where information was available which indicated that a subject received a different treatment for the entire course of their participation in the study (or period). In this case, the safety data for those subjects will be presented by the treatment actually received. In cases where a subject never received the treatment as assigned by randomization, then the safety data for that subject will be presented by the first treatment received.
- <u>Short-term completers dataset</u>: The short-term completers dataset will consist of all subjects in the full analysis dataset who completed the short-term double-blind treatment period. Whenever using the short term completers dataset, subjects will be presented in the treatment group to which they were randomized at the start of the short-term double-blind


treatment period (even if the treatment they received in the short-term or long-term was different).

Efficacy analyses will be performed using the full analysis dataset, which is considered as the primary efficacy dataset. Primary efficacy analysis will be reanalyzed using the evaluable subjects' dataset if more than 10% of the subjects in any treatment group are found to significantly violate the terms and conditions of the protocol. Otherwise, efficacy analysis will be restricted to the primary efficacy dataset.

Safety analyses will be based on the treated subjects dataset which consists of all subjects who received at least one dose of double-blind study medication.

#### 8.3 Endpoints

## 8.3.1 Primary Endpoint

The primary endpoint of this study is the change in HbA1c from baseline to Week 24.

#### 8.3.2 Secondary Endpoints

The secondary efficacy endpoints are:

- 1. Percent change from baseline to Week 24 in total daily insulin dose
- 2. Percent change from baseline to Week 24 in body weight
- 3. Change from baseline to Week 24 in the mean value of 24-hour glucose readings obtained from CGM
- 4. Change from baseline to Week 24 in mean amplitude of glucose excursion (MAGE) of 24-hour glucose readings obtained from CGM
- 5. Change from baseline to Week 24 in the percent of 24-hour glucose readings obtained from CGM that falls within the range of > 70 mg/dL and ≤ 180 mg/dL
- 6. Proportion of subjects achieving an HbA1c reduction from baseline to Week  $24 \ge 0.5\%$  and without severe hypoglycemia events.

#### 8.3.3 Safety

The safety endpoints include:

- The proportion of subjects with hypoglycemia events and the frequency and severity of the hypoglycemia events
- The proportion of subjects experiencing adverse events (AE), DKA events, and marked abnormalities in clinical laboratory tests
- The change from baseline at each post-baseline time point of assessment of selected safety clinical laboratory parameters, physical measurements, vital signs, and electrocardiogram data


## 8.3.4 Exploratory Endpoints

The efficacy exploratory endpoints of the study are:

1) Proportion of subjects with HbA1c reduction from baseline to Week 24 of at least 0.5% ( $\geq 0.5\%$ )

- 2) Proportion of subjects with HbA1C < 7.0% after 24 weeks of double-blinded treatment
- 3) Change from baseline to Week 24 in FPG
- 4) Change from baseline to Week 24 in the percent of 24-hour glucose readings obtained from CGM that falls within the hypoglycemic range of  $\leq 70 \text{ mg/dL}$
- 5) Change from baseline to Week 24 in seated systolic blood pressure among subjects with hypertension at baseline, defined as seated SBP  $\geq$  140 mmHg and/or seated DBP  $\geq$  90 mmHg
- 6) Change from baseline to Week 24 in average glucose values measured by 6-point self monitored blood glucose (SMBG)
- 7) Change from baseline to Week 24 in postprandial glucose values measured by 6-point self monitored blood glucose (SMBG)
- 8) Change from baseline to Week 24 in postprandial glucose values measured by CGM
- 9) Change from baseline to Week 24 in the standard deviation of 24-hour glucose readings obtained from CGM
- 10) Change from baseline to Week 24 in each of the 5 dimensions, as well as the health status index of the EQ-5D-3L questionnaire
- 11) Changes from baseline to Week 24 in the summary score for treatment satisfaction and scores for perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively, as measured by the Diabetes Treatment Satisfaction Questionnaire status (DTSQs)
- 12) Changes from baseline to Week 24 in the summary score of the Hypoglycemia Fear Survey (HFS-II) Worry Subscale between the dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
- 13) To explore the relationship between observed and/or model estimated pharmacokinetic measures of exposure (eg, AUCss, Cmax, Cmin) and efficacy and/or safety endpoints by using model-based approaches. This analysis will be provided in a separate report
- 14) Number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of  $\geq 0.5\%$

#### 8.4 Analyses

Analyses of the data from the short-term period will be conducted once all randomized subjects have either completed the short-term double-blind period or discontinued study medication from the short-term double-blind period. In addition all relevant queries must be resolved and the database must be locked for this period before the blind is broken for analyses.


Analyses of the data from both short-term double-blinded and long-term subject- and site-blinded treatment periods will be performed after all subjects have completed or have been discontinued from the study. In addition, all relevant queries must be resolved and the database must be locked for this study prior to analyses.

## 8.4.1 Demographics and Baseline Characteristics

Frequency distributions and summary statistics for demographic and baseline variables summarized in efficacy analyses will be computed by treatment group, as well as for all subjects combined. No statistical test will be carried out for comparison of any baseline measurement among the treatment groups.

## 8.4.2 Efficacy Analyses

Unless otherwise specified, efficacy analyses will be performed using the full analysis dataset.

## 8.4.2.1 Primary Efficacy Analyses

The primary endpoint is the change in HbA1c from baseline to Week 24. The primary estimand for the primary endpoint is *treatment difference at Week 24 if subjects did not discontinue randomized treatment*. In order to maintain an overall Type I error rate of 5% for the endpoint, a Dunnett and Tamhane step-up procedure will be used, which allows for the correlation of 0.5 between the standard normal deviate for each comparison (Dunnett and Tamhane 1992). Applying the Dunnett and Tamhane procedure, statistical significance will be declared for both doses at the two-sided 5% level if the two-sided p-values from both pairwise comparisons are smaller than 5%. If the larger p-value among the two pairwise comparisons is greater than 5% and the smaller p-value is below 2.62%, then statistical significance will be declared for the latter comparison.

The primary analysis of the change in HbA1c from baseline to Week 24 will be based on a longitudinal repeated measures analysis using 'direct likelihood'. The analysis will be based on the full analysis dataset who have a baseline assessment and any post-baseline double-blind treatment period assessment. The analysis will include all available data up to Week 24 or until premature discontinuation of randomized treatment, whichever occurs first. The analysis will be conducted regardless of insulin up-titration. The model is based on a missing at random (MAR) assumption with respect to missing data.

The SAS procedure PROC MIXED will be used. The preferred model will include the fixed categorical effects of treatment, week, randomization stratification factor (ie, one term for each combination of all stratification factors) and treatment-by-week interaction, as well as the continuous fixed covariates of baseline measurement and baseline measurement-by-week interaction. An unstructured matrix for the within-subject error variance-covariance will be used. The denominator degrees of freedom will be calculated according to the Kenward-Roger method. A number of back-up models will be defined in the statistical analysis plan in case of non-convergence of the preferred model or other issues. Point estimates and 95% confidence intervals for the mean change within each treatment group as well as the difference in mean change between the dapagliflozin treatment group and placebo will be calculated. P-values for


the differences in the Week 24 estimates between each dapagliflozin group and placebo will be calculated.

The ITT estimand, i.e., *treatment difference at Week 24 regardless of treatment discontinuation*, will be evaluated as the secondary estimand of the primary endpoint. The analysis of the ITT estimand will include all available data up to Week 24, regardless of insulin up-titration and regardless of premature discontinuation of randomized treatment.

Sensitivity analyses will be conducted for the primary efficacy endpoint to assess the robustness of the primary efficacy results, including sensitivity analysis with respect to the ITT estimand, sensitivity analyses based on missing-not-at-random (MNAR) assumptions with respect to missing data, and sensitivity analysis with respect to insulin up-titration.

## 8.4.2.2 Secondary Efficacy Analyses

Statistical tests for secondary efficacy endpoints will be only conducted if there is a statistically significant difference in the primary endpoint for both pairwise comparisons, i.e., dapagliflozin 5 mg vs. placebo and dapagliflozin 10mg vs. placebo. The same Dunnett and Tamhane step-up procedure will be applied to each secondary efficacy endpoint. Secondary efficacy endpoints will be tested in the order that they appear in the objectives section of the protocol and protocol synopsis. Statistical tests will be only performed for a given secondary endpoint if both comparisons for a proceeding secondary endpoint are significant. Otherwise, the testing procedure will stop at the secondary endpoint that does not reach statistical significance.

The percent change (using logarithmic transformation for the endpoint in the model) from baseline to Week 24 in total daily insulin dose and total body weight, the change from baseline to Week 24 in the mean value of 24-hour glucose readings obtained from CGM, mean amplitude of glucose excursions of 24-hour glucose readings obtained from CGM, and the percent of 24-hour glucose readings obtained from CGM that fall within the range of > 70 mg/dL and  $\leq$  180 mg/dL will be analyzed using a longitudinal repeated measures analysis, similarly to the model used for primary efficacy analysis. The proportion of subjects achieving an HbA1c reduction from baseline to Week 24 visit  $\geq$  0.5% without severe hypoglycemia events will be analyzed using a logistic regression model with adjustment for baseline value. In addition to point estimates and 95% confidence intervals, p-values will be calculated for all endpoints. Nominal p-values will be presented for endpoints where type 1 error is not controlled. All secondary efficacy analyses will use subjects in the primary efficacy dataset (ie, full analysis dataset) who have a baseline assessment and any post-baseline double-blind treatment period assessment.

## 8.4.2.3 Exploratory Efficacy Analyses

The proportion of subjects with HbA1c reduction from baseline to Week 24 last observation carried forward (LOCF) of at least 0.5% ( $\geq 0.5\%$ ) and the proportion of subjects with HbA1c at Week 24 LOCF < 7.0% will be summarized for each treatment group. For these analyses, LOCF refers to the Week 24 value, or the last post-baseline measurement prior to Week 24 if no measurement is available at Week 24. Poisson regression will be used to model number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of  $\geq 0.5\%$ . Point


Date: 18-May-2016 91

estimates and 2-sided 95% confidence intervals for the proportion in each treatment group and for the differences in proportions between each dapagliflozin treatment groups and the placebo treatment group will be calculated. No p-values will be generated.

The change from baseline to Week 24 in the following parameters will be analyzed using a longitudinal repeated measures model similar to the primary efficacy analysis:

- Fasting plasma glucose
- Percent of 24-hour glucose readings obtained from CGM that falls within the range of  $\leq 70 \text{ mg/dL}$
- Seated systolic blood pressure among subjects with hypertension at baseline, defined as seated SBP ≥ 140 mmHg and/or seated DBP ≥ 90 mmHg
- Average glucose values measured by 6-point SMBG
- Postprandial glucose values measured by 6-point SMBG
- Postprandial glucose values measured by CGM
- Standard deviation of 24-hour glucose readings obtained from CGM

## 8.4.3 Safety Analyses

The incidence of adverse events and of marked abnormalities in clinical laboratory tests will be summarized by treatment group.

The proportion of subjects with at least one hypoglycemic episode will be summarized by treatment group and by the severity of the events. The frequency of the hypoglycemia will also be summarized. Subjects with adjudicated DKA events will also be summarized by treatment group.

All AEs that are serious or that result in discontinuation of study therapy will be described in depth. Changes from baseline at each of the scheduled time points in each clinical laboratory parameter will be summarized by treatment group.

Changes from baseline at each of the scheduled time points in each selected safety clinical laboratory parameters, physical measurements, vital signs and electrocardiogram data will be summarized by treatment group.

## 8.4.4 Pharmacokinetic Analyses

The dapagliflozin plasma concentrations obtained by sampling of individual subjects will be used to build a population PK (PPK) model to estimate PK parameters (eg, oral clearance [CL/F], apparent volume of distribution [Vd/F], and absorption rate constant [ka]). Possible covariate effects on PK parameters may be identified and quantified. The estimated parameters will be used to derive individual exposure measures (eg, AUC, Cmin). Relationships between observed exposures, and/or these model-based estimates of exposures, and efficacy/safety endpoints (eg, changes from baseline in HbA1c, average daily glucose concentration, hypoglycemia) will be explored. The PK data and efficacy endpoint responses derived from this study may also be pooled with similar data from other studies to refine the model-based


Date: 18-May-2016 92

exposure-response relationship. Listings and summary statistics will be reported for the sampled pharmacokinetic measurements. The PPK and exposure-response analyses will be described in a separate report.

## 8.4.5 Biomarker Analyses

Not applicable

## 8.4.6 Outcomes Research Analyses

The change from baseline to Week 24 LOCF (Week 24 value or the last post-baseline measurement prior to Week 24 if no measurement is available at Week 24, [ie, last observation carried forward]) in each of the 5 dimensions of the EQ-5D-3L questionnaire will be analyzed with shift tables showing difference as to the respective classifications at baseline.

The change from baseline to Week 24 LOCF in the following will be analyzed as continuous variables: 1) health status index of the EQ-5D-3L questionnaire; 2) the summary score for treatment satisfaction and scores for perceived frequency of hyper- and perceived frequency of hypoglycemia, respectively, as measured by the Diabetes Treatment Satisfaction Questionnaire status (DTSQs); and 3) the summary score for HFS-II Worry Subscale. These will be analyzed using an ANCOVA model with treatment group as effect and baseline value and randomization stratification factor (ie, one term for each combination of all stratification factors) as covariates. Point estimates and 2-sided 95% confidence intervals for the mean change within each treatment group, as well as for the differences in the mean change between each dapagliflozin treatment group and the placebo treatment group will be calculated. No p-values will be generated.

All above mentioned analyses will use subjects in the primary efficacy dataset (ie, full analysis dataset) who have at least one baseline assessment and any post-baseline double-blind treatment period assessment.

#### 8.4.7 Other Analyses

Not applicable.

#### 8.5 Interim Analyses

There are no planned interim analyses for this study.

#### 9 STUDY MANAGEMENT

#### 9.1 Compliance

#### 9.1.1 Compliance with the Protocol and Protocol Revisions

The study shall be conducted as described in this approved protocol. All revisions to the protocol must be discussed with, and be prepared by BMS. The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion from the IRB/IEC of an amendment, except where necessary to eliminate an immediate hazard(s) to study subjects.


If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining IRB/IEC approval/favorable opinion, the deviation or change will be submitted as soon as possible to:

- IRB/IEC for review and approval/favorable opinion
- BMS
- Regulatory Authority(ies), if required by local regulations

Documentation of approval signed by the chairperson or designee of the IRB(s)/IEC(s) must be sent to BMS.

If an amendment substantially alters the study design or increases the potential risk to the subject: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from subjects currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new subjects prior to enrollment.

If the revision is done via an administrative letter, investigators must inform their IRB(s)/IEC(s).

## 9.1.2 Monitoring

Representatives of BMS/CRO must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable. Certain pages and/or electronic files may serve as the source documents, including but not limited to: CGM data, fingerstick blood glucose values recorded in the diary and meter data (SMBGs and ketones), insulin pump data, and the diary data as noted in Section 5.2.

In addition, the study may be evaluated by BMS internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to BMS.

## 9.1.3 Investigational Site Training

BMS will provide quality investigational staff training prior to study initiation. Training topics will include but are not limited to: good clinical practice (GCP), AE reporting, study details and procedure, electronic CRFs, study documentation, informed consent, and enrollment of WOCBP.

#### 9.2 Records

#### 9.2.1 Records Retention

The investigator must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period


Date: 18-May-2016 94

specified by BMS, whichever is longer. The investigator must contact BMS prior to destroying any records associated with the study.

BMS will notify the investigator when the study records are no longer needed.

If the investigator withdraws from the study (eg, relocation, retirement), the records shall be transferred to a mutually agreed upon designee (eg, another investigator, IRB). Notice of such transfer will be given in writing to BMS.

## 9.2.2 Study Drug Records

It is the responsibility of the investigator to ensure that a current disposition record of investigational product (those supplied by BMS) is maintained at each study site where study drug are inventoried and dispensed. Records or logs must comply with applicable regulations and guidelines and should include:

- Amount received and placed in storage area
- Amount currently in storage area
- Label identification number or batch number
- Amount dispensed to and returned by each subject, including unique subject identifiers
- Amount transferred to another area/site for dispensing or storage
- Nonstudy disposition (eg, lost, wasted)
- Amount destroyed at study site, if applicable
- Amount returned to BMS
- Retain samples for bioavailability/bioequivalence, if applicable
- Dates and initials of person responsible for Investigational Product dispensing/accountability, as per the Delegation of Authority Form

BMS will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

## 9.2.3 Case Report Forms

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for AEs and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the BMS electronic data capture tool, electronic CRFs will be prepared for all data collection fields except for fields specific to SAEs and pregnancy, which will be reported on the paper or electronic SAE form and Pregnancy Surveillance form, respectively. Spaces may be


Date: 18-May-2016 95

left blank only in those circumstances permitted by study-specific CRF completion guidelines provided by BMS.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF, including any paper or electronic SAE/pregnancy CRFs, must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a sub-investigator and who is delegated this task on the Delegation of Authority Form. For electronic CRFs, review and approval/signature is completed electronically through the BMS electronic data capture tool. The investigator must retain a copy of the CRFs including records of the changes and corrections.

Each individual electronically signing electronic CRFs must meet BMS training requirements and must only access the BMS electronic data capture tool using the unique user account provided by BMS. User accounts are not to be shared or reassigned to other individuals.

## 9.3 Clinical Study Report and Publications

A Signatory Investigator must be selected to sign the clinical study report.

For this protocol, the Signatory Investigator will be selected considering the following criteria:

- National Coordinating Investigator
- Involvement in trial design

The data collected during this study are confidential and proprietary to AZ. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the clinical trial agreement (CTAg) governing [Study site or Investigator] participation in the study. These requirements include, but are not limited to, submitting proposed publications to AZ at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTA.


Clinical Protocol BMS-512148

## 10 GLOSSARY OF TERMS

| Term | Definition |
|---|---|
| Adverse Reaction | An adverse event that is considered by either the investigator or BMS as related to the investigational product |
| Unexpected Adverse Reaction | An adverse reaction, the nature or severity of which is not consistent with the applicable product information (eg, Investigator Brochure for an unapproved investigational product) |
| Serious Adverse Event | Serious adverse event defined as any untoward medical occurrence that at any dose: results in death; is life threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization; results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; is an important medical event (defined as a medical event(s) that may not be immediately life threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the subject or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above). Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.). For reporting purposes only, BMS also considers the occurrence of pregnancy, overdose (regardless of association with an AE), and cancer as important medical events. |

Revised Protocol No.: 02 Date: 18-May-2016

# 11 LIST OF ABBREVIATIONS

| Term | Definition |
|-------|------------------------------------------|
| A1C | Glycosylated Hemoglobin |
| ADA | American Diabetes Association |
| AE | Adverse event |
| ALK-P | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUA | American Urological Association |
| AZ | AstraZeneca |
| BMI | Body mass index |
| BMS | Bristol-Myers Squibb |
| BP | Blood pressure |
| С | Celsius |
| CABG | Coronary artery bypass graft |
| CFR | Code of Federal Regulations |
| CEC | Clinical event committee |
| CGM | Continuous Glucose Monitoring |
| CHF | Congestive Heart Failure |
| CK | Creatine kinase |
| Cm | Centimeter |
| СРК | Creatine phosphokinase |
| CrCl | Creatinine Clearance |
| Cr | Creatinine |
| CRF | Case Report Form, paper or electronic |
| CRO | Contract Research Organization |
| CSII | Continuous subcutaneous insulin infusion |
| СТ | Computed Tomography |
| CTAg | Clinical Trial Agreement |
| CV | Cardiovascular |
| DBP | Diastolic blood pressure |

Revised Protocol No.: 02 Date: 18-May-2016

| Term | Definition |
|----------|-----------------------------------------------------|
| DKA | Diabetic Ketoacidosis |
| dL | Deciliter |
| DILI | Drug-induced liver injury |
| DMC | Data Monitoring Committee |
| DTSQs | Diabetes Treatment Satisfaction Questionnaire |
| DVT | Deep Vein Thrombosis |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| Eg | exempli gratia (for example) |
| EQ-5D-3L | Euro Quality of life 5 dimensions 3 levels |
| ET | Early Termination |
| FDA | Food and Drug Administration |
| FFA | Free Fatty Acid |
| FPG | Fasting Plasma Glucose |
| FSH | Follicle stimulating hormone |
| GCP | Good Clinical Practice |
| g/L | Grams/liter |
| g/dl | Grams/deciliter |
| GFR | Glomerular filtration rate |
| HbA1c | Glycosylated Hemoglobin |
| HBsAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| HCG | Human Chorionic Gonadotropin |
| HFS-II | Hypoglycemia Fear Survey II |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | Heart rate |
| HRQoL | Health related Quality of Life |
| HRT | Hormone replacement therapy |
| ICF | Informed Consent |


| Term | Definition |
|-------|-------------------------------------------|
| ICH | International Conference on Harmonisation |
| Ie | id est (that is) |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal products |
| IRB | Institutional Review Board |
| IU | International Unit |
| IUD | Intrauterine Device |
| IVRS | Interactive Voice Response System |
| Kg | kilogram |
| Lb | Pound |
| LFT | Liver function test |
| LOCF | Last observation carried forward |
| M | Meter |
| MAGE | Mean amplitude of glucose excursions |
| МСН | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |
| MDI | Multiple daily injections |
| Mg | milligram |
| mL | milliliter |
| MI | Myocardial infarction |
| Min | minute |
| Mmol | Millimole |
| MOA | Mechanism of Action |
| MODY | Maturity onset diabetes of young |
| NIMP | Non-investigational medicinal products |
| NSAID | Nonsteroidal anti-inflammatory drug |
| NYHA | New York Heart Association |
| PCI | Percutaneous Coronary Intervention |
| PE | Pulmonary Embolism |


v3.0 930087408 3.0

| Term | Definition |
|--------|------------------------------------------------|
| PK | Pharmacokinetics |
| PPK | Population Pharmacokinetics |
| PRO | Patient reported outcomes |
| PT | Prothrombin time |
| PTCA | Percutaneous transluminal coronary angioplasty |
| QD, qd | quaque die, once daily |
| RBC | Red blood cell |
| SA | Sickle cell trait |
| SAE | Serious adverse event |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SGLT-2 | Sodium-dependent glucose transporter 2 |
| SMBG | Self monitored blood glucose |
| SMQ | Standardized MedDRA Queries |
| SOP | Standard Operating Procedures |
| ТВ | Total bilirubin |
| TIA | Transient Ischemic Attack |
| TSH | Thyroid Stimulating Hormone |
| T1DM | Type 1 Diabetes Mellitus |
| T2DM | Type 2 Diabetes Mellitus |
| ULN | Upper limit of normal |
| UTI | Urinary Tract Infection |
| VAS | Visual Analogue Scale |
| WOCBP | women of childbearing potential |

Revised Protocol No.: 02 Date: 18-May-2016

#### 12 REFERENCES

- Daneman D. Type 1 Diabetes. Lancet 2006;367:847-58.
- <sup>2</sup> Cryer PE. Hypoglycaemia: The limiting factor in the glycaemic management of Type 1 and Type II Diabetes. Diabetologia 2002;45:937.948.
- Weinstock RS, Xing D, Maahs DM, Michels A, Rickels MR, Peters AL, et al. Severe hypoglycemia and diabetic ketoacidosis in adults with type 1 diabetes: results from the T1D Exchange clinic registry. J Clin Endocrinol Metab 2013;98(8):3411-9.
- <sup>4</sup> Kilpatrick ES, Rigby AS, Goode K, Atkin SL. Relating mean blood glucose and glucose variability to the risk of multiple episodes of hypoglycaemia in type 1 diabetes. Diabetologia. 2007;50(12):2553-61
- The Diabetes Control and Complications Trial Research Group. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin dependent diabetes mellitus. N Engl J Med 1993;329:977–986.
- Kilpatrick ES, Rigby AS, Atkin SL. Insulin resistance, the metabolic syndrome, and complication risk in type 1 diabetes: "double diabetes" in the Diabetes Control and Complications Trial. Diabetes Care. 2007;30(3):707-12.
- Ferriss JB, Webb D, Chaturvedi N, Fuller JH, Idzior-Walus B; The EURODIAB Prospective Complications Group. Weight gain is associated with improved glycaemic control but with adverse changes in plasma lipids and blood pressure in Type 1 diabetes. Diabet Med 2006;23(5):557-64.
- <sup>8</sup> Cleland SJ, Fisher BM, Colhoun HM, Sattar N, Petrie JR. Insulin resistance in type 1 diabetes: what is 'double diabetes' and what are the risks? Diabetologia. 2013;56(7):1462-70.
- Soedamah-Muthu SS, Chaturvedi N, Witte DR, Stevens LK, Porta M, Fuller JH for the EURODIAB Prospective Complications Study Group. Relationship between risk factors and mortality in type 1 diabetic patients in Europe: the EURODIAB Prospective Complications Study (PCS). Diabetes Care 2008;31(7):1360-6.
- Beck RW, Tamborlane WV, Bergenstal RM, Miller KM, DuBose SN, Hall CA for the T1D Exchange Clinic Network. The T1D exchange clinic registry. J Clin Endocrinol Metab 2012;97(12):4383-9.
- Investigator Brochure Version 07: Dapagliflozin (BMS-512148). Bristol-Myers Squibb Research and Development and AstraZeneca AB, 22-Dec-2010, BMS Document Control Number 930005487.
- Defronzo RA, Hompesch M, Kasichayanula S, Liu X, Hong Y, Pfister M, Morrow LA, Leslie BR, Boulton DW, Ching A, Lacreta FP, Griffen SC. Characterization of renal glucose reabsorption in response to dapagliflozin in healthy subjects and subjects with type 2 diabetes. Diabetes Care 2013;36:3169-3176.


v3.0 930087408 3.0

Perkins BA, Cherney DZ, Partridge H, Soleymanlou N, Tshirhart H, Zinman B, et al. Sodium-glucose cotransporter 2 inhibition and glycemc control in type 1 diabetes: results of an 8-week open-label proof-of-concept trial. Diabetes Care 2014;37:1480-83.

- Kestelman P. et. al., Efficacy of the Simultaneous Use of Condoms and Spermicides Family Planning Perspectives. Vol 23 (5); October 1991; Gabbay MB, Thomas J, Gibbs A, Hold P. A Randomized Crossover Trial of The Impact of Additional Spermicide on Condom Failure Rates. Sex Transm Dis 2008; 35: 862-8.
- Nicolle LE, Bradley S, Colgan R, Rice JC, Schaeffer A, Hooton TM. Infectious diseases society of America guidelines for the diagnosis and treatment of asymptomatic bacteriuria inadults. Clin Infect Dis 2005;40:643-54.
- US Preventative Services Taskforce. Recommendation Statement Screening or Asymptomatic Bacteriuria. Revised 2004. Available athttp://www.ahrq.gov/clinic/uspstf/uspsbact.htm
- European Association of Urology. Guidelines on the management of urinary and male genitaltract infections 2008. Available at http://www.uroweb.org/
- Bradley C (1994) The Diabetes Treatment Satisfaction Questionnaire: DTSQ. In Bradley C (ED) (1994) Handbook of Physchology and Dianetes: a guide to Psychological Measurement in diabetes research and practice. Chur, Switzerland: Harwood Academic Publishers.
- Gonder-Frederick L, Schmidt K, Vajda K, Greear M, Singh H, Shepard J, Cox D: Psychometric properties of the Hypoglycemia Fear Survey-II for adults with Type 1 diabetes. Diabetes Care 2011, 34:801-806.
- Dunnett CW and Tamhane AC. A step-up multiple test procedure. J of the American Statistical Association. 1992;87(417):162-170.

Revised Protocol No.: 02 Date: 18-May-2016

103

Page: 1

Protocol Number: MB102230 IND Number: 68,652

EUDRACT Number 2014-004599-49

Date: 18-May-2016

**Protocol MB102230:** A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Dapagliflozin as an Add-on to Insulin Therapy in Subjects with Type 1 Diabetes Mellitus -Study Two

Amendment Number 05 Site Number: All

#### **Study Director/Central Medical Monitor**

Lars Hansen, MD, PhD Route 206 & Province Line Road Lawrenceville, NJ 08543



#### **Bristol-Myers Squibb Research and Development**

Metabolics Clinical Research and Development
Avenue de Finlande 4
B-1420 Braine-l'Alleud, Belgium
Route 206 & Province Line Road
Lawrenceville, NJ 08543

This protocol amendment contains information that is confidential and proprietary to Bristol-Myers Squibb (BMS).

This amendment must be maintained with the referenced protocol.

Protocol Amendment 05 MB102230 BMS-512148 dapagliflozin

#### **Amendment Rationale:**

The primary purpose of this amendment is to provide study visit scheduling flexibility by allowing optional phone visits to be done at week -4, week 2 and for the Continuous Glucose Monitoring visits (weeks 10/11 and weeks 22/23) during the 24 week double blinded short term treatment period.

Additional changes in this amendment include:

- Adding an exploratory endpoint to compare the number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of  $\geq 0.5\%$  on dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin from baseline to Week 24 visit.
- Updating the guidance on DKA assessments and reporting to include the following:
  - Reductions in insulin doses of more than 20% are not recommended regardless of glucose values. If blood glucose is repeatedly low and a 20% reduction in total daily insulin dose cannot be avoided the daily dietary carbohydrate intake should be increased, as well as during and/or after elevated physical activity.
  - Investigators are recommended to advise subjects to take extra insulin and extra carbohydrates if elevated ketones are registered and to continue to measure blood ketones. Study medication should be interrupted during sick days if necessary
  - For subjects who report elevated ketones/ketosis or a DKA, it is recommended that the
    investigator consider reeducation concerning DKA at the next scheduled visit, at an unscheduled visit or by telephone contact
- Adding that if total daily insulin dose is reduced upon initiation of study medication, attempts must be made to titrate insulin back to baseline total daily insulin dose. It is not recommended to reduce total daily insulin dose by more than 20% compared to baseline at any time during the study unless medically indicated and close attention should be paid, especially in these subjects, to symptoms of, and risk factors for developing DKA.
- Revising the upper range of the Week -1 Visit: Central laboratory HbA1c to  $\leq 10.5\%$
- Adding multiple statistically related changes in this amendment including:
  - Adding the ITT estimand analysis and sensitivity analyses for the primary efficacy endpoint.
  - Replacing the single-step Dunnett procedure with the Dunnett and Tamhane step-up procedure for improved power and greater emphasis on primary endpoint.
  - Replacing "Randomized subjects dataset" with "Full analysis dataset".
  - Replacing the Zhang et al method with a general logistic regression model for implementation considerations.
  - Adding statistical method to model the added exploratory endpoint, number of number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of ≥ 0.5%
- Indicating that Tubal Ligation in this protocol is not considered surgical sterilization
- Removing the PK Sampling required at the Day 1 visit

Protocol Amendment 05
BMS-512148
MB102230
dapagliflozin

- Confirming that subjects are to record day and time of CGM sensor insertion if performed at home at week 11 and week 23
- Reinforcing that all results recorded in subject diary are to be reviewed by site staff during each study visit and that determination of a DKA event must be assessed and documented by the Principal Investigator or by a qualified sub-investigator
- Adding that blood ketone and glucose values associated with events that are deemed not to be a DKA event should be recorded on the non-DKA eCRF log page
- Including local injections such as intramuscular or intra-articular in the systemic corticosteroid therapy exclusion criteria as well as adding drops to the topical corticosteroids that are allowed in the study
- Clarifying that the Data Monitoring Committee will periodically evaluate the incidence of hypoglycemia and DKA events, as well as AEs, laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects.
- Adding multiple updates, confirmations and additions in the Study Flowchart

The changes included in the amendment apply to all subjects in the study with no impact expected on study conduct

#### **Changes to the Protocol:**

- 1. Cover Page, Study Director/Medical Monitor Contact Information: Updated Medical Director name and telephone number
- 2. Synopsis Other/Exploratory Objectives,  $14^{th}$  objective, Protocol Section 1.3.3 Other Exploratory Objectives,  $14^{th}$  objective: Added new objective for comparing the number of non-severe hypoglycemic events per subject in those achieving an HbA1c reduction of  $\geq 0.5\%$  on dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin from baseline to Week 24 visit
- 3. Synopsis Study Design, end of 2<sup>nd</sup> paragraph, Protocol Section 3 Investigational Plan, Section 3.1 Study Design and Duration, Protocol Section 4.4.1, Subjects entering the 24-week double-blinded short-term treatment period: Updated the higher end of the range of the Week -1 Visit: Central laboratory HbA1c to ≤ 10.5% in the third factor for randomization stratification
- 4. Synopsis Study Design, 3<sup>rd</sup> paragraph: Clarified the recommendation for daily insulin dose reduction is to be up to 20%
- 5. Synopsis, Figure 1, Study Schematic, Protocol 3.1-1 Study Design Schematic: Added Optional Phone visits for week -4, 2, 10, and 22
- 6. Synopsis Study Population, Key Inclusion Criteria, 4<sup>th</sup> bullet, Protocol Section 3.3.1 Inclusion Criteria 4b): Updated the higher end of the range of the Week -1 Visit: Central laboratory HbA1c to ≤ 10.5%
- 7. Synopsis Study Population, Key Exclusion Criteria, 6<sup>th</sup> bullet, Other Exclusion Criteria, fifth bullet, Protocol Section 3.3.2 Exclusion Criteria, 6) Other Exclusion Criteria, bullet e), Protocol Section 3.4.1 Prohibited and/or Restricted Treatments, 3<sup>rd</sup> bullet: Added local injections such as intramuscular or intra-articular, etc. as an example of systemic

- corticosteroid therapy excluded as well as adding drops to the topical corticosteroids that are allowed in the study
- 8. Synopsis Study Assessments, Safety Assessments: Added guidance that subjects must also be instructed that if attempts to contact the site are unsuccessful or if they are in urgent need of medical attention that they should seek medical attention. They should provide information to the health care provider on their participation in a placebo controlled clinical study evaluating the effects of the SGLT2i dapagliflozin in addition to their insulin treatment.
- 9. Synopsis Data Monitoring Committee, Protocol Section 7.4, Data Monitoring Committee: Clarified that DMC would periodically evaluate the incidence of hypoglycemia and DKA events, as well as AEs,
- 10. Synopsis Statistical Considerations, Sample Size, Protocol Section 8 Statistical Considerations, Section 8.1 Sample Size Determination:
  - a) Removed incorrect text in 2nd paragraph
  - b) Added new language for 243 subjects per treatment group with both baseline and at least one post baseline measurement, there is approximately 90% power to detect a difference in means of 0.35% between each dapagliflozin treatment group and placebo at the two-sided 0.0262 significance level (based on Dunnett and Tamhane step-up procedure), assuming a standard deviation (SD) of 1.1%.
- 11. Synopsis, Statistical Considerations, Statistical Approach / Assumptions, Protocol Section 8.4.2.1 Primary Efficacy Analyses
  - a) Removed second sentence in first paragraph and added The primary estimand for the primary endpoint is treatment difference at Week 24 if subjects did not discontinue randomized treatment.
  - b) Added In order to maintain an overall Type I error rate of 5% for the endpoint, a Dunnett and Tamhane step-up procedure will be used, which allows for the correlation of 0.5 between the standard normal deviate for each comparison (Dunnett and Tamhane 1992). Applying the Dunnett and Tamhane procedure, statistical significance will be declared for both doses at the two-sided 5% level if the two-sided p-values from both pairwise comparisons are smaller than 5%. If the larger p-value among the two pairwise comparisons is greater than 5% and the smaller p-value is below 2.62%, then statistical significance will be declared for the latter comparison.
  - c) Removed model will use subjects in the primary efficacy dataset (ie, randomized subjects dataset)
  - d) Added The analysis will be based on the full analysis dataset
  - e) Removed For subjects whose insulin dose is up-titrated by more than 25% of baseline insulin prior to randomization measurements, obtained after meeting the above insulin up-titration criteria will be excluded from the primary analysis but included in the sensitivity analysis. Multiple sensitivity analyses, including the sensitivity analyses using data regardless of insulin dose up-titration, will also be performed for the primary efficacy endpoint to assess
  - f) Added The analysis will include all available data up to Week 24 or until premature discontinuation of randomized treatment, whichever occurs first. The analysis will be conducted regardless of insulin up-titration. The model is based on a missing at random (MAR) assumption with respect to missing data

- g) Added will be evaluated as the secondary estimand of the primary endpoint. The analysis of the ITT estimand will include all available data up to Week 24, regardless of insulin up-titration and regardless of premature discontinuation of randomized treatment.
- h) Added Sensitivity analyses will be conducted for the primary efficacy endpoint to assess the robustness of the primary efficacy results, including sensitivity analysis with respect to the ITT estimand, sensitivity analyses based on missing-not-at-random (MNAR) assumptions with respect to missing data, and sensitivity analysis with respect to insulin up-titration.
- 12. Synopsis, Statistical Considerations, Statistical Approach / Assumptions, Protocol Section 8.4.2.2 Secondary Efficacy Analyses
  - a) Removed the original secondary efficacy analysis description
  - b) Added Statistical tests for secondary efficacy endpoints will be only conducted if there is a statistically significant difference in the primary endpoint for both pairwise comparisons, i.e., dapagliflozin 5 mg vs. placebo and dapagliflozin 10mg vs. placebo. The same Dunnett and Tamhane step-up procedure will be applied to each secondary efficacy endpoint. Secondary efficacy endpoints will be tested in the order that they appear in the objectives section of the protocol and protocol synopsis. Statistical tests will be only performed for a given secondary endpoint if both comparisons for a proceeding secondary endpoint are significant. Otherwise, the testing procedure will stop at the secondary endpoint that does not reach statistical significance
  - c) Replaced the Zhang et al method with a general logistic regression model for implementation considerations
  - d) End of last paragraph replaced However, no claim will be based on endpoints for which the statistical testing is not performed as per the testing strategy as described above. No claims can be made based on these p-values. A clear distinction will be made between p-values whereby claims can and cannot be made with Nominal p-values will be presented for endpoints where type 1 error is not controlled
  - e) Replaced randomized subject dataset with full analysis dataset
- 13. Section 3.3.1 Inclusion Criteria, 6) Age and Reproductive Status: Clarifed that tubal ligation is not considered surgically sterile
- 14. Section 5, Table 5.1-1 Flow chart for Protocol MB102229, Qualification and Lead-in Period:
  - a) Week -4: Added footnote c
  - b) Insert/calibrate CGM, Record Meals for 7 days Second week of CGM.: Added If a lead-in subject fails lead-in prior to the Day 1 visit, the CGM will not be required to be completed between the week-2 visit and the Day 1 visit (Please refer to Section 5.9.4.3)
  - c) 6-point SMBG profiles: Added If a lead-in subject fails prior to the Day 1 visit, the 6-point SMBG profile will not be required between the week -1 visit and the Day 1 visit
  - d) Pregnancy test (urine) WOCBP only: added footnote g for week -8 and week -4
  - e) Footnote c: Added details for Optional Phone Visit at week -4
  - f) Footnote g: Added If an optional phone visit is planned for week -4, the home pregnancy kit should be given to the subject at the week -8 visit.
- 15. Section 5, Table 5.1-2 Flow chart for Protocol MB102229, 24-week Double-blinded Short-term Treatment Period,
  - a) Week 2: Added footnote d

- b) Week 10 and Week 22: Added footnote e
- c) Insert/calibrate CGM: Added in Notes column If week 10 and week 22 are optional phone visits, please refer to footnote e below and Section 5.9.4.3 CGM.
- d) Insert/calibrate CGM, CGM Data Collection, data upload, and review, and Record Meals for7 days Second week of CGM: Added Note Please refer to Section 5.9.4.3
- e) Dispense subject diaries and provide instructions: Added footnote 1 in week 8 and week 18
- f) Dispense subject diaries and provide instructions: Added in Notes column At Day 1, collect Lead-In Period diaries and dispense the first diaries in the Short Term Treatment Period and added X to indicate the procedure needs to be done at week 10 and week 22 visits
- g) Review subject diaries, Adjust Insulin Dose, as needed, Assess Adverse Events, Assess Hypoglycemia Episodes, Assess DKA: Added X to indicate the procedure needs to be done at week 10 and week 22 visits
- h) PK sampling: Removed procedure requirement at Day 1
- i) Contact IVR system: Added footnote m at week 4, 8, 12, and 24
- j) Footnote d: Added the footnote with details for Optional Phone Visit at Week 2
- k) Footnote e: Added the footnote with details for Optional Phone Visit at Week 10 and/or Week 22
- 1) Footnote 1: Added the footnote If an optional phone visit is to be done at week 10, the subject diary should be given to the subject at week 8 and/or a new week 22 diary should be given at week 18
- m) Footnote m: Added the footnote to indicate that if visit is during the "off-treatment" or the Post Study Drug Study Follow-up phase (Section 3.6), the IVRS does not have to be contacted
- 16. Section 5, Table 5.1-3 Flow chart for Protocol MB102229, 28-week Subject and Site Blinded Long-term Treatment Period:
  - a) Included footnote a at week 52 to allow + 5 day visit window
  - b) Pregnancy test (urine) WOCBP only: Added and pregnancy logs to Notes
  - c) Contact IVR system: Added footnote c at week 32, 40, and 52
  - d) Footnote c: Added the footnote to indicate that if visit is during the "off-treatment" or the Post Study Drug Study Follow-up phase (Section 3.6), the IVRS does not have to be contacted
- 17. Section 5.2, Study Materials, Subject Diary:
  - a) Added to end of first bullet during each visit
  - b) Added to second bullet, day/time of CGM sensor insertion if performed at home at Weeks 11 and 23
    - i) Added fifth bullet Subjects are to record day and time of CGM sensor insertion if performed at home at week 11 and week 23
    - ii) Added at the end of the eighth bullet during each study visit. Determination of a DKA event must be assessed and documented by the Principal Investigator or by a qualified sub-investigator.

- 18. Section 5.3.3, Self-Monitored Blood Ketone Testing and Guidance on Management and Reporting of Diabetic Ketoacidosis Episodes:
  - a) Added guidance for reductions in insulin doses of more than 20% not recommended regardless of glucose values. If blood glucose is repeatedly low and a 20% reduction in total daily insulin dose cannot be avoided the daily dietary carbohydrate intake should be increased, as well as during and/or after elevated physical activity.
  - b) Added recommendation for the investigator to advise the subject to take extra insulin and extra carbohydrates if elevated ketones are registered and continue to measure blood ketones. If deemed necessary, dosing of study medication should be interrupted during sick days
  - c) Added guidance for the investigator to consider re-education concerning DKA at the next scheduled visit, at an un-scheduled visit or by telephone contact, as appropriate for subjects who report elevated ketones/ketosis
  - d) Added blood ketone and glucose values associated with events deemed not to be a DKA event should be recorded on the non-DKA eCRF log page.
  - e) Added reinforcement, that subjects who experience a DKA, it is recommended that the investigator schedules a telephone or site visit for re-education in prevention of ketosis and DKA
  - f) Section 5.3.4 Insulin Dosing Adjustment and Data Collection Guidelines: Added guidance that if total daily insulin dose is reduced upon initiation of study medication, attempts must be made to titrate insulin back to baseline total daily insulin dose. It is not recommended to reduce total daily insulin dose by more than 20% compared to baseline at any time during the study unless medically indicated and close attention should be paid, especially in these subjects, to symptoms of, and risk factors for developing DKA (See also Section 5.3.3).
- 19. Section 5.3.7 Guidance on Assessment of Hepatic Laboratory Abnormalities, Specialized Liver Laboratory Panel: Added clarification the Specialized Liver Lab Panel should only be done once for elevated liver enzymes per Appendix 3 Sustained Elevated Liver Safety Abnormalities Flow Chart unless liver discontinuation panel is required
- 20. Section 5.5 Pharmacokinetic Assessments: Removed PK Sampling at Day 1
- 21. Section 5.9.4.3 Continuous Glucose Monitoring (CGM): Added guidance on optional phone visits during CGM visits at week 10/11 and 22/23
- 22. Section 8 Statistical Considerations, Section 8.1 Sample Size Determination: Removed "For subjects whose insulin dose is up-titrated by more than 25% of insulin prior to randomization, measurements obtained after meeting the above insulin up-titration criteria will be excluded from the primary analysis of the primary efficacy endpoint."
- 23. Section 8.2 Populations for Analyses, Section 8.2.1 Definition of Analysis Datasets:
  - a) Randomized subjects dataset: Removed the section
  - b) Evaluable subjects dataset:
    - i) changed randomized subject dataset to full analysis dataset
    - ii) added through exclusion of subjects with important protocol deviations. Important protocol deviations are those that have the potential to impact the results of the primary analysis

- iii) removed It will exclude primary efficacy variable data which may have been affected by protocol deviations as determined by the medical monitor
- iv) added detailed exclusion criteria for the evaluable subjects dataset will be specified in the SAP
- v) replaced "data" with "subjects"
- c) Short-term completers dataset
  - i) changed randomized subject dataset to full analysis dataset
  - ii) deleted "changed randomized subject dataset to full analysis dataset"
- 24. Section 8.3.1 Primary Endpoint: removed second paragraph
- 25. Section 8.3.2 Secondary Endpoints: removed last paragraph
- 26. Section 8.3.4 Exploratory Endpoints:
  - a) added new exploratory endpoint of Number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of  $\geq 0.5\%$
  - b) removed the last paragraph
- 27. Section 8.4.2 Efficacy Analyses:
  - a) removed first sentence
  - b) added Unless otherwise specified, efficacy analyses will be performed using the full analysis dataset.
- 28. Section 8.4.2.2 Secondary Efficacy Analyses: removed last sentence in the section
- 29. Section 8.4.2.3 Exploratory Efficacy Analyses
  - a) added Poisson regression will be used to model number of non-severe hypoglycemic events per subject in those achieving a HbA1c reduction of  $\geq 0.5\%$
  - b) removed incorrect text in last paragraph
- 30. Section 8.4.6 Outcomes Research Analyses
  - a) changed randomized subject dataset to full analysis dataset
  - b) removed incorrect text in last paragraph
- 31 References
  - a) Deleted references 18) and 19)
  - b) Added new reference 18) Dunnett CW and Tamhane AC. A step-up multiple test procedure. J of the American Statistical Association. 1992;87(417):162-170

Please maintain a copy of this amendment with your protocol. Please provide a copy to your Investigational Review Board / Ethics Committee, unless agreed otherwise with BMS.

#### AMENDMENT ACKNOWLEDGMENT

I have read this Amendment and agree that it contains all necessary details for carrying out the changes described. I understand that it must be reviewed by the Institutional Review Board or Independent Ethics Committee overseeing the conduct of the study and approved or given favorable opinion by all necessary Health Authorities before implementation unless to eliminate an immediate hazard to subjects.

If this Amendment substantially alters the study design or increases potential risk to subjects, the consent form will be revised and submitted to the Institutional Review Board/Independent Ethics Committee for approval/positive opinion. I will use the new consent form for any new subjects prior to enrollment, and for subjects currently enrolled in the study if they are affected by the Amendment.

Investigator's printed name and signature

Date

PPD

Medical Monitor/Study Director (If required by applicable regulations and guidelines.) 07-JUN-7016

Protocol Number: MB102230

Site Number:

Amendment Number: 05